Replication of Prasugrel versus Clopidogrel in Patients with Acute Coronary Syndromes (TRITON-TIMI 38 Trial)

January 13, 2020

#### 1. RCT Details

This section provides a high-level overview of the RCT that the described real-world evidence study is trying to replicate as closely as possible given the remaining limitations inherent in the healthcare databases.

#### 1.1 Title

Prasugrel versus Clopidogrel in Patients with Acute Coronary Syndromes (TRITON-TIMI 38 trial)

### 1.2 <u>Intended aim(s)</u>

To compare prasugrel, a new thienopyridine, with clopidogrel, we randomly assigned 13,608 patients with moderate-to-high-risk acute coronary syndromes with scheduled percutaneous coronary intervention to receive prasugrel (a 60-mg loading dose and a 10-mg daily maintenance dose) or clopidogrel (a 300-mg loading dose and a 75-mg daily maintenance dose), for 6 to 15 months.

#### 1.3 Primary endpoint for replication and RCT finding

The primary efficacy end point was death from cardiovascular causes, nonfatal myocardial infarction, or nonfatal stroke. The key safety end point was major bleeding.

## 1.4 Required power for primary endpoint and noninferiority margin (if applicable)

We calculated that a total of 875 primary end points would be required for the study to have a 90% power to detect a 20% reduction in the relative risk of the primary end point among patients with unstable angina or non–ST-elevation myocardial infarction receiving prasugrel, as compared with clopidogrel.

### 1.5 Primary trial estimate targeted for replication

HR = 0.81 (95% CI 0.73–0.90) comparing prasugrel to clopidogrel (Wiviott et al., 2007)

## 2. Person responsible for implementation of replication in Aetion

Ajinkya Pawar, Ph.D. implemented the study design in the Aetion Evidence Platform. S/he is not responsible for the validity of the design and analytic choices. All implementation steps are recorded and the implementation history is archived in the platform.

Effectiveness research with Real World Data to support FDA's regulatory decision making: Protocol Template

## 3. Data Source(s)

United/Optum, MarketScan

## 4. Study Design Diagram

The study design diagram visualizes key aspects of the longitudinal study design for expedited review.



#### 5. Cohort Identification

## 5.1 Cohort Summary

This study will involve a new user, parallel group, cohort study design comparing prasugrel 90mg to clopidogrel 75mg. The patients will be required to have continuous enrollment during the baseline period of 180 days before initiation of prasugrel 90mg or a comparator drug (cohort entry date). Follow-up for the outcome (3P-MACE), begins the day after drug initiation.

## 5.2 <u>Important steps for cohort formation</u>

New users (defined as no use in 180 days prior to index date) of an exposure and a comparator drug will be identified.

### 5.2.1 Eligible cohort entry dates

Market availability of prasugrel in the U.S. started on 2009-07-10.

- For Marketscan: 2009-07-10 to 2017-12-31 (end of data availability).
- For Optum: 2009-07-10 to 2019-03-31 (end of data availability).

## 5.2.2 Specify <u>inclusion/exclusion</u> criteria for cohort entry and define the index date

Inclusion and exclusion criteria were adapted from the trial as closely as possible. Definitions for all inclusion/exclusion are provided in **Appendix A** and are summarized in the flowcharts below.

## 5.3 Flowchart of the study cohort assembly

| | Optum | | MarketScan | |
|---|---|---|---|---|
| | Less Excluded Patients | Remaining Patients | Less Excluded Patients | Remaining Patients |
| All patients | | 75,524,500 | | 191,990,035 |
| Patients meeting the cohort entry criteria of moderate to high risk Acute Coronary Syndrome undergoing PCI procedure | -75219388 | 305,112 | -191556394 | 433,641 |
| Patients with sufficient enrollment period in the claims database | -41910 | 263,202 | -120017 | 313,624 |
| Patients with moderate to high risk Acute Coronary Syndrome | -144114 | 119,088 | -165792 | 147,832 |
| Patients initiating clopidogrel 75mg or prasugrel 10mg within 14 days of discharge of PCI hospitalization | -56497 | 62,591 | -54511 | 93,321 |

| Patients without history of hemorrhagic stroke | -349 | 62,242 | -392 | 92,929 |
|---|---|---|---|---|
| Patients without intracranial neoplasm, AV malformation, or aneurysm | -186 | 62,056 | -202 | 92,727 |
| Patients without ischemic stroke occurring 90 days prior to PCI hospitalization | -163 | 61,893 | -255 | 92,472 |
| Patients with sufficient claims enrollment after PCI hospital discharge | -483 | 61,410 | -1191 | 91,281 |
| Parent: Final cohort | | 61,410 | | 91,281 |
| Did not meet cohort entry criteria | -80 | 61,330 | 0 | 91,281 |
| Excluded due to insufficient enrollment | 0 | 61,330 | 0 | 91,281 |
| Patients with no prior use of clopidogrel | -3135 | 58,195 | -3653 | 87,628 |
| Patients with no prior use of prasugrel | -535 | 57,660 | -958 | 86,670 |
| Patients without qualification in >1 exposure category | -18 | 57,642 | -20 | 86,650 |
| Patients age 18 years or older | -2 | 57,640 | 0 | 86,650 |
| Patients without cardiogenic shock during PCI hospitalization | -1811 | 55,829 | -2457 | 84,193 |
| Patients without refractory ventricular arrhythmias | -5341 | 50,488 | -7235 | 76,958 |
| Patients without New York Heart Association Class IV congestive heart failure | -416 | 50,072 | -265 | 76,693 |
| Patients without active internal bleeding or history of bleeding diathesis | -3974 | 46,098 | -3739 | 72,954 |
| Patients without thrombocytopenia (platelet count of less than 100,000/mm3) | 0 | 46,098 | 0 | 72,954 |
| Patients without anemia (hemoglobin <10 g/DI) | -886 | 45,212 | -2039 | 70,915 |
| Patients without a claim for thienopyridine 5 days or less before PCI hospitalization | -1 | 45,211 | -1 | 70,914 |
| Patients without daily treatments with NSAIDs or COX-2 inhibitors | -394 | 44,817 | -654 | 70,260 |
| Patients without concomitant medical illness that is potentially associated with reduced survival | -687 | 44,130 | -235 | 70,025 |
| Patients without severe hepatic dysfunction | -1755 | 42,375 | -2041 | 67,984 |
| Patients without issues on poor treatment compliance including alcoholism, mental illness, or drug dependence | -2927 | 39,448 | -1981 | 66,003 |
| Final cohort | | 39,448 | | 66,003 |

## 6. Variables

## 6.1 Exposure-related variables:

## Study drug:

The study exposure of interest is initiation of Prasugrel. Initiation will be defined by no use of Prasugrel or a comparator in the prior 6 months before treatment initiation (washout period).

Effectiveness research with Real World Data to support FDA's regulatory decision making: Protocol Template

#### Comparator agents:

- Initiators of prasugrel 10mg will be compared to initiators of-
  - Clopidogrel 75mg

#### 6.2 Preliminary covariates:

- Age
- Sex
- Combined Comorbidity Index (CCI), measured over the default baseline covariate assessment period, defined as 180 days prior to and including index date

Covariates listed above represent only a small subset of covariates that will ultimately be controlled for in the design and analysis. We use the covariates above only for initial feasibility analyses to judge whether there is likely to be sufficient overlap between treatment groups to proceed with the study. Remaining covariates are defined only after the study has passed the initial feasibility analysis and the initial power assessment and are listed in Table 1 (Appendix B).

### 6.3 Outcome variables and study follow-up:

#### 6.3.1 Outcome variables

Effectiveness outcomes of interest (definitions provided in **Appendix A**):

- <u>Primary outcome</u>: 3-point major adverse cardiovascular events (MACE), i.e., non-fatal myocardial infarction, non-fatal stroke, or CV mortality
- Secondary outcomes: Individual components:
  - o Hospital admission for MI (for purposes of this individual component, fatal MI is included)
  - Hospital admission for stroke (for purposes of this individual component, fatal stroke is included)
  - All-cause mortality/CV mortality:
    - All-cause inpatient mortality identified using discharge status codes will be used as a proxy for "CV mortality" in Marketscan
    - In Optum, all-cause inpatient mortality + all-cause mortality for Medicare Advantage patients is used

Control outcome of interest (control outcome only serve to assess aspects of study validity but are not further interpreted):

- 1. Major bleeding (we expect to see increased risk with prasugrel; Wiviott, 2007)
- 2. Pneumonia (we expect to see a null association)

## **Control outcome definition**

| Outcome | Definition | Comments |
|---|---|---|
| Control Outcomes | | |
| Major bleeding | Any inpatient diagnosis of major bleeding code list provided in <b>Appendix A</b> | Same code list used for both outcome and major bleed exclusion criteria |
| Pneumonia | Any inpatient diagnosis of pneumonia: * 481 - PNEUMOCOCCAL PNEUMONIA [STREPTOCOCCUS PNEUMONIAE PNEUMONIA] * 482 - OTHER BACTERIAL PNEUMONIA * 483 - PNEUMONIA DUE TO OTHER SPECIFIED ORGANISM * 485 - BRONCHOPNEUMONIA ORGANISM UNSPECIFIED * 486 - PNEUMONIA ORGANISM UNSPECIFIED * 487.0 - INFLUENZA WITH PNEUMONIA * 507 - PNEUMONITIS DUE TO SOLIDS AND LIQUIDS * 482.0 - PNEUMONIA DUE TO KLEBSIELLA PNEUMONIAE * 482.1 - PNEUMONIA DUE TO PSEUDOMONAS * 482.2 - PNEUMONIA DUE TO PSEUDOMONAS * 482.3 - PNEUMONIA DUE TO STREPTOCOCCUS * 482.3 - PNEUMONIA DUE TO STREPTOCOCCUS GROUP A * 482.3 - PNEUMONIA DUE TO STREPTOCOCCUS GROUP B * 482.3 - PNEUMONIA DUE TO STREPTOCOCCUS GROUP B * 482.3 - PNEUMONIA DUE TO OTHER STREPTOCOCCUS * 482.4 - PNEUMONIA DUE TO STAPHYLOCOCCUS * 482.4 - PNEUMONIA DUE TO STAPHYLOCOCCUS * 482.4 - PNEUMONIA DUE TO STAPHYLOCOCCUS * 482.4 - PNEUMONIA DUE TO STAPHYLOCOCCUS * 482.4 - PNEUMONIA DUE TO STAPHYLOCOCCUS UNSPECIFIED * 482.4 - PNEUMONIA DUE TO STAPHYLOCOCCUS UNSPECIFIED * 482.4 - PNEUMONIA DUE TO STAPHYLOCOCCUS UNSPECIFIED * 482.4 - PNEUMONIA DUE TO STAPHYLOCOCCUS UNSPECIFIED * 482.4 - PNEUMONIA DUE TO STAPHYLOCOCCUS UNSPECIFIED * 482.4 - PNEUMONIA DUE TO STAPHYLOCOCCUS AUREUS * 482.4 - PNEUMONIA DUE TO STAPHYLOCOCCUS BACTERIA * 482.8 - PNEUMONIA DUE TO OTHER SPECIFIED BACTERIA * 482.8 - PNEUMONIA DUE TO OTHER GRAM-NEGATIVE BACTERIA * 482.8 - PNEUMONIA DUE TO OTHER GRAM-NEGATIVE BACTERIA * 482.8 - PNEUMONIA DUE TO OTHER SPECIFIED BACTERIA * 482.8 - PNEUMONIA DUE TO OTHER SPECIFIED BACTERIA * 482.8 - PNEUMONIA DUE TO OTHER SPECIFIED BACTERIA * 482.8 - PNEUMONIA DUE TO OTHER SPECIFIED BACTERIA * 482.8 - PNEUMONIA DUE TO OTHER SPECIFIED BACTERIA * 482.9 - BACTERIAL PNEUMONIA UNSPECIFIED * 483.1 - PNEUMONIA DUE TO OTHER SPECIFIED BACTERIA | and major bleed exclusion criteria PPV = 85% (Aronsky, et al.; 2005); Note- The corresponding ICD-10 codes will also be used |

| * 507.0 - PNEUMONITIS DUE TO INHALATION OF FOOD OR VOMITUS |
|--------------------------------------------------------------|
| * 507.1 - PNEUMONITIS DUE TO INHALATION OF OILS AND ESSENCES |
| * 507.8 - PNEUMONITIS DUE TO OTHER SOLIDS AND LIQUIDS |

### 6.3.2 Study follow-up

Both as-treated (AT) and intention-to-treat (ITT) analyses will be conducted with treatment defined as the index drug on the day of cohort entry. Because adherence in the real-world databases is expected to be much worse than in the trial, the AT analysis is the **primary** analysis, as it targets the relative hazard of outcomes on treatment.

For the AT analyses, the follow-up will start the day after initiation of prasugrel and comparator and will continue until the earliest date of the following events:

- The first occurrence of the outcome of interest, unless otherwise specified for selected outcomes,
- The date of end of continuous registration in the database,
- End of the study period,
- Measured death event occurs,
- Nursing home admission
  - Nursing home admissions are considered a censoring event because the data sources utilized typically provide little to no data on a patient, particularly on drug utilization, after admission. We will utilize this as an exclusion reason for cohorts for the same reason.
- The date of drug discontinuation, defined as the date of the last continuous treatment episode of the index drug (prasugrel and comparator) plus a defined grace period (i.e., 30 days after the end of the last prescription's days' supply in main analyses).
- The date of augmentation or switching from an exposure to a comparator
- Initiation of ticagrelor

For the ITT analyses, the censoring based on the augmentation/switching and treatment discontinuation will be replaced with a maximum allowed follow-up time of 365 days.

## 7. Initial Feasibility Analysis

### Aetion report links:

Optum: https://bwh-dope.aetion.com/projects/details/989/results/46156/result/0 Marketscan: https://bwh-dope.aetion.com/projects/details/990/results/46157/result/0

Date conducted: December 15, 2019

Complete Aetion feasibility analysis using age, sex, and CCI as the only covariates and the primary endpoint (Section 6.3.1) as the outcome. No measures of association will be computed nor will incidence rates stratified by treatment group.

- Report patient characteristics by treatment group
- Report summary parameters of the overall study population
- Report median follow-up time by treatment group
- Report reasons for censoring in the overall study population

#### 8. Initial Power Assessment

## Aetion report links:

Optum: https://bwh-dope.aetion.com/projects/details/989/results/46159/result/0
Marketscan: https://bwh-dope.aetion.com/projects/details/990/results/46158/result/0

Date conducted: December 15, 2019

In order to complete the initial power analysis, the dummy outcome of a 90-day gap in database enrollment will be used. This outcome is used to ensure that no information on the comparative risks of the outcomes of interest are available at this stage. Complete a 1:1 PS-matched comparative analysis using this outcome. PS should include only 3 covariates: age, sex, and combined comorbidity index. Power calculations are based on the formulas from Chow et al. (2008).

In order to complete the initial power analysis, the dummy outcome of a 90-day gap in database enrollment will be used. This outcome is used to ensure that no information on the comparative risks of the outcomes of interest are available at this stage.

Effectiveness research with Real World Data to support FDA's regulatory decision making: Protocol Template

Complete a 1:1 PS-matched comparative analysis using this outcome. PS should include only 3 covariates: age, sex, and combined comorbidity index. Power calculations are based on the formulas from Chow et al. (2008).

| Reviewed by PI: | Jessica Franklin | Date reviewed: | 12/16/19 |
|-------------------------|------------------|----------------|----------|
| Reviewed by FDA: | David Martin | Date reviewed: | 1/2/20 |
| Reasons for stopping | | | |
| analysis (if required): | | | |

## 9. Balance Assessment after PS matching

## Aetion report links (Prasugrel vs. clopidogrel):

Optum: https://bwh-dope.aetion.com/projects/details/989/results/46940/result/0
Marketscan: https://bwh-dope.aetion.com/projects/details/990/results/46941/result/0

Date conducted: 01/05/2020

After review of initial feasibility and power analyses, complete creation of the remaining covariates (see Table 1 below for list of covariates). Again, using the dummy outcome of a 90-day gap in database enrollment, complete a 1:1 PS-matched analysis. The PS should include the complete list of covariates (excluding laboratory values, which are missing in some patients).

• Provide plot of PS distributions stratified by treatment group.

Note- Please refer to Appendix B.

Report covariate balance after matching.

Note- For Table 1, please refer to Appendix B.

• Report reasons for censoring by treatment group.

| Overall | Referent | Exposure |
|---------|----------|----------|

Effectiveness research with Real World Data to support FDA's regulatory decision making

| Dummy Outcome | 0 (0.00%) | 0 (0.00%) | 0 (0.00%) |
|---|---|---|---|
| Death | 123 (0.28%) | 70 (0.32%) | 53 (0.24%) |
| Start of an additional exposure | 3,840 (8.75%) | 580 (2.64%) | 3,260 (14.86%) |
| End of index exposure | 22,870 (52.14%) | 11,391 (51.94%) | 11,479 (52.34%) |
| Specified date reached | 3,735 (8.51%) | 2,262 (10.31%) | 1,473 (6.72%) |
| End of patient enrollment | 12,361 (28.18%) | 7,033 (32.07%) | 5,328 (24.29%) |
| Switch to ticagrelor (for censoring) + nursing home admission | 935 (2.13%) | 596 (2.72%) | 339 (1.55%) |

• Report follow-up time by treatment group.

| Median Follow-Up Time (Days) [IQR] | | |
|------------------------------------|---------------|---------------|
| Patient Group Optum Marketscan | | |
| Overall Patient Population | 276 [98-453] | 312 [122-481] |
| Referent | 332 [124-532] | 344 [144-530] |
| Exposure | 222 [82-405] | 281 [111-443] |

• Report overall risk of the primary outcome.

| | Optum | Marketscan |
|--------------------------------|-------|------------|
| Risk per 1,000 patients (MACE) | 58.63 | 45.09 |

#### 10. Final Power Assessment

## Date conducted:

- Re-calculate power in the appropriate excel table, using the revised number of matched patients from the PS-match in Section 9. All other parameters in the table should be the same as in Section 8. If the study is to be implemented in more than one database, copy and paste excel sheet to report power for each database separately and for the pooled analysis that uses data from all databases together. Power calculations are based on the formulas from Chow et al. (2008).
  - Pooled
    - For prasugrel 10mg vs. clopidogrel 75mg (Primary outcome- MACE)

| Superiority Analysis | | Non-inferiority Analysis | |
|---|---|---|---|
| Number of patients matched | | Number of patients matched | |
| Reference | 21,932 | Reference | 21,932 |
| Exposed | 21,932 | Exposed | 21,932 |
| Risk per 1,000 patients | 51.86 | Risk per 1,000 patients | 51.86 |
| Desired HR from RCT | 0.8 | Assumed HR from RCT | 1 |
| Alpha (2-sided) | 0.05 | Alpha (2-sided) | 0.05 |
| | | Non-inferiority margin | 1.3 |
| Number of events expected | 2274.78704 | Number of events expected | 2274.78704 |
| Power | 0.999612288 | Power | 0.999991333 |

## o Optum

For prasugrel 10mg vs. clopidogrel 75mg (Primary outcome- MACE)

| Superiority Analysis | | Non-inferiority Analysis | |
|---|---|---|---|
| Number of patients matched | | Number of patients matched | |
| Reference | 6,835 | Reference | 6,835 |
| Exposed | 6,835 | Exposed | 6,835 |
| Risk per 1,000 patients | 58.63 | Risk per 1,000 patients | 58.63 |
| Desired HR from RCT | 0.8 | Assumed HR from RCT | 1 |
| Alpha (2-sided) | 0.05 | Alpha (2-sided) | 0.05 |
| | | Non-inferiority margin | 1.3 |
| Number of events expected | 801.4721 | Number of events expected | 801.4721 |
| Power | 0.884670943 | Power | 0.960270972 |

#### MarketScan

For prasugrel 10mg vs. clopidogrel 75mg (Primary outcome- MACE)

| Tot prasagret total vs. clopidogret 75 mg (1 milary outcome-winee) | | | |
|---|---|---|---|
| Superiority Analysis | | Non-inferiority Analysis | |
| Number of patients matched | | Number of patients matched | |
| Reference | 15,097 | Reference | 15,097 |
| Exposed | 15,097 | Exposed | 15,097 |
| Risk per 1,000 patients | 45.09 | Risk per 1,000 patients | 45.09 |
| Desired HR from RCT | 0.8 | Assumed HR from RCT | 1 |
| Alpha (2-sided) | 0.05 | Alpha (2-sided) | 0.05 |
| | | Non-inferiority margin | 1.3 |
| Number of events expected | 1361.44746 | Number of events expected | 1361.44746 |
| Power | 0.984488939 | Power | 0.998013942 |

• Stop analyses until balance and final power assessment are reviewed by primary investigators, FDA, and assigned members of advisory board. Reviewers evaluate the results of the analyses described above in Sections 9 and 10, including numbers of patients, balance in patient characteristics, follow-up time, and reasons for censoring by treatment group, as well as overall rates of outcomes and study power.

| Reviewed by PI: | Jessica Franklin | Date reviewed: | 12/16/19 |
|-------------------------|------------------|----------------|------------|
| Reviewed by FDA: | David Martin | Date reviewed: | 01/02/2020 |
| Reasons for stopping | | | |
| analysis (if required): | | | |

## 11. Study Confidence and Concerns

### Deadline for voting on study confidence and listing concerns: 1/10/20

- If final feasibility and power analyses are reviewed and approved, proceed to the remaining protocol steps.
- All study team and advisory board members that review this protocol should at this stage provide their level of confidence for the
  success of the RWD study in the <u>Google Form</u>. This form also provides space for reviewers to list any concerns that they feel may
  contribute to a failure to replicate the findings of the RCT, including differences in study populations, poor measurement of study
  variables, or residual confounding. All responses will be kept confidential and individual-level results will only be shared with the
  individual respondent.

## 12. Register study protocol on clinicalTrials.gov

#### Date conducted:

• Register the study on <u>clinicalTrials.gov</u> and upload this document.

### 13. Comparative Analyses

### Aetion report name:

Date conducted:

## 13.1 For primary analysis:

• In the PS-matched cohort from Section 9, calculate the HR for each outcome for prasugrel versus clopidogrel patients using a Cox proportional hazards model.

## 13.2 <u>For secondary analyses:</u>

• In both pre-matched cohorts, perform asymmetrical trimming to remove patients with PS values below the 2.5<sup>th</sup> percentile of treated patients and above the 97.5<sup>th</sup> percentile of untreated patients. In the trimmed cohort, calculate the HR for prasugrel versus referent patients using a Cox proportional hazards model, adjusting for deciles of the PS.

Effectiveness research with Real World Data to support FDA's regulatory decision making

## 14. Requested Results

## 14.1 Results from primary and secondary analyses;

| Analysis | No. exposed events | No. referent events | Exposed rate | Referent rate | HR (95% CI) |
|---|---|---|---|---|---|
| Crude | | | | | |
| Primary analysis | | | | | |
| Analysis 2 | | | | | |
| *** | | | | | |

HR, Hazard Ratio; Cl, Confidence Interval.

#### **15. References**

Aronsky, Dominik, et al. Accuracy of Administrative Data for Identifying Patients with Pneumonia. American Journal of Medical Quality. 2005: 20(6);319–28. doi:10.1177/1062860605280358.

Chow S, Shao J, Wang H. 2008. Sample Size Calculations in Clinical Research. 2nd Ed. Chapman & Hall/CRC Biostatistics Series. page 177

Wiviott et al. Prasugrel versus Clopidogrel in Patients with Acute Coronary Syndromes. N Engl J Med. 2007; 357:2001-15.

| ıs |
|--------------------|
| in claims |
| t for the analysis |

| 3 | For women of childbearing potential only, test negative for pregnancy between ACS presentation and enrollment (based on a<br>urine or serum pregnancy test) and agree to use a reliable method of birth control during the study | N/A<br>(We account for this criteria as an exclusion criteria) | |
|---|---|---|---|
| | EXCLUSION CRITERIA Cardiovascular exclusion criteria | (We docume for all a official as an excitation official) | |
| | Cardiovascular exclusion criteria | Measured during index hospitalization in inpatient setting, any position | |
| 1 | Cardiogenic shock at the time of randomization | Cardiogenic shock:<br>ICD-9: 785.51<br>ICD-10: R57.0 | |
| 2 | Refractory ventricular arrhythmias | Measured 180 days prior to drug initiation in any diagnosis position and inpetient or outpatient setting Ventriouser teachysardia ICD-9: 42-17.2 Ventriouser fibrillistion ICD-9: 42-7.4x ICD-10: 149.0x | |
| 3 | New York Heart Association class IV congestive heart failure | Measured 180 days prior to drug Initiation in any diagnosis position and inpetient or outpatient setting. Heart failure diagnosis: Any of ICD-9 codes: 428x, 398.91, 402.01, 402.11, 402.91, 404.01, 404.11, 404.91, 404.03, 404.13, 404.93 AND Oxygen use: E0425 E0425 E0430 E0431 E0433 E0434 E0435 E0439 E0440 E0441 E0442 E0432 E0444 E047 E1309 E1391 E1392 E1405 E1406 K0738 S\$120 S\$121 ICD-9 V46.2 (Other dependence on machines, supplemental oxygen), ICD-10 299.81 (Dependence on Supplemental oxygen) | |
| | Bleeding risk exclusion criteria | | |
| 4 | Fibrin-specific fibrinolytic therapy less than 24 h before randomization | N/A | |
| 5 | Non-fibrin-specific fibrinolytic therapy less than 48 h before randomization | N/A | |
| 6 | Active internal bleeding or history of bleeding diathesis | Messured 180 days prior to drug initiation in any diagnosis position and inpetient or outpatient setting. For active internal bleeding, refer to the sheet "Bleeding" or Bleeding disthesis: (CD-9: | Cunningham A, Stein CM, Chung CP, Daugherty JR, Smalley WE, Ray WA. An automated database case definition for serious bleeding related to oral anticoagulant use. Pharmacoepidemiol Drug Saf. 2011;20(6):560-566. doi:10.1002/pds.2109 Huybrechts KF, Gogalakrishnan C, Bartels DB, Zint K, Gurusamy WK, Landon J, et al. Safety and effectiveness of dabigatran and other direct oral anticoagulants compared to warfarin in patients with straif libritiation. Clin Pharmacol Ther. 2019 |
| 7 | Clinical findings, in the judgment of the investigator, associated with an increased risk of bleeding | 286.x Coagulation defects 287.x Purpura and other hemorrhagic conditions | Dec 23. |
| | Any of the following: a) History of hemorrhagic streke | Measured any time prior to index hospitalization in any diagnosis position, inpatient or outpatient setting Hemorrhagic stroke: ICD-9: 430 xx, 431.xx ICD-10: I60 xx, 161.xx, | Patorno, Elisabetta et al. 'Cardiovascular outcomes associated with canagliflozin versus other non-giflozin antidiabetic drugs; population based cohort study.' BMJ 2018;360:k119 http://dx.doi.org/10.1136/hmj.k119 Patorno, Elisabetta et al. 'Empagliflozin and the Risk of Heart Failure Hospitalization in Routine Clinical Care: A First Analysis from the Empagliflozin Comparative Effectiveness and Safety (EMPRISE) Study.' Circulation. 2019 Apr 8. doi: 10.1161/CIRCUATIONAHA.118.039117 |
| 8 | b) Intracranial neoplasm, arteriovenous malformation, or aneurysm | Measured 180 days prior to drug initiation in any diagnosis position and inpatient or outpatient setting intraoranial neoplasm (IDO-9: 191x, 255.0, 225.2, 225.4 (IDO-10: C71x, D32x, D33x, AW maiformation (of brain) (IDO-9: 747.81 (IDO-10: C928.2) Corebral Aneuropen (IDO-9: 437.3) (IDO-10: 107.1 | |
| | c) Ischemic stroke within 3 months prior to screening | Measured 90 days prior to Index hospitalization in any position, inpatient setting, isohemic stroke: ICD-9: 433.xx, 434.xx, 436.xx ICD-10: I63.xx I65.xx I66.xx | Patorno, Elisabetta et al. "Cardiovascular outcomes associated with canagliflozin versus other non-giflozin antidiabetic drugs: population based cohort study." BMJ 2018;360:k119 http://dx.doi.org/10.1136/bmj.k119 Patorno, Elisabetta et al. "Empagliflozin and the Risk of Heart Failure Hospitalization in Routine Clinical Care: A First Analysis from the Empagliflozin Comparative Effectiveness and Safety (EMPRISE) Study." Circulation. 2019 Apr 8. doi: 10.1161/circilcul.2110AVAH.2116.039117 |
| 9 | International normalized ratio known to be greater than 1.5 at the time of screening | N/A | |
| 10 | Platelet count of less than 100000/mm3 at the time of screening | Measured during index hospitalization in inpatient setting, any position<br>Thrombocytopenia:<br>ICD-10: D98, D694.x, D69.5x, D69.2x, D69.3x<br>ICD-9: 287.3x, 287.4x | |
| 11 | Anemia (hemoglobin b10 g/dL) at the time of screening | Measured during Index hospitalization in Inpatient setting, any position ICD-9: 280.0 Iron deficiency anemia secondary to blood loss (chronic) 285.1 (Acute posthemorrhagic anemia), 285.9 (Anemia unspecified) | |

| Prior/concomitant therapy exclusion criteria | |
|---|---|
| Prescription for following drugs 5 days prior to index hospitalization One or more doses of a thienopyridine 5 d or less before PCI Clopidogrei, prasugrei, or ticlopidine | |
| 13 Oral anticoagulation or other antiplatelet therapy that cannot be safely discontinued for the duration of the study N/A | |
| More than 150 days of supply out of 180 days prior to drug initiation 14 Daily treatment with nonsteroidal antiinflammatory drugs (NSAIDs) or cyclooxygenase-2 inhibitors (COX-2 inhibitors) NSAID: aspirin, ibuprofen, naproxen >> OTC cannot be captured COX-2 inhibitors: celecoxib | |
| General exclusion criteria | |
| General exclusion criteria 15 Investigative site personnel directly affiliated with the study or immediate family N/A | |
| investigative size personned underly animates with the study of nimerostate raininy investigative size personned underly animates with the study of nimerostate raininy investigative size personned in the study of | |
| Employed by Europeany, one industries Limited, analoms analysis of order of several property of the Limit Study arrounds and the Limit Study arrounds on the Limit Study a | |
| Treatment within the last 30 d with an investigational origing or are presently enrolled in another origing or device study N/A 18 Previously completed or withdrawn from this study or any other study investigating prasugrel N/A | |
| 19 Women who are known to be pregnant, have given by past 90 d. property of the property of th | |
| Gagne, Josh patients between the control of the investigator is associated with reduced survival Following Index score measured 180 days prior to drug initiation 10.1016/j.j. Sun, Jennyl Sun, Jenny | sh J et. al. "A combined comorbidity score predicted mortality in elderly<br>etter than existing scores." J Clin Epidemiol. 2011 Jul;64(7):749-59. doi:<br>j.jclinepi.2010.10.004.<br>W et. al. "Validation of the Combined Comorbidity Index of Charlson and<br>to Predict 30-bay Mortality Across ICD-9 and ICD-10." Med Care. 2018 |
| Seg.56(9):8 Measured 180 days prior to drug initiation in any diagnosis position and inpatient or Patorno, Elic | :812. doi: 10.1097/MLR.000000000000954. |
| 21 Known severe hepatic dysfunction Llwer disease Patorno, Eli (CD-9 diagnosis: 070.x, \$70.xx, \$70.xx, \$70.xx, \$73.xx, \$45.0x, \$45.0x, \$45.0x, \$78.2x, \$78.2x, \$78.9x In Routine C (CD-9 procedure codes: Effectivene | rk119 http://dx.doi.org/10.1136/bmj.k119 Ilisabetta et al. "Empagliflozin and the Risk of Heart Failure Hospitalization Clinical Care: A First Analysis from the Empagliflozin Comparative ess and Safety (EMPRISE) Study." Circulation. 2019 Apr 8. doi: CIRCULATIONAHA.118.039177 |
| 22 Any condition associated with poor treatment compliance including alcoholism, mental illness, or drug dependence Any condition associated with poor treatment compliance including alcoholism, mental illness, or drug dependence Observable (1.09-CM codes: 290.11, 290.3x, 290.41, 291.0x, 292.81, 293.xx; 100.10 Demontal: (1.09-CM codes: 290.xx, 294.1x, 294.8x, 311.19, 331.82; (CD-10-CM codes: 700.7x, 700.7x), 607.0x, 960.0x, 967.xx, 969.4x, 960.6x, 960.7x, 969.4x, 960.6x, 960.7x, | ilisabetta et al. "Cardiovascular outcomes associated with canagliflozin<br>er non-gliflozin antidabetic drugs: population based cohort study." BMJ<br>ktil-19 http://dx.olo.org/10.1138/bmj.kt.19<br>ilisabetta et al. "Empagliflozin and the Risk of Heart Failure Hospitalization<br>Clinical Care: A First Analysis from the Empagliflozin Comparative<br>ess and Safety (EMPRSES) Study." Circulation. 2019 Apr 8. doi:<br>CIRCULATIONAHA.118.039177 |
| 23 Intolerance of or allergy to aspirin, tilopidine, or clopidogrel N/A | |
| 24 May be unable to cooperate with protocol requirements and follow-up procedures N/A | |
| 177 | |

| Trial ID | pNDA14 |
|---|---|
| Trial Name (with web links) | TRITON-TIMI 38 |
| Trial Name (with pdf links) | TRITON-TIMI 38 |
| <u>NCT</u> | NCT00097591 |
| Trial category | Primary indication |
| Run-in period Description | |
| Run-in period? | ? |
| Therapeutic Area | Cardiology/Vascular Diseases |
| Study batch | Antiplatelets |
| RCT Category | 1a-Intended S with label change |
| <b>Brand Name</b> | <u>Efient</u> |
| <b>Generic Name</b> | prasugrel |
| Sponsor | Eli Lilly |
| <u>Year</u> | 2009 |
| | Primary composite endpoint of death from |
| Measurable endpoint | cardiovascular causes, nonfatal myocardial |
| I Wicasarabic Chaponic | infarction, or nonfatal stroke. The key |
| | safety end point was major bleeding. |
| <u>Exposure</u> | Prasugrel |
| <u>Comparator</u> | Clopidogrel |
| | patients with moderate-to-high-risk acute |
| <u>Population</u> | coronary syndromes with scheduled |
| | percutaneous coronary intervention |
| Trial finding | HR = 0.81 (95% CI 0.73–0.90) |
| <u>Notes</u> | |
| No. of Patients | 13,608 |
| Non-inferiority margin | - |
| Assay Sens. Outcome | |
| Assay Sens. Endpoint (from trial) | |
| Finding for potential Assay Sens. | |
| Outcome from trial- | |
| Power | 0.90 to detect 20% reduction in the relative |
| | risk |
| Blinding | Double-blinded |

| Statistical Method | |
|---------------------|---------------------------------------|
| | for the prevention of thrombotic |
| Approval indication | cardiovascular complications in acute |
| | coronary syndromes |

## Mortality-Dependent on data source.

1. All-cause mortality / inpatient mortality Identified using the vital status file-

#### Medicare

Identified using the discharge status codes-

#### Optum-

- 20 = EXPIRED
- 21 = EXPIRED TO BE DEFINED AT STATE LEVEL
- 22 = EXPIRED TO BE DEFINED AT STATE LEVEL
- 23 = EXPIRED TO BE DEFINED AT STATE LEVEL
- 24 = EXPIRED TO BE DEFINED AT STATE LEVEL
- 25 = EXPIRED TO BE DEFINED AT STATE LEVEL
- 26 = EXPIRED TO BE DEFINED AT STATE LEVEL
- 27 = EXPIRED TO BE DEFINED AT STATE LEVEL
- 28 = EXPIRED TO BE DEFINED AT STATE LEVEL
- 29 = EXPIRED TO BE DEFINED AT STATE LEVEL
- 40 = EXPIRED AT HOME (HOSPICE)
- 41 = EXPIRED IN A MEDICAL FACILITY (HOSPICE)
- 42 = EXPIRED PLACE UNKNOWN (HOSPICE)

#### Truven-

- 20 Died
- 22 Died
- 23 Died
- 24 Died
- 25 Died
- 26 Died
- 27 Died
- 28 Died
- 29 Died
- 40 Other died status or Expired at home (Hospice claims only) (depends on year)
- 41 Other died status or Expired in medical facility (Hospice claims only) (depends on year)

- 42 Other died status or Expired place unknown (Hospice claims only) (depends on year)
- 21 Died or Disch./Transf. to court/law enforcement (depends on year)

## 2. CV mortality

Information on CV mortality through data linkage with the National Death Index (NDI) will be available for Medicare at a later date. We will conduct secondary analyses using CV mortality at that time.

| Major bleeding control outcome: 1 inpatient (any position) | |
|---|---|
| Major bleeding exclusion criteria: 1 inpatient (any position) or 2 outpatient diagnosis (separated by 7-365 days) | |
| 562.02 | (ICD9) DIVERTICULOSIS OF SMALL INTESTINE WITH HEMORRHAGE |
| 562.03 | (ICD9) DIVERTICULITIS OF SMALL INTESTINE WITH HEMORRHAGE |
| 562.12 | (ICD9) DIVERTICULOSIS OF COLON WITH HEMORRHAGE |
| 562.13 | (ICD9) DIVERTICULITIS OF COLON WITH HEMORRHAGE |
| 568.81 | (ICD9) HEMOPERITONEUM (NONTRAUMATIC) |
| 569.3 | (ICD9) HEMORRHAGE OF RECTUM AND ANUS |
| 569.83 | (ICD9) PERFORATION OF INTESTINE |
| 569.85 | (ICD9) ANGIODYSPLASIA OF INTESTINE WITH HEMORRHAGE |
| 569.86 | (ICD9) DIEULAFOY LESION (HEMORRHAGIC) OF INTESTINE |
| 578 | (ICD9) HEMATEMESIS |
| 578.9 | (ICD9) HEMORRHAGE OF GASTROINTESTINAL TRACT UNSPECIFIED |
| 423 | (ICD9) HEMOPERICARDIUM |
| 432 | (ICD9) NONTRAUMATIC EXTRADURAL HEMORRHAGE |
| 432.1 | (ICD9) SUBDURAL HEMORRHAGE |
| 432.9 | (ICD9) UNSPECIFIED INTRACRANIAL HEMORRHAGE |
| 459 | (ICD9) HEMORRHAGE UNSPECIFIED |
| 531 | (ICD9) ACUTE GASTRIC ULCER WITH HEMORRHAGE |
| 531 | (ICD9) ACUTE GASTRIC ULCER WITH HEMORRHAGE WITHOUT OBSTRUCTION |
| 531.01 | (ICD9) ACUTE GASTRIC ULCER WITH HEMORRHAGE WITH OBSTRUCTION |
| 531.2 | (ICD9) ACUTE GASTRIC ULCER WITH HEMORRHAGE AND PERFORATION |
| 531.2 | (ICD9) ACUTE GASTRIC ULCER WITH HEMORRHAGE AND PERFORATION WITHOUT OBSTRUCTION |
| 531.21 | (ICD9) ACUTE GASTRIC ULCER WITH HEMORRHAGE AND PERFORATION WITH OBSTRUCTION |
| 531.4 | (ICD9) CHRONIC OR UNSPECIFIED GASTRIC ULCER WITH HEMORRHAGE |
| 531.4 | (ICD9) CHRONIC OR UNSPECIFIED GASTRIC ULCER WITH HEMORRHAGE WITHOUT OBSTRUCTION |
| 531.41 | (ICD9) CHRONIC OR UNSPECIFIED GASTRIC ULCER WITH HEMORRHAGE WITH OBSTRUCTION |
| 531.6 | (ICD9) CHRONIC OR UNSPECIFIED GASTRIC ULCER WITH HEMORRHAGE AND PERFORATION |
| 531.6 | (ICD9) CHRONIC OR UNSPECIFIED GASTRIC ULCER WITH HEMORRHAGE AND PERFORATION WITHOUT OBSTRUCTION |
| 531.61 | (ICD9) CHRONIC OR UNSPECIFIED GASTRIC ULCER WITH HEMORRHAGE AND PERFORATION WITH OBSTRUCTION |

| 532 | (ICD9) ACUTE DUODENAL ULCER WITH HEMORRHAGE |
|---|---|
| 532 | (ICD9) ACUTE DUODENAL ULCER WITH HEMORRHAGE WITHOUT OBSTRUCTION |
| 532.01 | (ICD9) ACUTE DUODENAL ULCER WITH HEMORRHAGE WITH OBSTRUCTION |
| 532.2 | (ICD9) ACUTE DUODENAL ULCER WITH HEMORRHAGE AND PERFORATION |
| 532.2 | (ICD9) ACUTE DUODENAL ULCER WITH HEMORRHAGE AND PERFORATION WITHOUT OBSTRUCTION |
| 532.21 | (ICD9) ACUTE DUODENAL ULCER WITH HEMORRHAGE AND PERFORATION WITH OBSTRUCTION |
| 532.4 | (ICD9) CHRONIC OR UNSPECIFIED DUODENAL ULCER WITH HEMORRHAGE |
| 532.4 | (ICD9) CHRONIC OR UNSPECIFIED DUODENAL ULCER WITH HEMORRHAGE WITHOUT OBSTRUCTION |
| 532.41 | (ICD9) CHRONIC OR UNSPECIFIED DUODENAL ULCER WITH HEMORRHAGE WITH OBSTRUCTION |
| 532.6 | (ICD9) CHRONIC OR UNSPECIFIED DUODENAL ULCER WITH HEMORRHAGE AND PERFORATION |
| 532.6 | (ICD9) CHRONIC OR UNSPECIFIED DUODENAL ULCER WITH HEMORRHAGE AND PERFORATION WITHOUT OBSTRUCTION |
| 532.61 | (ICD9) CHRONIC OR UNSPECIFIED DUODENAL ULCER WITH HEMORRHAGE AND PERFORATION WITH OBSTRUCTION |
| 533 | (ICD9) ACUTE PEPTIC ULCER OF UNSPECIFIED SITE WITH HEMORRHAGE |
| 533 | (ICD9) ACUTE PEPTIC ULCER OF UNSPECIFIED SITE WITH HEMORRHAGE WITHOUT OBSTRUCTION |
| 533.01 | (ICD9) ACUTE PEPTIC ULCER OF UNSPECIFIED SITE WITH HEMORRHAGE WITH OBSTRUCTION |
| 533.2 | (ICD9) ACUTE PEPTIC ULCER OF UNSPECIFIED SITE WITH HEMORRHAGE AND PERFORATION |
| 533.2 | (ICD9) ACUTE PEPTIC ULCER OF UNSPECIFIED SITE WITH HEMORRHAGE AND PERFORATION WITHOUT OBSTRUCTION |
| 533.21 | (ICD9) ACUTE PEPTIC ULCER OF UNSPECIFIED SITE WITH HEMORRHAGE AND PERFORATION WITH OBSTRUCTION |
| 533.4 | (ICD9) CHRONIC OR UNSPECIFIED PEPTIC ULCER OF UNSPECIFIED SITE WITH HEMORRHAGE |
| 533.4 | (ICD9) CHRONIC OR UNSPECIFIED PEPTIC ULCER OF UNSPECIFIED SITE WITH HEMORRHAGE WITHOUT OBSTRUCTION |
| 533.41 | (ICD9) CHRONIC OR UNSPECIFIED PEPTIC ULCER OF UNSPECIFIED SITE WITH HEMORRHAGE WITH OBSTRUCTION |
| 533.6 | (ICD9) CHRONIC OR UNSPECIFIED PEPTIC ULCER OF UNSPECIFIED SITE WITH HEMORRHAGE AND PERFORATION |
| 533.6 | (ICD9) CHRONIC OR UNSPECIFIED PEPTIC ULCER OF UNSPECIFIED SITE WITH HEMORRHAGE AND PERFORATION WITHOUT OBSTRUCTION |
| 533.61 | (ICD9) CHRONIC OR UNSPECIFIED PEPTIC ULCER OF UNSPECIFIED SITE WITH HEMORRHAGE AND PERFORATION WITH OBSTRUCTION |
| 534 | (ICD9) ACUTE GASTROJEJUNAL ULCER WITH HEMORRHAGE |
| 534 | (ICD9) ACUTE GASTROJEJUNAL ULCER WITH HEMORRHAGE WITHOUT OBSTRUCTION |

| 534.01 | (ICD9) ACUTE GASTROJEJUNAL ULCER WITH HEMORRHAGE WITH OBSTRUCTION |
|---|---|
| 534.2 | (ICD9) ACUTE GASTROJEJUNAL ULCER WITH HEMORRHAGE AND PERFORATION |
| 534.2 | (ICD9) ACUTE GASTROJEJUNAL ULCER WITH HEMORRHAGE AND PERFORATION WITHOUT OBSTRUCTION |
| 534.21 | (ICD9) ACUTE GASTROJEJUNAL ULCER WITH HEMORRHAGE AND PERFORATION WITH OBSTRUCTION |
| 534.4 | (ICD9) CHRONIC OR UNSPECIFIED GASTROJEJUNAL ULCER WITH HEMORRHAGE |
| 534.4 | (ICD9) CHRONIC OR UNSPECIFIED GASTROJEJUNAL ULCER WITH HEMORRHAGE WITHOUT OBSTRUCTION |
| 534.41 | (ICD9) CHRONIC OR UNSPECIFIED GASTROJEJUNAL ULCER WITH HEMORRHAGE WITH OBSTRUCTION |
| 534.6 | (ICD9) CHRONIC OR UNSPECIFIED GASTROJEJUNAL ULCER WITH HEMORRHAGE AND PERFORATION |
| 534.6 | (ICD9) CHRONIC OR UNSPECIFIED GASTROJEJUNAL ULCER WITH HEMORRHAGE AND PERFORATION WITHOUT OBSTRUCTION |
| 534.61 | (ICD9) CHRONIC OR UNSPECIFIED GASTROJEJUNAL ULCER WITH HEMORRHAGE AND PERFORATION WITH OBSTRUCTION |
| 578.1 | (ICD9) BLOOD IN STOOL |
| 719.1 | (ICD9) HEMARTHROSIS |
| 719.1 | (ICD9) HEMARTHROSIS SITE UNSPECIFIED |
| 719.11 | (ICD9) HERARTHROSIS INVOLVING SHOULDER REGION |
| 719.12 | (ICD9) HEMARTHORSIS INVOLVING UPPER ARM |
| 719.13 | (ICD9) HEMARTHROSIS INVOLVING FOREARM |
| 719.14 | (ICD9) HEMARTHROSIS INVOLVING HAND |
| 719.15 | (ICD9) HEMARTHROSIS INVOLVING PELVIC REGION AND THIGH |
| 719.16 | (ICD9) HEMARTHROSIS INVOLVING LOWER LEG |
| 719.17 | (ICD9) HEMARTHROSIS INVOLVING ANKLE AND FOOT |
| 719.18 | (ICD9) HEMARTHROSIS INVOLVING OTHER SPECIFIED SITES |
| 719.19 | (ICD9) HEMARTHROSIS INVOLVING MULTIPLE SITES |
| 430 | (ICD9) SUBARACHNOID HEMORRHAGE |
| 431 | (ICD9) INTRACEREBRAL HEMORRHAGE |
| 131.2 | (ICD10) Hemopericardium, not elsewhere classified |
| 160.00 | (ICD10) Nontraumatic subarachnoid hemorrhage from unspecified carotid siphon and bifurcation |
| 160.01 | (ICD10) Nontraumatic subarachnoid hemorrhage from right carotid siphon and bifurcation |
| 160.02 | (ICD10) Nontraumatic subarachnoid hemorrhage from left carotid siphon and bifurcation |
| 160.10 | (ICD10) Nontraumatic subarachnoid hemorrhage from unspecified middle cerebral artery |
| 160.11 | (ICD10) Nontraumatic subarachnoid hemorrhage from right middle cerebral artery |
| 160.12 | (ICD10) Nontraumatic subarachnoid hemorrhage from left middle cerebral artery |

| - | | |
|---|---|---|
| | 160.2 | (ICD10) Nontraumatic subarachnoid hemorrhage from anterior communicating artery |
| | 160.30 | (ICD10) Nontraumatic subarachnoid hemorrhage from unspecified posterior communicating artery |
| | 160.31 | (ICD10) Nontraumatic subarachnoid hemorrhage from right posterior communicating artery |
| | 160.32 | (ICD10) Nontraumatic subarachnoid hemorrhage from left posterior communicating artery |
| | 160.4 | (ICD10) Nontraumatic subarachnoid hemorrhage from basilar artery |
| | 160.50 | (ICD10) Nontraumatic subarachnoid hemorrhage from unspecified vertebral artery |
| | 160.51 | (ICD10) Nontraumatic subarachnoid hemorrhage from right vertebral artery |
| | 160.52 | (ICD10) Nontraumatic subarachnoid hemorrhage from left vertebral artery |
| | 160.6 | (ICD10) Nontraumatic subarachnoid hemorrhage from other intracranial arteries |
| | 160.7 | (ICD10) Nontraumatic subarachnoid hemorrhage from unspecified intracranial artery |
| | 160.8 | (ICD10) Other nontraumatic subarachnoid hemorrhage |
| | 160.9 | (ICD10) Nontraumatic subarachnoid hemorrhage, unspecified |
| | 161.0 | (ICD10) Nontraumatic intracerebral hemorrhage in hemisphere, subcortical |
| | 161.1 | (ICD10) Nontraumatic intracerebral hemorrhage in hemisphere, cortical |
| | 161.2 | (ICD10) Nontraumatic intracerebral hemorrhage in hemisphere, unspecified |
| | 161.3 | (ICD10) Nontraumatic intracerebral hemorrhage in brain stem |
| | 161.4 | (ICD10) Nontraumatic intracerebral hemorrhage in cerebellum |
| | 161.5 | (ICD10) Nontraumatic intracerebral hemorrhage, intraventricular |
| | 161.6 | (ICD10) Nontraumatic intracerebral hemorrhage, multiple localized |
| | 161.8 | (ICD10) Other nontraumatic intracerebral hemorrhage |
| | 161.9 | (ICD10) Nontraumatic intracerebral hemorrhage, unspecified |
| | 162.00 | (ICD10) Nontraumatic subdural hemorrhage, unspecified |
| | 162.01 | (ICD10) Nontraumatic acute subdural hemorrhage |
| | 162.02 | (ICD10) Nontraumatic subacute subdural hemorrhage |
| | 162.03 | (ICD10) Nontraumatic chronic subdural hemorrhage |
| | 162.1 | (ICD10) Nontraumatic extradural hemorrhage |
| | 162.9 | (ICD10) Nontraumatic intracranial hemorrhage, unspecified |
| | K25.0 | (ICD10) Acute gastric ulcer with hemorrhage |
| | K25.2 | (ICD10) Acute gastric ulcer with both hemorrhage and perforation |
| | K25.4 | (ICD10) Chronic or unspecified gastric ulcer with hemorrhage |
| | K25.6 | (ICD10) Chronic or unspecified gastric ulcer with both hemorrhage and perforation |
| | K26.0 | (ICD10) Acute duodenal ulcer with hemorrhage |
| | K26.2 | (ICD10) Acute duodenal ulcer with both hemorrhage and perforation |

| K26.4 | (ICD10) Chronic or unspecified duodenal ulcer with hemorrhage |
|---|---|
| K26.6 | (ICD10) Chronic or unspecified duodenal ulcer with both hemorrhage and perforation |
| K27.0 | (ICD10) Acute peptic ulcer, site unspecified, with hemorrhage |
| K27.2 | (ICD10) Acute peptic ulcer, site unspecified, with both hemorrhage and perforation |
| K27.4 | (ICD10) Chronic or unspecified peptic ulcer, site unspecified, with hemorrhage |
| K27.6 | (ICD10) Chronic or unspecified peptic ulcer, site unspecified, with both hemorrhage and perforation |
| K28.0 | (ICD10) Acute gastrojejunal ulcer with hemorrhage |
| K28.2 | (ICD10) Acute gastrojejunal ulcer with both hemorrhage and perforation |
| K28.4 | (ICD10) Chronic or unspecified gastrojejunal ulcer with hemorrhage |
| K28.6 | (ICD10) Chronic or unspecified gastrojejunal ulcer with both hemorrhage and perforation |
| K55.21 | (ICD10) Angiodysplasia of colon with hemorrhage |
| K56.60 | (ICD10) Unspecified intestinal obstruction |
| K57.01 | (ICD10) Diverticulitis of small intestine with perforation and abscess with bleeding |
| K57.11 | (ICD10) Diverticulosis of small intestine without perforation or abscess with bleeding |
| K57.13 | (ICD10) Diverticulitis of small intestine without perforation or abscess with bleeding |
| K57.21 | (ICD10) Diverticulitis of large intestine with perforation and abscess with bleeding |
| K57.31 | (ICD10) Diverticulosis of large intestine without perforation or abscess with bleeding |
| K57.33 | (ICD10) Diverticulitis of large intestine without perforation or abscess with bleeding |
| K57.41 | (ICD10) Diverticulitis of both small and large intestine with perforation and abscess with bleeding |
| K57.51 | (ICD10) Diverticulosis of both small and large intestine without perforation or abscess with bleeding |
| K57.53 | (ICD10) Diverticulitis of both small and large intestine without perforation or abscess with bleeding |
| K57.81 | (ICD10) Diverticulitis of intestine, part unspecified, with perforation and abscess with bleeding |
| K57.91 | (ICD10) Diverticulosis of intestine, part unspecified, without perforation or abscess with bleeding |
| K57.93 | (ICD10) Diverticulitis of intestine, part unspecified, without perforation or abscess with bleeding |
| K62.5 | (ICD10) Hemorrhage of anus and rectum |
| K63.1 | (ICD10) Perforation of intestine (nontraumatic) |
| K63.81 | (ICD10) Dieulafoy lesion of intestine |
| K66.1 | (ICD10) Hemoperitoneum |
| K92.0 | (ICD10) Hematemesis |
| K92.1 | (ICD10) Melena |
| K92.2 | (ICD10) Gastrointestinal hemorrhage, unspecified |
| M25.00 | (ICD10) Hemarthrosis, unspecified joint |
| M25.011 | (ICD10) Hemarthrosis, right shoulder |

| M25.012 | (ICD10) Hemarthrosis, left shoulder |
|---------|-------------------------------------------------------------|
| M25.019 | (ICD10) Hemarthrosis, unspecified shoulder |
| M25.021 | (ICD10) Hemarthrosis, right elbow |
| M25.022 | (ICD10) Hemarthrosis, left elbow |
| M25.029 | (ICD10) Hemarthrosis, unspecified elbow |
| M25.031 | (ICD10) Hemarthrosis, right wrist |
| M25.032 | (ICD10) Hemarthrosis, left wrist |
| M25.039 | (ICD10) Hemarthrosis, unspecified wrist |
| M25.041 | (ICD10) Hemarthrosis, right hand |
| M25.042 | (ICD10) Hemarthrosis, left hand |
| M25.049 | (ICD10) Hemarthrosis, unspecified hand |
| M25.051 | (ICD10) Hemarthrosis, right hip |
| M25.052 | (ICD10) Hemarthrosis, left hip |
| M25.059 | (ICD10) Hemarthrosis, unspecified hip |
| M25.061 | (ICD10) Hemarthrosis, right knee |
| M25.062 | (ICD10) Hemarthrosis, left knee |
| M25.069 | (ICD10) Hemarthrosis, unspecified knee |
| M25.071 | (ICD10) Hemarthrosis, right ankle |
| M25.072 | (ICD10) Hemarthrosis, left ankle |
| M25.073 | (ICD10) Hemarthrosis, unspecified ankle |
| M25.074 | (ICD10) Hemarthrosis, right foot |
| M25.075 | (ICD10) Hemarthrosis, left foot |
| M25.076 | (ICD10) Hemarthrosis, unspecified foot |
| M25.08 | (ICD10) Hemarthrosis, other specified site |
| R58 | (ICD10) Hemorrhage, not elsewhere classified |
| R04 | (ICD10) Hemorrhage from respiratory passages |
| R04.0 | (ICD10) Epistaxis |
| R04.1 | (ICD10) Hemorrhage from throat |
| R04.2 | (ICD10) Hemoptysis |
| R04.8 | (ICD10) Hemorrhage from other sites in respiratory passages |
| R04.81 | (ICD10) Acute idiopathic pulmonary hemorrhage in infants |
| R04.89 | (ICD10) Hemorrhage from other sites in respiratory passages |
| R04.9 | (ICD10) Hemorrhage from respiratory passages, unspecified |

| R31 | (ICD10) Hematuria |
|---|---|
| R31.0 | (ICD10) Gross hematuria |
| R31.1 | (ICD10) Benign essential microscopic hematuria |
| R31.2 | (ICD10) Other microscopic hematuria |
| R31.21 | |
| R31.29 | |
| R31.9 | (ICD10) Hematuria, unspecified |
| 784.7 | (ICD9) EPISTAXIS |
| 784.8 | (ICD9) HEMORRHAGE FROM THROAT |
| 599.7 | (ICD9) HEMATURIA |
| 599.7 | (ICD9) HEMATURIA UNSPECIFIED |
| 599.71 | (ICD9) GROSS HEMATURIA |
| 599.72 | (ICD9) MICROSCOPIC HEMATURIA |
| 786.3 | (ICD9) HEMOPTYSIS |
| 786.3 | (ICD9) HEMOPTYSIS UNSPECIFIED |
| 786.31 | (ICD9) ACUTE IDIOPATHIC PULMONARY HEMORRHAGE IN INFANTS |
| 786.39 | (ICD9) OTHER HEMOPTYSIS |
| The occurrence | ce of Inpatient with the following attributes: Procedure Code (Any Position) is any of: { "44.43", "43255", "0W3P8ZZ" } |
| 44.43 | (ICD9) ENDOSCOPIC CONTROL OF GASTRIC OR DUODENAL BLEEDING |
| 77.70 | (HCPCS) Esophagogastroduodenoscopy, flexible, transoral; with control of bleeding, any method / Upper |
| 43255 | gastrointestinal endoscopy including esophagus, stomach, and either the duodenum and/or jejunum as |
| 70200 | appropriate; with control of bleeding, any method |
| 0W3P8ZZ | (ICD10) Control Bleeding in Gastrointestinal Tract, Via Natural or Artificial Opening Endoscopic |



The c-statistics for the propensity score model, pre-matching was 0.744. The post-matching c-statistic was 0.538.

The c-statistics for the propensity score model, pre-matching was 0.722. The post-matching c-statistic was 0.528.



Figure 64: Post-matching propensity score overlap



Figure 64: Post-matching propensity score overlap

Table 1: Prasugrel 10 mg vs Clopidogrel 75 mg

| | Unmatched | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|
| | Opt | um | Truven | | | | POO | LED | |
| Variable | Clopidogrel 75mg | Prasugrel 10mg | St. Diff. | Clopidogrel 75mg | Prasugrel 10mg | St. Diff. | Clopidogrel 75mg | Ticagrelor 90mg | St. Diff. |
| Number of patients | 32,556 | 6,872 | | 50,795 | 15,187 | | 83,351 | 22,059 | |
| Age | | | | | | | | | |
| mean (sd) | 65.63 (12.12) | 58.97 (10.27) | 0.59 | 60.92 (11.98) | 56.08 (8.96) | 0.46 | 62.76 (12.03) | 56.98 (9.39) | 0.54 |
| median [IQR] | 67.00 [57.00, 75.00] | 59.00 [52.00, 67.00] | 0.71 | 60.00 [53.00, 68.00] | 57.00 [50.00, 62.00] | 0.28 | 62.73 (12.03) | 57.62 (9.39) | 0.47 |
| Age categories | | | | | | | | | |
| 18 - 54; n (%) | 6,488 (19.9%) | 2,342 (34.1%) | -0.32 | 15,420 (30.4%) | 6,296 (41.5%) | -0.23 | 21,908 (26.3%) | 8,638 (39.2%) | -0.28 |
| 55 - 64; n (%) | 7,900 (24.3%) | 2,300 (33.5%) | -0.20 | 19,596 (38.6%) | 6,745 (44.4%) | -0.12 | 27,496 (33.0%) | 9,045 (41.0%) | -0.17 |
| 65 - 74; n (%) | 9,646 (29.6%) | 1,861 (27.1%) | 0.06 | 7,876 (15.5%) | 1,834 (12.1%) | 0.10 | 17,522 (21.0%) | 3,695 (16.8%) | 0.11 |
| >= 75; n (%) | 8,522 (26.2%) | 369 (5.4%) | 0.59 | 7,903 (15.6%) | 312 (2.1%) | 0.49 | 16,425 (19.7%) | 0,681 (3.1%) | 0.54 |
| Gender-United | | , , | | , , , | , , | | , , , | , , , | |
| Males; n (%) | 21,743 (66.8%) | 5,279 (76.8%) | -0.22 | 36,413 (71.7%) | 12,111 (79.7%) | -0.19 | 58,156 (69.8%) | 17,390 (78.8%) | -0.21 |
| Females; n (%) | 10,813 (33.2%) | 1,593 (23.2%) | 0.22 | 14,382 (28.3%) | 3,076 (20.3%) | 0.19 | 25,195 (30.2%) | 4,669 (21.2%) | 0.21 |
| Region | | , , , | | , , , | , , , | | , , , | , , , | |
| Northeast; n (%) | 3,792 (11.6%) | 520 (7.6%) | 0.14 | 9,397 (18.5%) | 2,412 (15.9%) | 0.07 | 13,189 (15.8%) | 2,932 (13.3%) | 0.07 |
| South; n (%) | 13,415 (41.2%) | 3,530 (51.4%) | -0.21 | 15,086 (29.7%) | 3,797 (25.0%) | 0.11 | 28,501 (34.2%) | 7,327 (33.2%) | 0.02 |
| Midwest; n (%) | 9,686 (29.8%) | 1,655 (24.1%) | 0.13 | 17,860 (35.2%) | 6,576 (43.3%) | -0.17 | 27,546 (33.0%) | 8,231 (37.3%) | -0.09 |
| West; n (%) | 5,663 (17.4%) | 1,167 (17.0%) | 0.01 | 7,896 (15.5%) | 2,181 (14.4%) | 0.03 | 13,559 (16.3%) | 3,348 (15.2%) | 0.03 |
| Unknown+missing; n (%) | N/A | N/A | #VALUE! | 556 (1.1%) | 221 (1.5%) | -0.04 | 556 (0.7%) | 221 (1.0%) | -0.03 |
| CV Covariates | | | | | | | | | |
| Ischemic heart disease; n (%) | 32,556 (100.0%) | 6,872 (100.0%) | #DIV/0! | 50,795 (100.0%) | 15,187 (100.0%) | #DIV/0! | 83,351 (100.0%) | 22,059 (100.0%) | #DIV/0! |
| Acute MI; n (%) | 30,440 (93.5%) | 6,584 (95.8%) | -0.10 | 49,272 (97.0%) | 14,846 (97.8%) | -0.05 | 79712 (95.6%) | 21430 (97.1%) | -0.08 |
| ACS/unstable angina; n (%) | 13,130 (40.3%) | 2,491 (36.2%) | 0.08 | 16,600 (32.7%) | 4,707 (31.0%) | 0.04 | 29730 (35.7%) | 7198 (32.6%) | 0.07 |
| Old MI; n (%) | 4,370 (13.4%) | 739 (10.8%) | 0.08 | 3,850 (7.6%) | 1,014 (6.7%) | 0.03 | 8220 (9.9%) | 1753 (7.9%) | 0.07 |
| Stable angina; n (%) | 6,311 (19.4%) | 1,068 (15.5%) | 0.10 | 5,813 (11.4%) | 1,663 (11.0%) | 0.01 | 12,124 (14.5%) | 2,731 (12.4%) | 0.06 |
| Coronary atherosclerosis and other forms of chronic ischemic heart disease; n (%) | 31,630 (97.2%) | 6,662 (96.9%) | 0.02 | 46,490 (91.5%) | 13,861 (91.3%) | 0.01 | 78,120 (93.7%) | 20,523 (93.0%) | 0.03 |
| Other atherosclerosis with ICD10; n (%) | 560 (1.7%) | 97 (1.4%) | 0.02 | 782 (1.5%) | 157 (1.0%) | 0.05 | 1342 (1.6%) | 254 (1.2%) | 0.03 |
| Previous cardiac procedure (CABG or PTCA or Stent); n (%) | 31,882 (97.9%) | 6,786 (98.7%) | -0.06 | 49,694 (97.8%) | 14,936 (98.3%) | -0.04 | 81576 (97.9%) | 21722 (98.5%) | -0.05 |
| History of CABG or PTCA; n (%) | 9,533 (29.3%) | 1,631 (23.7%) | 0.13 | 7,438 (14.6%) | 1,995 (13.1%) | 0.04 | 16,971 (20.4%) | 3,626 (16.4%) | 0.10 |
| Any stroke; n (%) | 2,400 (7.4%) | 287 (4.2%) | 0.14 | 2,470 (4.9%) | 390 (2.6%) | 0.12 | 4,870 (5.8%) | 0,677 (3.1%) | 0.13 |
| Ischemic stroke (w and w/o mention of cerebral infarction); n (%) | 2,399 (7.4%) | 287 (4.2%) | 0.14 | 2,470 (4.9%) | 390 (2.6%) | 0.12 | 4,869 (5.8%) | 0,677 (3.1%) | 0.13 |
| Hemorrhagic stroke; n (%) | 1 (0.0%) | 0 (0.0%) | #DIV/0! | 1 (0.0%) | 0 (0.0%) | #DIV/0! | 2 (0.0%) | 0 (0.0%) | #DIV/0! |
| TIA; n (%) | 480 (1.5%) | 46 (0.7%) | 0.08 | 523 (1.0%) | 63 (0.4%) | 0.07 | 1003 (1.2%) | 109 (0.5%) | 0.08 |
| Other cerebrovascular disease; n (%) | 450 (1.4%) | 43 (0.6%) | 0.08 | 388 (0.8%) | 46 (0.3%) | 0.07 | 838 (1.0%) | 89 (0.4%) | 0.07 |
| Late effects of cerebrovascular disease; n (%) | 396 (1.2%) | 28 (0.4%) | 0.09 | 291 (0.6%) | 21 (0.1%) | 0.08 | 687 (0.8%) | 49 (0.2%) | 0.09 |
| Cerebrovascular procedure; n (%) | 16 (0.0%) | 1 (0.0%) | #DIV/0! | 34 (0.1%) | 1 (0.0%) | 0.04 | 50 (0.1%) | 2 (0.0%) | 0.04 |
| Heart failure (CHF); n (%) | 6,838 (21.0%) | 941 (13.7%) | 0.19 | 7,137 (14.1%) | 1,632 (10.7%) | 0.10 | 13,975 (16.8%) | 2,573 (11.7%) | 0.15 |
| Peripheral Vascular Disease (PVD) or PVD<br>Surgery ; n (%) | 2,702 (8.3%) | 361 (5.3%) | 0.12 | 2,268 (4.5%) | 413 (2.7%) | 0.10 | 4,970 (6.0%) | 0,774 (3.5%) | 0.12 |

Table 1: Prasugrel 10 mg vs Clopidogrel 75 mg

| Atrial fibrillation; n (%) | 4,283 (13.2%) | 413 (6.0%) | 0.25 | 4,104 (8.1%) | 574 (3.8%) | 0.18 | 8,387 (10.1%) | 0,987 (4.5%) | 0.22 |
|---|---|---|---|---|---|---|---|---|---|
| Other cardiac dysrhythmia; n (%) | 9,981 (30.7%) | 1,632 (23.7%) | 0.16 | 10,768 (21.2%) | 2,653 (17.5%) | 0.09 | 20,749 (24.9%) | 4,285 (19.4%) | 0.13 |
| Cardiac conduction disorders; n (%) | 4,606 (14.1%) | 639 (9.3%) | 0.15 | 4,344 (8.6%) | 958 (6.3%) | 0.09 | 8950 (10.7%) | 1597 (7.2%) | 0.12 |
| Other CVD; n (%) | 11,182 (34.3%) | 1,890 (27.5%) | 0.15 | 12,049 (23.7%) | 3,160 (20.8%) | 0.07 | 23,231 (27.9%) | 5,050 (22.9%) | 0.12 |
| Diabetes-related complications | | | | | | | | | |
| Diabetic retinopathy; n (%) | 742 (2.3%) | 140 (2.0%) | 0.02 | 641 (1.3%) | 152 (1.0%) | 0.03 | 1,383 (1.7%) | 0,292 (1.3%) | 0.03 |
| Diabetes with other ophthalmic | 61 (0.2%) | 6 (0.1%) | 0.03 | 426 (0.8%) | 109 (0.7%) | 0.01 | 0,487 (0.6%) | 0,115 (0.5%) | 0.01 |
| manifestations; n (%) | | | | | | | | | |
| Retinal detachment, vitreous hemorrhage, | 15 (0.0%) | 1 (0.0%) | #DIV/0! | 15 (0.0%) | 4 (0.0%) | #DIV/0! | 30 (0.0%) | 5 (0.0%) | #DIV/0! |
| vitrectomy; n (%) | | | | | | | | | |
| Retinal laser coagulation therapy; n (%) | 63 (0.2%) | 11 (0.2%) | 0.00 | 103 (0.2%) | 28 (0.2%) | 0.00 | 166 (0.2%) | 39 (0.2%) | 0.00 |
| Occurrence of Diabetic Neuropathy; n (%) | 2,028 (6.2%) | 331 (4.8%) | 0.06 | 1,485 (2.9%) | 353 (2.3%) | 0.04 | 3,513 (4.2%) | 0,684 (3.1%) | 0.06 |
| Occurrence of diabetic nephropathy with ICD10 ; n (%) | 1,915 (5.9%) | 238 (3.5%) | 0.11 | 994 (2.0%) | 203 (1.3%) | 0.05 | 2,909 (3.5%) | 0,441 (2.0%) | 0.09 |
| Hypoglycemia; n (%) | 396 (1.2%) | 71 (1.0%) | 0.02 | 608 (1.2%) | 138 (0.9%) | 0.03 | 1,004 (1.2%) | 0,209 (0.9%) | 0.03 |
| Hyperglycemia; n (%) | 2,444 (7.5%) | 521 (7.6%) | 0.00 | 2,152 (4.2%) | 697 (4.6%) | -0.02 | 4,596 (5.5%) | 1,218 (5.5%) | 0.00 |
| Disorders of fluid electrolyte and acid-base balance; n (%) | 4,694 (14.4%) | 808 (11.8%) | 0.08 | 4,163 (8.2%) | 1,078 (7.1%) | 0.04 | 8,857 (10.6%) | 1,886 (8.5%) | 0.07 |
| Diabetic ketoacidosis; n (%) | 127 (0.4%) | 22 (0.3%) | 0.02 | 182 (0.4%) | 53 (0.3%) | 0.02 | 309 (0.4%) | 75 (0.3%) | 0.02 |
| Hyperosmolar hyperglycemic nonketotic syndrome (HONK); n (%) | 81 (0.2%) | 18 (0.3%) | -0.02 | 54 (0.1%) | 14 (0.1%) | 0.00 | 135 (0.2%) | 32 (0.1%) | 0.03 |
| Diabetes with peripheral circulatory | 946 (2.9%) | 101 (1.5%) | 0.10 | 537 (1.1%) | 126 (0.8%) | 0.03 | 1,483 (1.8%) | 0,227 (1.0%) | 0.07 |
| disorders with ICD-10; n (%) | , | . , . , | | , | - ( / | | , , | -, ( , | |
| Diabetic Foot; n (%) | 374 (1.1%) | 54 (0.8%) | 0.03 | 378 (0.7%) | 92 (0.6%) | 0.01 | 752 (0.9%) | 146 (0.7%) | 0.02 |
| Gangrene ; n (%) | 39 (0.1%) | 4 (0.1%) | 0.00 | 30 (0.1%) | 9 (0.1%) | 0.00 | 69 (0.1%) | 13 (0.1%) | 0.00 |
| Lower extremity amputation; n (%) | 145 (0.4%) | 22 (0.3%) | 0.02 | 67 (0.1%) | 23 (0.2%) | -0.03 | 212 (0.3%) | 45 (0.2%) | 0.02 |
| Osteomyelitis; n (%) | 99 (0.3%) | 16 (0.2%) | 0.02 | 110 (0.2%) | 21 (0.1%) | 0.03 | 209 (0.3%) | 37 (0.2%) | 0.02 |
| Skin infections ; n (%) | 1,316 (4.0%) | 240 (3.5%) | 0.03 | 1,628 (3.2%) | 437 (2.9%) | 0.02 | 2,944 (3.5%) | 0,677 (3.1%) | 0.02 |
| Erectile dysfunction; n (%) | 856 (2.6%) | 240 (3.5%) | -0.05 | 1,014 (2.0%) | 329 (2.2%) | -0.01 | 1,870 (2.2%) | 0,569 (2.6%) | -0.03 |
| Diabetes with unspecified complication; n | 759 (2.3%) | 148 (2.2%) | 0.01 | 696 (1.4%) | 246 (1.6%) | -0.02 | 1,455 (1.7%) | 0,394 (1.8%) | -0.01 |
| (%) | , , | . , | | , , | . , | | . , , | . , , | |
| Diabetes mellitus without mention of complications; n (%) | 10,901 (33.5%) | 2,146 (31.2%) | 0.05 | 13,531 (26.6%) | 3,957 (26.1%) | 0.01 | 24,432 (29.3%) | 6,103 (27.7%) | 0.04 |
| Hypertension: 1 inpatient or 2 outpatient claims within 365 days; n (%) | 26,001 (79.9%) | 5,031 (73.2%) | 0.16 | 33,778 (66.5%) | 9,642 (63.5%) | 0.06 | 59,779 (71.7%) | 14,673 (66.5%) | 0.11 |
| Hyperlipidemia ; n (%) | 26,353 (80.9%) | 5,585 (81.3%) | -0.01 | 32,023 (63.0%) | 10,002 (65.9%) | -0.06 | 58,376 (70.0%) | 15,587 (70.7%) | -0.02 |
| Edema; n (%) | 1,711 (5.3%) | 184 (2.7%) | 0.13 | 1,267 (2.5%) | 262 (1.7%) | 0.06 | 2,978 (3.6%) | 0,446 (2.0%) | 0.10 |
| Renal Dysfunction (non-diabetic) ; n (%) | 6,929 (21.3%) | 936 (13.6%) | 0.20 | 5,898 (11.6%) | 1,168 (7.7%) | 0.13 | 12,827 (15.4%) | 2,104 (9.5%) | 0.18 |
| Occurrence of acute renal disease ; n (%) | 2,912 (8.9%) | 403 (5.9%) | 0.11 | 2,293 (4.5%) | 488 (3.2%) | 0.07 | 5205 (6.2%) | 891 (4.0%) | 0.10 |
| Occurrence of chronic renal insufficiency;<br>n (%) | 4,727 (14.5%) | 549 (8.0%) | 0.21 | 3,259 (6.4%) | 558 (3.7%) | 0.12 | 7,986 (9.6%) | 1,107 (5.0%) | 0.18 |
| n (%)<br>Chronic kidney disease ; n (%) | 4,603 (14.1%) | 526 (7.7%) | 0.21 | 3,172 (6.2%) | 537 (3.5%) | 0.13 | 7,775 (9.3%) | 1,063 (4.8%) | 0.18 |
| CKD Stage 3-4; n (%) | 2,896 (8.9%) | 296 (4.3%) | 0.21 | 1,875 (3.7%) | 284 (1.9%) | 0.13 | 4,771 (5.7%) | 0,580 (2.6%) | 0.16 |
| CND 3(age 3-4, 11 (/0) | 2,030 (0.3/0) | 230 (4.370) | 0.15 | 1,013 (3.170) | 204 (1.3/0) | 0.11 | 7,111 (3.1/0) | 0,300 (2.070) | 0.10 |

Table 1: Prasugrel 10 mg vs Clopidogrel 75 mg

| Occurrence of hypertensive nephropathy; n (%) | 3,749 (11.5%) | 412 (6.0%) | 0.20 | 2,431 (4.8%) | 415 (2.7%) | 0.11 | 6180 (7.4%) | 827 (3.7%) | 0.16 |
|---|---|---|---|---|---|---|---|---|---|
| Occurrence of miscellaneous renal | 2,374 (7.3%) | 359 (5.2%) | 0.09 | 1,923 (3.8%) | 418 (2.8%) | 0.06 | 4,297 (5.2%) | 0,777 (3.5%) | 0.08 |
| insufficiency ; n (%)<br>Glaucoma or cataracts ; n (%) | 4,247 (13.0%) | 576 (8.4%) | 0.15 | 4,713 (9.3%) | 902 (5.9%) | 0.13 | 8,960 (10.7%) | 1,478 (6.7%) | 0.14 |
| Cellulitis or abscess of toe; n (%) | 276 (0.8%) | 33 (0.5%) | 0.13 | 173 (0.3%) | 48 (0.3%) | 0.00 | 449 (0.5%) | 81 (0.4%) | 0.14 |
| Foot ulcer; n (%) | 376 (1.2%) | 52 (0.8%) | 0.04 | 379 (0.7%) | 92 (0.6%) | 0.00 | 755 (0.9%) | 144 (0.7%) | 0.01 |
| Bladder stones; n (%) | 57 (0.2%) | 7 (0.1%) | 0.04 | 48 (0.1%) | 8 (0.1%) | 0.00 | 105 (0.1%) | 15 (0.1%) | 0.02 |
| Kidney stones; n (%) | 729 (2.2%) | 143 (2.1%) | 0.03 | 48 (0.1%)<br>857 (1.7%) | 258 (1.7%) | 0.00 | , , | 0,401 (1.8%) | 0.00 |
| Urinary tract infections (UTIs); n (%) | | | 0.01 | | | 0.00 | 1,586 (1.9%) | | 0.01 |
| , , , , , | 2,281 (7.0%) | 303 (4.4%) | 0.11 | 2,080 (4.1%) | 441 (2.9%) | -0.01 | 4,361 (5.2%) | 0,744 (3.4%) | 0.09 |
| Dipstick urinalysis; n (%) | 7,433 (22.8%) | 1,375 (20.0%) | | 10,098 (19.9%) | 3,062 (20.2%) | | 17,531 (21.0%) | 4,437 (20.1%) | |
| Non-dipstick urinalysis; n (%) | 3,761 (11.6%) | 666 (9.7%) | 0.06 | 3,775 (7.4%) | 1,224 (8.1%) | -0.03 | 7,536 (9.0%) | 1,890 (8.6%) | 0.01 |
| Urine function test; n (%) | 682 (2.1%) | 108 (1.6%) | 0.04 | 934 (1.8%) | 189 (1.2%) | 0.05 | 1,616 (1.9%) | 0,297 (1.3%) | 0.05 |
| Cytology; n (%) | 332 (1.0%) | 45 (0.7%) | 0.03 | 497 (1.0%) | 87 (0.6%) | 0.04 | 829 (1.0%) | 132 (0.6%) | 0.04 |
| Cystos; n (%) | 468 (1.4%) | 61 (0.9%) | 0.05 | 640 (1.3%) | 113 (0.7%) | 0.06 | 1108 (1.3%) | 174 (0.8%) | 0.05 |
| Other Covariates | | | | | | | | | |
| Liver disease; n (%) | 11 (0.0%) | 2 (0.0%) | #DIV/0! | 9 (0.0%) | 6 (0.0%) | #DIV/0! | 0,020 (0.0%) | 0,008 (0.0%) | #DIV/0! |
| Osteoarthritis; n (%) | 5,215 (16.0%) | 796 (11.6%) | 0.13 | 4,978 (9.8%) | 1,170 (7.7%) | 0.07 | 10,193 (12.2%) | 1,966 (8.9%) | 0.11 |
| Other arthritis, arthropathies and | 11,251 (34.6%) | 2,072 (30.2%) | 0.09 | 13,878 (27.3%) | 3,718 (24.5%) | 0.06 | 25,129 (30.1%) | 5,790 (26.2%) | 0.09 |
| musculoskeletal pain; n (%) | | | | | | | | | |
| Dorsopathies; n (%) | 7,629 (23.4%) | 1,462 (21.3%) | 0.05 | 9,142 (18.0%) | 2,497 (16.4%) | 0.04 | 16,771 (20.1%) | 3,959 (17.9%) | 0.06 |
| Fractures; n (%) | 758 (2.3%) | 116 (1.7%) | 0.04 | 879 (1.7%) | 209 (1.4%) | 0.02 | 1,637 (2.0%) | 0,325 (1.5%) | 0.04 |
| Falls ; n (%) | 742 (2.3%) | 85 (1.2%) | 0.08 | 316 (0.6%) | 54 (0.4%) | 0.03 | 1058 (1.3%) | 139 (0.6%) | 0.07 |
| Osteoporosis; n (%) | 1,494 (4.6%) | 137 (2.0%) | 0.15 | 1,313 (2.6%) | 149 (1.0%) | 0.12 | 2,807 (3.4%) | 0,286 (1.3%) | 0.14 |
| Hyperthyroidism; n (%) | 181 (0.6%) | 34 (0.5%) | 0.01 | 189 (0.4%) | 37 (0.2%) | 0.04 | 370 (0.4%) | 71 (0.3%) | 0.02 |
| Hypothyroidism ; n (%) | 4,397 (13.5%) | 682 (9.9%) | 0.11 | 4,244 (8.4%) | 992 (6.5%) | 0.07 | 8,641 (10.4%) | 1,674 (7.6%) | 0.10 |
| Other disorders of thyroid gland; n (%) | 750 (2.3%) | 131 (1.9%) | 0.03 | 867 (1.7%) | 225 (1.5%) | 0.02 | 1,617 (1.9%) | 0,356 (1.6%) | 0.02 |
| Depression; n (%) | 3,047 (9.4%) | 634 (9.2%) | 0.01 | 3,332 (6.6%) | 907 (6.0%) | 0.02 | 6,379 (7.7%) | 1,541 (7.0%) | 0.03 |
| Anxiety; n (%) | 3,443 (10.6%) | 720 (10.5%) | 0.00 | 3,184 (6.3%) | 1,000 (6.6%) | -0.01 | 6,627 (8.0%) | 1,720 (7.8%) | 0.01 |
| Sleep_Disorder; n (%) | 2,282 (7.0%) | 594 (8.6%) | -0.06 | 3,772 (7.4%) | 1,215 (8.0%) | -0.02 | 6,054 (7.3%) | 1,809 (8.2%) | -0.03 |
| Dementia; n (%) | 487 (1.5%) | 22 (0.3%) | 0.13 | 413 (0.8%) | 38 (0.3%) | 0.07 | 900 (1.1%) | 60 (0.3%) | 0.10 |
| Delirium; n (%) | 197 (0.6%) | 20 (0.3%) | 0.04 | 147 (0.3%) | 23 (0.2%) | 0.02 | 344 (0.4%) | 43 (0.2%) | 0.04 |
| Psychosis; n (%) | 19 (0.1%) | 2 (0.0%) | 0.04 | 16 (0.0%) | 2 (0.0%) | #DIV/0! | 35 (0.0%) | 4 (0.0%) | #DIV/0! |
| Obesity; n (%) | 6,887 (21.2%) | 1,604 (23.3%) | -0.05 | 7,002 (13.8%) | 2,329 (15.3%) | -0.04 | 13,889 (16.7%) | 3,933 (17.8%) | -0.03 |
| Overweight; n (%) | 1,386 (4.3%) | 255 (3.7%) | 0.03 | 816 (1.6%) | 259 (1.7%) | -0.01 | 2,202 (2.6%) | 0,514 (2.3%) | 0.02 |
| Smoking; n (%) | 14,928 (45.9%) | 3,204 (46.6%) | -0.01 | 15,361 (30.2%) | 4,812 (31.7%) | -0.03 | 30,289 (36.3%) | 8,016 (36.3%) | 0.00 |
| Alcohol abuse or dependence; n (%) | 4 (0.0%) | 0 (0.0%) | #DIV/0! | 504 (1.0%) | 170 (1.1%) | -0.01 | 508 (0.6%) | 170 (0.8%) | -0.02 |
| Drug abuse or dependence; n (%) | 8 (0.0%) | 2 (0.0%) | #DIV/0! | 2 (0.0%) | 0 (0.0%) | #DIV/0! | 10 (0.0%) | 2 (0.0%) | #DIV/0! |
| COPD; n (%) | 5,055 (15.5%) | 674 (9.8%) | 0.17 | 4,803 (9.5%) | 964 (6.3%) | 0.12 | 9,858 (11.8%) | 1,638 (7.4%) | 0.15 |
| Asthma; n (%) | 2,227 (6.8%) | 403 (5.9%) | 0.17 | 2,515 (5.0%) | 621 (4.1%) | 0.12 | 4,742 (5.7%) | | 0.13 |
| * * * | | | | | | | | 1,024 (4.6%) | |
| Obstructive sleep apnea; n (%) | 2,734 (8.4%) | 634 (9.2%) | -0.03 | 3,200 (6.3%) | 1,045 (6.9%) | -0.02 | 5,934 (7.1%) | 1,679 (7.6%) | -0.02 |
| Pneumonia; n (%) | 1,627 (5.0%) | 238 (3.5%) | 0.07 | 1,716 (3.4%) | 358 (2.4%) | 0.06 | 3,343 (4.0%) | 0,596 (2.7%) | 0.07 |
| Imaging; n (%) | 698 (2.1%) | 132 (1.9%) | 0.01 | 4,713 (9.3%) | 133 (0.9%) | 0.39 | 1138 (1.4%) | 265 (1.2%) | 0.02 |
| Other Medications | 47 504 (5 4 50) | 2 742 /54 52/ | 0.01 | 20 474 (50 20) | 0.004 (=0.00) | 0.01 | 47.055 (50.50) | 42.022./52.22** | 0.00 |
| Use of ACE inhibitors; n (%) | 17,584 (54.0%) | 3,742 (54.5%) | -0.01 | 29,471 (58.0%) | 9,091 (59.9%) | -0.04 | 47,055 (56.5%) | 12,833 (58.2%) | -0.03 |
| Use of ARBs; n (%) | 5,799 (17.8%) | 1,182 (17.2%) | 0.02 | 8,108 (16.0%) | 2,346 (15.4%) | 0.02 | 13,907 (16.7%) | 3,528 (16.0%) | 0.02 |
| Use of Loop Diuretics - United; n (%) | 3,974 (12.2%) | 449 (6.5%) | 0.20 | 4,290 (8.4%) | 720 (4.7%) | 0.15 | 8,264 (9.9%) | 1,169 (5.3%) | 0.17 |
| Use of other diuretics- United; n (%) | 1,162 (3.6%) | 249 (3.6%) | 0.00 | 1,686 (3.3%) | 520 (3.4%) | -0.01 | 2,848 (3.4%) | 0,769 (3.5%) | -0.01 |

Table 1: Prasugrel 10 mg vs Clopidogrel 75 mg

| Use of nitrates-United; n (%) | 14,693 (45.1%) | 2,981 (43.4%) | 0.03 | 24,231 (47.7%) | 6,928 (45.6%) | 0.04 | 38,924 (46.7%) | 9,909 (44.9%) | 0.04 |
|---|---|---|---|---|---|---|---|---|---|
| Use of other hypertension drugs; n (%) | 2,065 (6.3%) | 271 (3.9%) | 0.11 | 2,486 (4.9%) | 513 (3.4%) | 0.08 | 4,551 (5.5%) | 0,784 (3.6%) | 0.09 |
| Use of digoxin- United; n (%) | 517 (1.6%) | 49 (0.7%) | 0.08 | 749 (1.5%) | 94 (0.6%) | 0.09 | 1266 (1.5%) | 143 (0.6%) | 0.09 |
| Use of Anti-arrhythmics; n (%) | 897 (2.8%) | 88 (1.3%) | 0.11 | 1,065 (2.1%) | 171 (1.1%) | 0.08 | 1962 (2.4%) | 259 (1.2%) | 0.09 |
| Use of COPD/asthma meds- United; n (%) | 4,160 (12.8%) | 750 (10.9%) | 0.06 | 6,088 (12.0%) | 1,656 (10.9%) | 0.03 | 10,248 (12.3%) | 2,406 (10.9%) | 0.04 |
| Use of statins; n (%) | 29,217 (89.7%) | 6,272 (91.3%) | -0.05 | 45,797 (90.2%) | 13,815 (91.0%) | -0.03 | 75,014 (90.0%) | 20,087 (91.1%) | -0.04 |
| Use of other lipid-lowering drugs; n (%) | 2,494 (7.7%) | 609 (8.9%) | -0.04 | 4,655 (9.2%) | 1,435 (9.4%) | -0.01 | 7,149 (8.6%) | 2,044 (9.3%) | -0.02 |
| Use of oral anticoagulants (Dabigatran,<br>Rivaroxaban, Apixaban, Warfarin); n (%) | 2,662 (8.2%) | 171 (2.5%) | 0.26 | 3,286 (6.5%) | 393 (2.6%) | 0.19 | 5,948 (7.1%) | 0,564 (2.6%) | 0.21 |
| Use of heparin and other low-molecular weight heparins; n (%) | 330 (1.0%) | 29 (0.4%) | 0.07 | 2 (0.0%) | 3 (0.0%) | #DIV/0! | 332 (0.4%) | 32 (0.1%) | 0.06 |
| Use of NSAIDs; n (%) | 4,155 (12.8%) | 898 (13.1%) | -0.01 | 6,384 (12.6%) | 1,965 (12.9%) | -0.01 | 10,539 (12.6%) | 2,863 (13.0%) | -0.01 |
| Use of oral corticosteroids; n (%) | 5,465 (16.8%) | 953 (13.9%) | 0.08 | 7,355 (14.5%) | 2,031 (13.4%) | 0.03 | 12,820 (15.4%) | 2,984 (13.5%) | 0.05 |
| Use of bisphosphonate (United); n (%) | 604 (1.9%) | 58 (0.8%) | 0.10 | 773 (1.5%) | 82 (0.5%) | 0.10 | 1377 (1.7%) | 140 (0.6%) | 0.10 |
| Use of opioids- United; n (%) | 7,601 (23.3%) | 1,567 (22.8%) | 0.01 | 11,530 (22.7%) | 3,264 (21.5%) | 0.03 | 19,131 (23.0%) | 4,831 (21.9%) | 0.03 |
| Use of antidepressants; n (%) | 5,200 (16.0%) | 1,058 (15.4%) | 0.02 | 7,509 (14.8%) | 2,093 (13.8%) | 0.03 | 12,709 (15.2%) | 3,151 (14.3%) | 0.03 |
| Use of antipsychotics; n (%) | 292 (0.9%) | 44 (0.6%) | 0.03 | 396 (0.8%) | 108 (0.7%) | 0.01 | 0,688 (0.8%) | 0,152 (0.7%) | 0.01 |
| Use of anticonvulsants; n (%) | 3,010 (9.2%) | 498 (7.2%) | 0.07 | 3,327 (6.5%) | 789 (5.2%) | 0.06 | 6,337 (7.6%) | 1,287 (5.8%) | 0.07 |
| Use of lithium- United; n (%) | 31 (0.1%) | 7 (0.1%) | 0.00 | 60 (0.1%) | 17 (0.1%) | 0.00 | 91 (0.1%) | 24 (0.1%) | 0.00 |
| Use of Benzos- United; n (%) | 2,919 (9.0%) | 668 (9.7%) | -0.02 | 5,195 (10.2%) | 1,421 (9.4%) | 0.03 | 8,114 (9.7%) | 2,089 (9.5%) | 0.01 |
| Use of anxiolytics/hypnotics- United; n (%) | 1,506 (4.6%) | 352 (5.1%) | -0.02 | 2,651 (5.2%) | 818 (5.4%) | -0.01 | 4,157 (5.0%) | 1,170 (5.3%) | -0.01 |
| Use of dementia meds- United; n (%) | 178 (0.5%) | 14 (0.2%) | 0.05 | 252 (0.5%) | 13 (0.1%) | 0.07 | 430 (0.5%) | 27 (0.1%) | 0.07 |
| Use of antiparkinsonian meds- United; n<br>(%) | 547 (1.7%) | 63 (0.9%) | 0.07 | 652 (1.3%) | 118 (0.8%) | 0.05 | 1,199 (1.4%) | 0,181 (0.8%) | 0.06 |
| Entresto (sacubitril/valsartan); n (%) <b>Labs</b> | 22 (0.1%) | 2 (0.0%) | 0.04 | 3 (0.0%) | 2 (0.0%) | #DIV/0! | 25 (0.0%)<br>0 | 4 (0.0%)<br>0 | #DIV/0! |
| Labs<br>Lab values- HbA1c (%) ; n (%) | 3,678 (11.3%) | 668 (9.7%) | 0.05 | 559 (1.1%) | 130 (0.9%) | 0.02 | 4,237 (5.1%) | 0,798 (3.6%) | 0.07 |
| Lab values-HbA1c (%) (within 3 months); n | 2,396 (7.4%) | 415 (6.0%) | 0.05 | 395 (0.8%) | 79 (0.5%) | 0.02 | 2,791 (3.3%) | 0,494 (2.2%) | 0.07 |
| (%) | 2,330 (7.470) | 413 (0.0%) | 0.00 | 333 (0.8%) | 75 (0.5%) | 0.04 | 2,791 (3.370) | 0,434 (2.270) | 0.07 |
| Lab values- HbA1c (%) (within 6 months) ; n<br>(%) | 3,678 (11.3%) | 668 (9.7%) | 0.05 | 559 (1.1%) | 130 (0.9%) | 0.02 | 4,237 (5.1%) | 0,798 (3.6%) | 0.07 |
| Lab values- BNP; n (%) | 257 (0.8%) | 31 (0.5%) | 0.04 | 41 (0.1%) | 6 (0.0%) | 0.04 | 298 (0.4%) | 37 (0.2%) | 0.04 |
| Lab values- BNP (within 3 months); n (%) | 200 (0.6%) | 26 (0.4%) | 0.03 | 37 (0.1%) | 5 (0.0%) | 0.04 | 237 (0.3%) | 31 (0.1%) | 0.04 |
| Lab values- BNP (within 6 months); n (%) | 257 (0.8%) | 31 (0.5%) | 0.04 | 41 (0.1%) | 6 (0.0%) | 0.04 | 298 (0.4%) | 37 (0.2%) | 0.04 |
| Lab values- BUN (mg/dl); n (%) | 6,259 (19.2%) | 1,248 (18.2%) | 0.03 | 444 (0.9%) | 144 (0.9%) | 0.00 | 6,703 (8.0%) | 1,392 (6.3%) | 0.07 |
| Lab values- BUN (mg/dl) (within 3 months); | 4,032 (12.4%) | 755 (11.0%) | 0.04 | 306 (0.6%) | 95 (0.6%) | 0.00 | 4,338 (5.2%) | 0,850 (3.9%) | 0.06 |
| n (%) | | | | | | | | | |
| Lab values- BUN (mg/dl) (within 6 months);<br>n (%) | 6,259 (19.2%) | 1,248 (18.2%) | 0.03 | 444 (0.9%) | 144 (0.9%) | 0.00 | 6,703 (8.0%) | 1,392 (6.3%) | 0.07 |
| Lab values- Creatinine (mg/dl); n (%) | 6,410 (19.7%) | 1,279 (18.6%) | 0.03 | 467 (0.9%) | 153 (1.0%) | -0.01 | 6,877 (8.3%) | 1,432 (6.5%) | 0.07 |
| Lab values- Creatinine (mg/dl) (within 3 months); n (%) | 4,139 (12.7%) | 775 (11.3%) | 0.04 | 317 (0.6%) | 100 (0.7%) | -0.01 | 4,456 (5.3%) | 0,875 (4.0%) | 0.06 |

Table 1: Prasugrel 10 mg vs Clopidogrel 75 mg

| Lab values- Creatinine (mg/dl) (within 6 months); n (%) | 6,410 (19.7%) | 1,279 (18.6%) | 0.03 | 467 (0.9%) | 153 (1.0%) | -0.01 | 6,877 (8.3%) | 1,432 (6.5%) | 0.07 |
|---|---|---|---|---|---|---|---|---|---|
| Lab values- HDL level (mg/dl); n (%) | 4,980 (15.3%) | 1,064 (15.5%) | -0.01 | 506 (1.0%) | 130 (0.9%) | 0.01 | 5,486 (6.6%) | 1,194 (5.4%) | 0.05 |
| Lab values- HDL level (mg/dl) (within 3 months); n (%) | 3,015 (9.3%) | 623 (9.1%) | 0.01 | 333 (0.7%) | 85 (0.6%) | 0.01 | 3,348 (4.0%) | 0,708 (3.2%) | 0.04 |
| Lab values- HDL level (mg/dl) (within 6 months); n (%) | 4,980 (15.3%) | 1,064 (15.5%) | -0.01 | 506 (1.0%) | 130 (0.9%) | 0.01 | 5,486 (6.6%) | 1,194 (5.4%) | 0.05 |
| Lab values- LDL level (mg/dl); n (%) | 5,080 (15.6%) | 1,074 (15.6%) | 0.00 | 571 (1.1%) | 135 (0.9%) | 0.02 | 5,651 (6.8%) | 1,209 (5.5%) | 0.05 |
| Lab values- LDL level (mg/dl) (within 3 | 3,064 (9.4%) | 626 (9.1%) | 0.01 | 400 (0.8%) | 87 (0.6%) | 0.02 | 3,464 (4.2%) | 0,713 (3.2%) | 0.05 |
| months); n (%) | | ( | | (0.0,1) | J. (3.37.) | | 5, 15 1 (11=11) | 2,1 = (0.=,1) | |
| Lab values- LDL level (mg/dl) (within 6 months); n (%) | 5,080 (15.6%) | 1,074 (15.6%) | 0.00 | 571 (1.1%) | 135 (0.9%) | 0.02 | 5,651 (6.8%) | 1,209 (5.5%) | 0.05 |
| Lab values- NT-proBNP; n (%) | 36 (0.1%) | 7 (0.1%) | 0.00 | 1 (0.0%) | 0 (0.0%) | #DIV/0! | 37 (0.0%) | 7 (0.0%) | #DIV/0! |
| Lab values- NT-proBNP (within 3 months); n (%) | 28 (0.1%) | 6 (0.1%) | 0.00 | 1 (0.0%) | 0 (0.0%) | #DIV/0! | 29 (0.0%) | 6 (0.0%) | #DIV/0! |
| Lab values- NT-proBNP (within 6 months);<br>n (%) | 36 (0.1%) | 7 (0.1%) | 0.00 | 1 (0.0%) | 0 (0.0%) | #DIV/0! | 37 (0.0%) | 7 (0.0%) | #DIV/0! |
| Lab values- Total cholesterol (mg/dl); n (%) | 5,029 (15.4%) | 1,068 (15.5%) | 0.00 | 510 (1.0%) | 131 (0.9%) | 0.01 | 5,539 (6.6%) | 1,199 (5.4%) | 0.05 |
| Lab values-Total cholesterol (mg/dl)<br>(within 3 months); n (%) | 3,031 (9.3%) | 621 (9.0%) | 0.01 | 339 (0.7%) | 85 (0.6%) | 0.01 | 3,370 (4.0%) | 0,706 (3.2%) | 0.04 |
| Lab values- Total cholesterol (mg/dl) | 5,029 (15.4%) | 1,068 (15.5%) | 0.00 | 510 (1.0%) | 131 (0.9%) | 0.01 | 5,539 (6.6%) | 1,199 (5.4%) | 0.05 |
| (within 6 months); n (%) | | , , , | | , , | , , | | | | |
| Lab values-Triglyceride level (mg/dl); n (%) | 4,942 (15.2%) | 1,070 (15.6%) | -0.01 | 497 (1.0%) | 129 (0.8%) | 0.02 | 5,439 (6.5%) | 1,199 (5.4%) | 0.05 |
| Lab values-Triglyceride level (mg/dl)<br>(within 3 months); n (%) | 2,969 (9.1%) | 623 (9.1%) | 0.00 | 325 (0.6%) | 84 (0.6%) | 0.00 | 3,294 (4.0%) | 0,707 (3.2%) | 0.04 |
| Lab values- Triglyceride level (mg/dl)<br>(within 6 months); n (%) | 4,942 (15.2%) | 1,070 (15.6%) | -0.01 | 497 (1.0%) | 129 (0.8%) | 0.02 | 5,439 (6.5%) | 1,199 (5.4%) | 0.05 |
| Lab result number- HbA1c (%) mean (only 2 to 20 included) | 3,659 | 664 | | 434 | 118 | | 0 | 0 | |
| mean (sd) | 7.12 (1.74) | 7.18 (1.76) | -0.03 | 8.08 (1.93) | 8.20 (1.99) | -0.06 | 7.71 (1.86) | 7.88 (1.92) | -0.09 |
| median [IQR] | 6.60 [5.90, 7.80] | 6.60 [5.90, 8.00] | 0.00 | 7.57 [6.70, 9.20] | 7.60 [6.80, 9.42] | -0.02 | 7.19 (1.86) | 7.29 (1.92) | -0.05 |
| Missing; n (%) | 28,897 (88.8%) | 6,208 (90.3%) | -0.05 | 50,361 (99.1%) | 15,069 (99.2%) | -0.01 | 79,258 (95.1%) | 21,277 (96.5%) | -0.07 |
| Lab result number- BNP mean | 257 | 31 | | 41 | 6 | | 0 | 0 | |
| mean (sd) | 286.40 (807.84) | 181.63 (295.19) | 0.17 | 462.66 (983.56) | 98.17 (120.28) | 0.52 | 393.81 (918.93) | 124.17 (192.63) | 0.41 |
| median [IQR] | 100.00 [36.25,<br>242.10] | 66.10 [31.00,<br>164.33] | 0.06 | 159.00 [30.50,<br>397.00] | 55.00 [30.75, 161.50] | 0.15 | 135.96 (918.93) | 58.46 (192.63) | 0.12 |
| Missing; n (%) | 32,299 (99.2%) | 6,841 (99.5%) | -0.04 | 50,754 (99.9%) | 15,181 (100.0%) | -0.04 | 83,053 (99.6%) | 22,022 (99.8%) | -0.04 |
| Lab result number-BUN (mg/dl) mean | 6,259 | 1,248 | | 444 | 144 | | 0 | 0 | |
| mean (sd) | 18.65 (8.48) | 17.48 (7.01) | 0.15 | 333.36 (6,643.25) | 1,684.66 (14,140.00) | -0.12 | 210.44 (5186.05) | 1165.29 (11732.70) | -0.11 |
| median [IQR] | 17.00 [14.00, 21.50] | 16.00 [13.00, 20.00] | 0.13 | 16.00 [13.50, 20.50] | 16.33 [13.00, 21.00] | 0.00 | 16.39 (5186.05) | 16.23 (11732.70) | 0.00 |
| Missing; n (%) | 26,297 (80.8%) | 5,624 (81.8%) | -0.03 | 50,351 (99.1%) | 15,043 (99.1%) | 0.00 | 76,648 (92.0%) | 20,667 (93.7%) | -0.07 |
| Lab result number- Creatinine (mg/dl)<br>mean (only 0.1 to 15 included) | 6,323 | 1,270 | | 426 | 137 | | 0 | 0 | |
| mean (sd) | 1.09 (0.54) | 1.04 (0.43) | 0.10 | 1.04 (0.77) | 1.06 (0.53) | -0.03 | 1.06 (0.69) | 1.05 (0.50) | 0.02 |
| median [IQR] | 0.99 [0.84, 1.18] | 0.98 [0.83, 1.14] | 0.02 | 0.95 [0.82, 1.09] | 1.00 [0.82, 1.19] | -0.08 | 0.97 (0.69) | 0.99 (0.50) | -0.03 |
| - | - | | | | | | | | • |
Table 1: Prasugrel 10 mg vs Clopidogrel 75 mg

| Missing; n (%) | 26,233 (80.6%) | 5,602 (81.5%) | -0.02 | 50,369 (99.2%) | 15,050 (99.1%) | 0.01 | 76,602 (91.9%) | 20,652 (93.6%) | -0.07 |
|---|---|---|---|---|---|---|---|---|---|
| Lab result number- HDL level (mg/dl) mean (only =<5000 included) | 4,980 | 1,064 | | 505 | 128 | | 0 | 0 | |
| mean (sd) | 46.47 (14.25) | 44.40 (12.70) | 0.15 | 40.89 (12.55) | 41.43 (11.97) | -0.04 | 43.07 (13.24) | 42.36 (12.20) | 0.06 |
| median [IQR] | 44.00 [37.00, 54.00] | 43.00 [36.00, 51.00] | 0.07 | 39.50 [34.00, 47.00] | 40.00 [33.00, 47.00] | -0.04 | 41.26 (13.24) | 40.93 (12.20) | 0.03 |
| Missing; n (%) | 27,576 (84.7%) | 5,808 (84.5%) | 0.01 | 50,290 (99.0%) | 15,059 (99.2%) | -0.02 | 77,866 (93.4%) | 20,867 (94.6%) | -0.05 |
| Lab result number- LDL level (mg/dl) mean (only =<5000 included) | 4,959 | 1,056 | | 493 | 120 | | 0 | 0 | |
| mean (sd) | 105.33 (44.86) | 108.39 (47.33) | -0.07 | 97.96 (50.99) | 99.60 (50.63) | -0.03 | 100.84 (48.69) | 102.34 (49.63) | -0.03 |
| median [IQR] | 104.00 [77.00,<br>132.00] | 109.75 [81.00,<br>135.75] | -0.12 | 96.50 [69.00, 129.00] | 100.00 [71.00,<br>135.50] | -0.07 | 99.43 (48.69) | 103.04 (49.63) | -0.07 |
| Missing; n (%) | 27,597 (84.8%) | 5,816 (84.6%) | 0.01 | 50,302 (99.0%) | 15,067 (99.2%) | -0.02 | 77,899 (93.5%) | 20,883 (94.7%) | -0.05 |
| Lab result number-Total cholesterol | 5,021 | 1,066 | | 508 | 129 | | 0 | 0 | |
| (mg/dl) mean (only =<5000 included) | | | | | | | | | |
| mean (sd) | 189.22 (50.40) | 195.25 (47.32) | -0.12 | 188.61 (58.77) | 191.70 (62.84) | -0.05 | 188.85 (55.65) | 192.81 (58.45) | -0.07 |
| median [IQR] | 184.00 [155.50,<br>217.00] | 192.00 [163.38,<br>224.00] | -0.16 | 185.50 [152.00,<br>223.00] | 187.00 [148.50,<br>223.00] | -0.02 | 184.91 (55.65) | 188.56 (58.45) | -0.06 |
| Missing; n (%) | 27,535 (84.6%) | 5,806 (84.5%) | 0.00 | 50,287 (99.0%) | 15,058 (99.2%) | -0.02 | 77,822 (93.4%) | 20,864 (94.6%) | -0.05 |
| Lab result number-Triglyceride level | 4,939 | 1,070 | | 496 | 127 | | 0 | 0 | |
| (mg/dl) mean (only =<5000 included) | | | | | | | | | |
| mean (sd) | 169.72 (134.74) | 186.28 (155.47) | -0.11 | 211.56 (177.58) | 215.24 (191.85) | -0.02 | 195.22 (162.20) | 206.22 (181.30) | -0.06 |
| median [IQR] | 138.50 [99.00,<br>199.00] | 150.00 [106.00,<br>215.25] | -0.08 | 168.00 [116.00,<br>243.12] | 160.50 [110.00,<br>229.00] | 0.04 | 156.48 (162.20) | 157.23 (181.30) | 0.00 |
| Missing; n (%) | 27,617 (84.8%) | 5,802 (84.4%) | 0.01 | 50,299 (99.0%) | 15,060 (99.2%) | -0.02 | 77,916 (93.5%) | 20,862 (94.6%) | -0.05 |
| Lab result number- Hemoglobin mean | 4,722 | 930 | | 321 | 90 | | 0 | 0 | |
| (only >0 included) | | | | | | | | | |
| mean (sd) | 13.97 (1.77) | 14.57 (1.65) | -0.35 | 443.73 (7,701.64) | 14.32 (1.38) | 0.08 | 275.87 (6012.28) | 14.40 (1.47) | 0.06 |
| median [IQR] | 14.10 [12.90, 15.20] | 14.70 [13.60, 15.70] | -0.35 | 13.80 [12.92, 15.20] | 14.43 [13.67, 15.15] | 0.00 | 13.92 (6012.28) | 14.51 (1.47) | 0.00 |
| Missing; n (%) | 27,834 (85.5%) | 5,942 (86.5%) | -0.03 | 50,474 (99.4%) | 15,097 (99.4%) | 0.00 | 78,308 (93.9%) | 21,039 (95.4%) | -0.07 |
| Lab result number- Serum sodium mean (only > 90 and < 190 included) | 6,132 | 1,249 | | 425 | 138 | | 0 | 0 | |
| mean (sd) | 139.85 (2.82) | 139.76 (2.52) | 0.03 | 138.74 (2.71) | 138.76 (2.93) | -0.01 | 139.17 (2.75) | 139.07 (2.81) | 0.04 |
| median [IQR] | 140.00 [138.00,<br>142.00] | 140.00 [138.00,<br>141.00] | 0.00 | 139.00 [137.00,<br>140.50] | 139.00 [137.00,<br>141.00] | 0.00 | 139.39 (2.75) | 139.31 (2.81) | 0.03 |
| Missing; n (%) | 26,424 (81.2%) | 5,623 (81.8%) | -0.02 | 50,370 (99.2%) | 15,049 (99.1%) | 0.01 | 76,794 (92.1%) | 20,672 (93.7%) | -0.06 |
| Lab result number- Albumin mean (only >0 and <=10 included) | 5,624 | 1,178 | | 360 | 115 | | 0 | 0 | |
| mean (sd) | 4.20 (0.34) | 4.29 (0.32) | -0.27 | 4.07 (0.63) | 4.13 (0.53) | -0.10 | 4.12 (0.54) | 4.18 (0.47) | -0.12 |
| median [IQR] | 4.20 [4.00, 4.40] | 4.30 [4.10, 4.50] | -0.30 | 4.15 [4.00, 4.40] | 4.20 [4.00, 4.40] | -0.09 | 4.17 (0.54) | 4.23 (0.47) | -0.12 |
| Missing; n (%) | 26,932 (82.7%) | 5,694 (82.9%) | -0.01 | 50,435 (99.3%) | 15,072 (99.2%) | 0.01 | 77,367 (92.8%) | 20,766 (94.1%) | -0.05 |
| Lab result number- Glucose (fasting or random) mean (only 10-1000 included) | 6,067 | 1,242 | | 408 | 132 | | 0 | 0 | |
| mean (sd) | 124.84 (56.69) | 120.87 (51.78) | 0.07 | 168.32 (67.53) | 165.62 (78.32) | 0.04 | 151.34 (63.52) | 151.68 (71.12) | -0.01 |
| median [IQR] | 105.00 [93.00,<br>135.00] | 103.00 [92.50,<br>130.00] | 0.04 | 149.00 [119.00,<br>202.50] | 143.90 [111.00,<br>189.50] | 0.07 | 131.81 (63.52) | 131.16 (71.12) | 0.01 |

Table 1: Prasugrel 10 mg vs Clopidogrel 75 mg

| Lab result number Protassium mean (only 1.277 1.377 1.317 0.00 0.0 | Missing; n (%) | 26,489 (81.4%) | 5,630 (81.9%) | -0.01 | 50,387 (99.2%) | 15,055 (99.1%) | 0.01 | 76,876 (92.2%) | 20,685 (93.8%) | -0.06 |
|---|---|---|---|---|---|---|---|---|---|---|
| mean bod | Lab result number-Potassium mean (only | 6,316 | 1,277 | | 437 | 141 | | 0 | 0 | |
| medin (IQR) | 1-7 included) | | | | | | | | | |
| Missing, n (N) | mean (sd) | 4.39 (0.45) | 4.40 (0.42) | -0.02 | 4.30 (0.46) | 4.32 (0.47) | -0.04 | 4.34 (0.46) | 4.34 (0.46) | 0.00 |
| Combridity Scores CLIBAD days-1009 and ICD10 CLIBAD days-1009 and IC | median [IQR] | 4.40 [4.10, 4.66] | 4.40 [4.10, 4.70] | 0.00 | 4.30 [4.00, 4.60] | 4.30 [4.00, 4.65] | 0.00 | 4.34 (0.46) | 4.33 (0.46) | 0.02 |
| CCC 150 days -1CD9 and ICD10 median (DR) 2.89 (2.14) 2.20 (1.02) 0.35 1.95 (1.72) 1.61 (1.42) 0.22 2.32 (1.90) 1.79 (1.56) 0.05 | Missing; n (%) | 26,240 (80.6%) | 5,595 (81.4%) | -0.02 | 50,358 (99.1%) | 15,046 (99.1%) | 0.00 | 76,598 (91.9%) | 20,641 (93.6%) | -0.07 |
| mean [sd] | Comorbidity Scores | | | | | | | | | |
| median | CCI (180 days)- ICD9 and ICD10 | | | | | | | | | |
| Frailty Score (mean): Empirical Version 365 daysmean (sb) | mean (sd) | 2.89 (2.14) | 2.20 (1.82) | 0.35 | 1.95 (1.72) | 1.61 (1.42) | 0.22 | 2.32 (1.90) | 1.79 (1.56) | 0.30 |
| Frailty Score (mean): Empirical Version 365 daysmean (sb) | median [IQR] | 2.00 [1.00, 4.00] | 2.00 [1.00, 3.00] | 0.00 | 1.00 [1.00, 3.00] | 1.00 [1.00, 2.00] | 0.00 | 1.39 (1.90) | 1.31 (1.56) | 0.05 |
| mean (s) | Frailty Score (mean): Empirical Version 365 | | | | | | | | | |
| median IOR | days, | | | | | | | | | |
| Healthcare Utilization Any hospitalization; n (%) Any hospitalization; n (%) Any hospitalization; n (%) Any hospitalization during prior 21-180 days; n (%) Endocrinologist Visit; n (%) Endoc | mean (sd) | 0.19 (0.05) | 0.17 (0.04) | 0.44 | 0.17 (0.04) | 0.16 (0.03) | 0.28 | 0.18 (0.04) | 0.16 (0.03) | 0.57 |
| Any hospitalization; n (%) Any hospitalization; n (%) Any hospitalization; n (%) Any hospitalization during prior 31-180 days, n (%) Endocrinologist Visit; n (%) Endocrinologist Visit; n (%) Endocrinologist Visit; n (%) Endocrinologist Visit; n (%) Endocrinologist Visit; d (31 days prior); n (%) Endocrinologist Visit; d (31 days prior); n (%) Endocrinologist Visit; d (31 days prior); n (%) Endocrinologist Visit; d (31 days prior); n (%) Endocrinologist Visit; d (31 days prior); n (%) Internal medicine/family medicine visits; n (%) Internal medicin | median [IQR] | 0.18 [0.16, 0.21] | 0.17 [0.15, 0.19] | 0.22 | 0.17 [0.15, 0.19] | 0.16 [0.14, 0.18] | 0.28 | 0.17 (0.04) | 0.16 (0.03) | 0.28 |
| Any hospitalization during prior 31-180 days; n (%) | Healthcare Utilization | | | | | | | | | |
| days, n (%) Endocrinologist Visit; n (%) Endocrinologist Visit; n (%) Endocrinologist Visit; n (%) Endocrinologist Visit; n (%) Endocrinologist Visit; (30 days prior); n (%) Endocrinologist Visit; (31 to 180 days Prior); n (%) Endocrinologist Visit; (31 to 180 days Prior); n (%) Endocrinologist Visit; (31 to 180 days Prior); n (%) Internal medicine/family medicinevisits; n (%) Internal medicine/family medicinevisits; n (%) Internal medicine/family medicinevisits; n (%) Internal medicine/family medicinevisits (30 days prior); n (%) Internal medicine/family medicinevisits (31 to 180 days Prior); n (%) Internal medicine/family medicinevisits | Any hospitalization; n (%) | 32,547 (100.0%) | 6,871 (100.0%) | #DIV/0! | 50,794 (100.0%) | 15,186 (100.0%) | #DIV/0! | 83,341 (100.0%) | 22,057 (100.0%) | #DIV/0! |
| Endocrinologist Visit; (1) (8) (8) (1,241 (4,1%) 327 (4,8%) -0.03 1,666 (3,3%) 558 (3,7%) -0.02 3,007 (3,6%) 0,885 (4,0%) -0.02 Endocrinologist Visit; (31 to 180 days prior); n (%) (85 (2,6%) 194 (2,8%) -0.01 1,002 (2,0%) 339 (2,2%) -0.01 1,854 (2,2%) 0,533 (2,4%) -0.01 prior); n (%) (8) (10 ternal medicine/family medicine visits; n (%) (8) (11 ternal medicine/family medicine visits; n (%) (11 ternal medicine/family medicine visits; n (%) (12 1,000 (2,0%) 1,000 (2,0%) (1,0%) (1,0% | Any hospitalization during prior 31-180 | 1,329 (4.1%) | 212 (3.1%) | 0.05 | 1,545 (3.0%) | 367 (2.4%) | 0.04 | 2,874 (3.4%) | 0,579 (2.6%) | 0.05 |
| Endocrinologist Visit (30 days prior); n (%) Endocrinologist Visit (31 to 180 days prior); n (%) Endocrinologist Visit (31 to 180 days prior); n (%) Internal medicine/family medicine visits; n (%) Internal medicine/family medicine visits (30 days prior); n (%) Internal medicine/family medicine visits (30 days prior); n (%) Internal medicine/family medicine visits (31 to 180 days prior); n (%) Internal medicine/family medicine visits (30 days prior); n (%) Internal medicine/fa | days; n (%) | | | | | | | | | |
| Endocrinologist Visit (31 to 180 days prior); n (%) Internal medicine/family medicine visits; n (%) Internal medicine/family medicine visits; n (%) Internal medicine/family medicine visits; n (%) Internal medicine/family medicine visits; 21,362 (65.6%) 3,940 (57.3%) 0.17 20,203 (39.8%) 5,719 (37.7%) 0.04 41,565 (49.9%) 9,659 (43.8%) 0.12 (30 days prior); n (%) Internal medicine/family medicine visits (30 days prior); n (%) Internal medicine/family medicine visits (31 to 180 days | Endocrinologist Visit; n (%) | 1,341 (4.1%) | 327 (4.8%) | -0.03 | 1,666 (3.3%) | 558 (3.7%) | -0.02 | 3,007 (3.6%) | 0,885 (4.0%) | -0.02 |
| Endocrinologist Visit (31 to 180 days prior); n (%) Internal medicine/family medicine visits; n (%) Internal medicine/family medicine visits; n (%) Internal medicine/family medicine visits; n (%) Internal medicine/family medicine visits; 21,362 (65.6%) 3,940 (57.3%) 0.17 20,203 (39.8%) 5,719 (37.7%) 0.04 41,565 (49.9%) 9,659 (43.8%) 0.12 (30 days prior); n (%) Internal medicine/family medicine visits (30 days prior); n (%) Internal medicine/family medicine visits (31 to 180 days | Endocrinologist Visit (30 days prior); n (%) | 689 (2.1%) | 175 (2.5%) | -0.03 | 891 (1.8%) | 317 (2.1%) | -0.02 | 1,580 (1.9%) | 0,492 (2.2%) | -0.02 |
| prior); n (%) Internal medicine/family medicine visits; n (%) (%) Internal medicine/family medicine visits (30 days prior); n (%) Internal medicine/family medicine visits (31 to 180 days prior); n (%) Number of Cardiologist visits (31 to 180 days prior); n (%) Electrocardiogram; n (%) Electrocardiogr | | | | | | | | | | |
| Internal medicine/family medicine visits; n (%) | Endocrinologist Visit (31 to 180 days | 852 (2.6%) | 194 (2.8%) | -0.01 | 1,002 (2.0%) | 339 (2.2%) | -0.01 | 1,854 (2.2%) | 0,533 (2.4%) | -0.01 |
| (%) Internal medicine/family medicine visits (30 days prior); n (%) Internal medicine/family medicine visits (31 to 180 days prior); n (%) Internal medicine/family medicine visits (31 to 180 days prior); n (%) Internal medicine/family medicine visits (30 days prior); n (%) Internal medicine/family medicine visits (31 to 180 days prior); n (%) Internal medicine/family medicine visits (30 days prior); n (%) Internal medicine/family medicine visits (30 days (31 to 180 days prior); n (%) Internal medicine/family medicine visits (31 to 180 days prior); n (%) Internal prior, n (%) Internal prior, n (%) Internal prior, n (%) Internal prior, n (%) Inte | prior); n (%) | | | | | | | | | |
| Internal medicine/family medicine visits (30 days prior); n (%) | Internal medicine/family medicine visits; n | 25,743 (79.1%) | 4,863 (70.8%) | 0.19 | 32,636 (64.3%) | 9,499 (62.5%) | 0.04 | 58,379 (70.0%) | 14,362 (65.1%) | 0.10 |
| (30 days prior); n (%) Internal medicine/family medicine visits (31 to 180 days prior); n (%) Cardiologist visit; n (%) Cardiologist visit; n (%) Sumber of Cardiologist visits (30 days prior); n (%) Number of Cardiologist visits (30 days prior); n (%) Number of Cardiologist visits (31 to 180 days prior); n (%) Number of Cardiologist visits (31 to 180 days prior); n (%) Number of Cardiologist visits (31 to 180 days prior); n (%) Electrocardiogram; n (%) Use of glucose test strips; n (%) Dialysis; n (%) 164 (0.5%) 27 (0.4%) 0.01 188 (0.44) 0.02 188 (0.44) 0.03 188 (0.44) 0.05 188 (0.44) 0.06 188 (0.42) 0.64 188 (0.44) 0.11 0.12 0.14 0.15 0.15 0.16 0.15 0.16 0.16 0.17 0.16 0.17 0.18 0.19 0.10 0.10 0.10 0.10 0.10 0.10 0.10 | (%) | | | | | | | | | |
| Internal medicine/family medicine visits (31 to 180 days prior); n (%) Cardiologist visit; n (%) Cardiologist visits; n (%) Cardiologist visits; n (%) Number of Cardiologist visits (30 days prior); n (%) Number of Cardiologist visits (30 days prior); n (%) Number of Cardiologist visits (30 days prior); n (%) Number of Cardiologist visits (30 days prior); n (%) Number of Cardiologist visits (31 to 180 days prior); n (%) Number of Cardiologist visits (31 to 180 days prior); n (%) Electrocardiogram; n (%) Electrocardiogram; n (%) Use of glucose test strips; n (%) Dialysis; n (%) 164 (0.5%) 27 (0.4%) Number of Hospitalizations median [IQR] Number of Hospitalidays median [IQR] Number of hospital days mean (sd) 4.12 (3.05) 3.71 (2.07) 3.05 (44.4%) 0.21 26,087 (51.4%) 7,448 (49.0%) 7,448 (49.0%) 7,448 (49.0%) 0.03 47,448 (49.0%) 0.05 43,967 (52.7%) 10,498 (47.6%) 0.10 43,967 (52.7%) 10,498 (47.6%) 0.11 17,435 (34.3%) 5,005 (33.0%) 0.03 48,741 (58.5%) 11,628 (52.7%) 0.12 Number (Cardiologist visits (30 days 31,169 (95.7%) 6,604 (96.1%) -0.02 14,457 (28.5%) 4,266 (28.1%) 0.01 45,626 (54.7%) 10,870 (49.3%) 0.11 10,628 (52.7%) 0.12 11,628 (52.7%) 0.12 11,628 (52.7%) 0.12 11,628 (52.7%) 0.13 11,628 (52.7%) 0.14 10,628 (64.4.7%) 11,628 (52.7%) 0.12 Nam(6.6.8.1) 11,628 (52.7%) 0.12 11,628 (52.7%) 0.12 11,628 (52.7%) 0.13 11,628 (52.7%) 0.14 10,628 (64.4.7%) 11,628 (52.7%) 0.12 11,628 (52.7%) 0.12 11,628 (52.7%) 0.11 10,628 (52.7%) 11,628 (52.7%) 11 | Internal medicine/family medicine visits | 21,362 (65.6%) | 3,940 (57.3%) | 0.17 | 20,203 (39.8%) | 5,719 (37.7%) | 0.04 | 41,565 (49.9%) | 9,659 (43.8%) | 0.12 |
| (31 to 180 days prior); n (%) Cardiologist visit; n (%) Number of Cardiologist visits; (30 days prior); n (%) Number of Cardiologist visits (31 to 180 days prior); n (%) Number of Cardiologist visits (31 to 180 days prior); n (%) Number of Cardiologist visits (31 to 180 days prior); n (%) Number of Cardiologist visits (31 to 180 days prior); n (%) Electrocardiogram; n (%) Luse of glucose test strips; n (%) Dialysis; n (%) 1040 (1.3%) 1050 (1.0%) 1060 (1.5%) 1070 (1.0%) 1060 (1.0%) 1070 (1.0%) | (30 days prior) ; n (%) | | | | | | | | | |
| Cardiologist visit; n (%) Number of Cardiologist visits (30 days prior); n (%) Relectrocardiogram; n (%) 10,299 (93.1%) 10,349 (95.7%) 10,341 (92.3%) 11,435 (34.3%) 11,435 (34.3%) 11,436 (28.1%) 11,436 (28.1%) 11,436 (42.1%) 11,439 (14.0%) 2,232 (10.1%) 11,639 (14.0%) 2,331 (14.0%) 2,331 (10.1%) 11,639 (14.0%) 2,331 (10.1%) 11,639 (14.0%) 2,332 (10.1%) 11,639 (14.0%) 2,331 (10.1%) 3,34 | • | 17,880 (54.9%) | 3,050 (44.4%) | 0.21 | 26,087 (51.4%) | 7,448 (49.0%) | 0.05 | 43,967 (52.7%) | 10,498 (47.6%) | 0.10 |
| Number of Cardiologist visits (30 days prior); n (%) Number of Cardiologist visits (31 to 180 days prior); n (%) Electrocardiogram; n (%) Use of glucose test strips; n (%) Independent of Cardiologist visits (31 to 180 days prior); n (%) Electrocardiogram; n (%) Use of glucose test strips; n (%) Independent of Cardiologist visits (31 to 180 days prior); n (%) Electrocardiogram; n (%) Use of glucose test strips; n (%) Independent of Cardiologist visits (31 to 180 days prior); n (%) Electrocardiogram; n (%) Use of glucose test strips; n (%) Independent of Cardiologist visits (31 to 180 days prior); n (%) Electrocardiogram; n (%) Use of glucose test strips; n (%) Independent of Cardiologist visits (31 to 180 days prior); n (%) Independent of Cardiologist visits (31 to 180 days prior); n (%) Electrocardiogram; n (%) Independent of Cardiologist visits (31 to 180 days prior); n (%) Independent of Cardiologist visits (10 days prior); n (%) Independent of Cardiolo | (31 to 180 days prior) ; n (%) | | | | | | | | | |
| prior); n (%) Number of Cardiologist visits (31 to 180 days prior); n (%) Electrocardiogram; n (%) Use of glucose test strips; n (%) Use of glucose test strips; n (%) 164 (0.5%) 170 (1.0%) 188 (0.4%) 191 (13.4%) 10.11 10.12 10.12 10.12 10.13 10.14 10.15 10 | | 31,306 (96.2%) | 6,623 (96.4%) | | 17,435 (34.3%) | 5,005 (33.0%) | | 48,741 (58.5%) | 11,628 (52.7%) | 0.12 |
| Number of Cardiologist visits (31 to 180 days prior); n (%) Electrocardiogram; n (%) Use of glucose test strips; n (%) Dialysis; n (%) mean (sd)median [IQR]median [IQR]median [IQR]median [IQR]median [IQR]median [IQR]medisd)mean (sd)median [IQR]median [IQR]median [IQR]mean (sd)median [IQR]median [IQR] | | 31,169 (95.7%) | 6,604 (96.1%) | -0.02 | 14,457 (28.5%) | 4,266 (28.1%) | 0.01 | 45,626 (54.7%) | 10,870 (49.3%) | 0.11 |
| days prior); n (%) Electrocardiogram; n (%) Electrocardiogram; n (%) Use of glucose test strips; n (%) Dialysis; n (%) Index (0.5%) Add (0.10%) Add (0.10% | | | | | | | | | | |
| Electrocardiogram; n (%) 30,299 (93.1%) 6,341 (92.3%) 0.03 29,074 (57.2%) 8,281 (54.5%) 0.05 59,373 (71.2%) 14,622 (66.3%) 0.11 Use of glucose test strips; n (%) 420 (1.3%) 70 (1.0%) 0.03 477 (0.9%) 157 (1.0%) -0.01 0,897 (1.1%) 0,227 (1.0%) 0.01 Dialysis; n (%) 164 (0.5%) 27 (0.4%) 0.01 188 (0.4%) 20 (0.1%) 0.06 352 (0.4%) 47 (0.2%) 0.04 number of different/distinct medication prescriptionsmean (sd) 9.12 (4.59) 8.43 (4.41) 0.15 8.69 (4.31) 8.22 (4.10) 0.11 8.86 (4.42) 8.29 (4.20) 0.13median [IQR] 8.00 [6.00, 12.00] 7.00 [5.00, 11.00] 0.22 8.00 [5.00, 11.00] 7.00 [5.00, 10.00] 0.24 8.00 (4.42) 7.00 (4.20) 0.23 Number of Hospitalizationsmean (sd) 1.12 (0.38) 1.09 (0.31) 0.09 1.10 (0.33) 1.07 (0.28) 0.10 1.11 (0.35) 1.08 (0.29) 0.09median [IQR] 1.00 [1.00, 1.00] 1.00 [1.00, 1.00] 0.00 1.00 [1.00, 1.00] 0.00 1.00 (0.35) 1.00 (0.29) 0.00 Number of hospital daysmean (sd) 4.12 (3.05) 3.71 (2.07) 0.16 3.87 (2.26) 3.60 (1.70) 0.14 3.97 (2.60) 3.63 (1.82) 0.15 | | 5,961 (18.3%) | 919 (13.4%) | 0.13 | 5,678 (11.2%) | 1,313 (8.6%) | 0.09 | 11,639 (14.0%) | 2,232 (10.1%) | 0.12 |
| Use of glucose test strips; n (%) Dialysis; n (%) Index (0.5%) Dialysis; n | | | | | | | | | | |
| Dialysis; n (%) number of different/distinct medication prescriptionsmean (sd)median [IQR] Number of Hospitalizationsmean (sd)mean (sd)mean (sd)mean (sd)mean (sd)median [IQR] Number of Hospitalizationsmean (sd)mean (sd)mean (sd)mean (sd)mean (sd)mean (sd)median [IQR]mean (sd)mean (sd) | • • • • | ' ' | | | . , , | . , , | | . , , | . , , | |
| number of different/distinct medication prescriptions 9.12 (4.59) 8.43 (4.41) 0.15 8.69 (4.31) 8.22 (4.10) 0.11 8.86 (4.42) 8.29 (4.20) 0.13 median [IQR] 8.00 [6.00, 12.00] 7.00 [5.00, 11.00] 0.22 8.00 [5.00, 11.00] 7.00 [5.00, 10.00] 0.24 8.00 (4.42) 7.00 (4.20) 0.23 Number of Hospitalizations mean (sd) 1.12 (0.38) 1.09 (0.31) 0.09 1.10 (0.33) 1.07 (0.28) 0.10 1.11 (0.35) 1.08 (0.29) 0.09 median [IQR] 1.00 [1.00, 1.00] 1.00 [1.00, 1.00] 1.00 [1.00, 1.00] 0.00 1.00 [1.00, 1.00] 0.00 1.00 [0.00, 1.00] 0.00 1.00 (0.35) 1.00 (0.29) 0.00 Number of hospital days mean (sd) 4.12 (3.05) 3.71 (2.07) 0.16 3.87 (2.26) 3.60 (1.70) 0.14 3.97 (2.60) 3.63 (1.82) 0.15 | | ` ' | , , | | , , | , , | | | | |
| prescriptionsmean (sd)median [IQR]median [IQR]mean (sd)median [IQR]median [IQR]mean (sd)mean (sd)median [IQR]mean (sd)mean (sd) | | 164 (0.5%) | 27 (0.4%) | 0.01 | 188 (0.4%) | 20 (0.1%) | 0.06 | 352 (0.4%) | 47 (0.2%) | 0.04 |
| mean (sd) 9.12 (4.59) 8.43 (4.41) 0.15 8.69 (4.31) 8.22 (4.10) 0.11 8.86 (4.42) 8.29 (4.20) 0.13median [IQR] 8.00 [6.00, 12.00] 7.00 [5.00, 11.00] 0.22 8.00 [5.00, 11.00] 7.00 [5.00, 10.00] 0.24 8.00 (4.42) 7.00 (4.20) 0.23 Number of Hospitalizationsmean (sd) 1.12 (0.38) 1.09 (0.31) 0.09 1.10 (0.33) 1.07 (0.28) 0.10 1.11 (0.35) 1.08 (0.29) 0.09 Number of hospital daysmean (sd) 4.12 (3.05) 3.71 (2.07) 0.16 3.87 (2.26) 3.60 (1.70) 0.14 3.97 (2.60) 3.63 (1.82) 0.15 | • | | | | | | | | | |
| median [IQR] 8.00 [6.00, 12.00] 7.00 [5.00, 11.00] 0.22 8.00 [5.00, 11.00] 7.00 [5.00, 10.00] 0.24 8.00 (4.42) 7.00 (4.20) 0.23 Number of Hospitalizationsmean (sd) 1.12 (0.38) 1.09 (0.31) 0.09 1.10 (0.33) 1.07 (0.28) 0.10 1.11 (0.35) 1.08 (0.29) 0.09 median [IQR] 1.00 [1.00, 1.00] 1.00 [1.00, 1.00] 0.00 1.00 [1.00, 1.00] 0.00 1.00 [0.35) 1.00 (0.29) 0.00 Number of hospital daysmean (sd) 4.12 (3.05) 3.71 (2.07) 0.16 3.87 (2.26) 3.60 (1.70) 0.14 3.97 (2.60) 3.63 (1.82) 0.15 | | | | | | | | | | |
| Number of Hospitalizationsmean (sd)median [IQR]median [IQR]median solutionsmean (sd)median solutionsmean (sd)mean solutionsmean solutions | | | | | , , | | | | , , | |
| mean (sd) 1.12 (0.38) 1.09 (0.31) 0.09 1.10 (0.33) 1.07 (0.28) 0.10 1.11 (0.35) 1.08 (0.29) 0.09 1.00 [1.00, 1.00] 1.00 [1.00, 1.00] 1.00 [1.00, 1.00] 1.00 [1.00, 1.00] 1.00 [1.00, 1.00] 0.00 1.00 (0.35) 1.00 (0.29) 0.00 Number of hospital days 1.00 (sd) 1.00 (sd | | 8.00 [6.00, 12.00] | 7.00 [5.00, 11.00] | 0.22 | 8.00 [5.00, 11.00] | 7.00 [5.00, 10.00] | 0.24 | 8.00 (4.42) | 7.00 (4.20) | 0.23 |
| median [IQR] 1.00 [1.00, 1.00] 1.00 [1.00, 1.00] 0.00 1.00 [1.00, 1.00] 0.00 1.00 [1.00, 1.00] 0.00 1.00 (0.35) 1.00 (0.29) 0.00 Number of hospital days 4.12 (3.05) 3.71 (2.07) 0.16 3.87 (2.26) 3.60 (1.70) 0.14 3.97 (2.60) 3.63 (1.82) 0.15 | - | | | | | | | | | |
| Number of hospital daysmean (sd) 4.12 (3.05) 3.71 (2.07) 0.16 3.87 (2.26) 3.60 (1.70) 0.14 3.97 (2.60) 3.63 (1.82) 0.15 | mean (sd) | 1.12 (0.38) | 1.09 (0.31) | 0.09 | 1.10 (0.33) | 1.07 (0.28) | 0.10 | 1.11 (0.35) | 1.08 (0.29) | 0.09 |
| mean (sd) 4.12 (3.05) 3.71 (2.07) 0.16 3.87 (2.26) 3.60 (1.70) 0.14 3.97 (2.60) 3.63 (1.82) 0.15 | | 1.00 [1.00, 1.00] | 1.00 [1.00, 1.00] | 0.00 | 1.00 [1.00, 1.00] | 1.00 [1.00, 1.00] | 0.00 | 1.00 (0.35) | 1.00 (0.29) | 0.00 |
| | Number of hospital days | | | | | | | | | |
| median [IQR] 3.00 [3.00, 4.00] 3.00 [3.00, 4.00] 0.00 3.00 [3.00, 4.00] 0.00 3.00 (2.60) 3.00 (1.82) 0.00 | mean (sd) | 4.12 (3.05) | 3.71 (2.07) | 0.16 | 3.87 (2.26) | 3.60 (1.70) | 0.14 | 3.97 (2.60) | 3.63 (1.82) | 0.15 |
| | median [IQR] | 3.00 [3.00, 4.00] | 3.00 [3.00, 4.00] | 0.00 | 3.00 [3.00, 4.00] | 3.00 [3.00, 4.00] | 0.00 | 3.00 (2.60) | 3.00 (1.82) | 0.00 |

Table 1: Prasugrel 10 mg vs Clopidogrel 75 mg

| Number of Emergency Department (ED) visits | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|
| mean (sd) | 1.07 (1.31) | 0.88 (1.12) | 0.16 | 3.06 (5.31) | 3.09 (5.66) | -0.01 | 2.28 (4.23) | 2.40 (4.74) | -0.03 |
| median [IQR] | 1.00 [0.00, 1.00] | 1.00 [0.00, 1.00] | 0.00 | 2.00 [0.00, 4.00] | 2.00 [0.00, 4.00] | 0.00 | 1.61 (4.23) | 1.69 (4.74) | -0.02 |
| Number of Office visits | | | | | | | | | |
| mean (sd) | 3.42 (3.55) | 2.95 (3.26) | 0.14 | 3.00 (3.50) | 2.64 (3.14) | 0.11 | 3.16 (3.52) | 2.74 (3.18) | 0.13 |
| median [IQR] | 2.00 [1.00, 5.00] | 2.00 [1.00, 4.00] | 0.00 | 2.00 [1.00, 4.00] | 2.00 [1.00, 4.00] | 0.00 | 2.00 (3.52) | 2.00 (3.18) | 0.00 |
| Number of Endocrinologist visits | | | | | | | | | |
| mean (sd) | 0.17 (1.23) | 0.19 (1.29) | -0.02 | 0.14 (1.13) | 0.18 (1.30) | -0.03 | 0.50 (1.20) | 0.40 (1.25) | 0.08 |
| median [IQR] | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 | 0.39 (1.20) | 0.31 (1.25) | 0.07 |
| Number of internal medicine/family | | | | | | | | | |
| medicine visits | | | | | | | | | |
| mean (sd) | 7.06 (10.34) | 5.39 (9.08) | 0.17 | 3.96 (6.97) | 3.52 (6.05) | 0.07 | 5.17 (8.45) | 4.10 (7.13) | 0.14 |
| median [IQR] | 4.00 [1.00, 9.00] | 3.00 [0.00, 7.00] | 0.10 | 2.00 [0.00, 5.00] | 2.00 [0.00, 5.00] | 0.00 | 2.78 (8.45) | 2.31 (7.13) | 0.06 |
| Number of Cardiologist visits | | | | | | | | | |
| mean (sd) | 9.87 (6.11) | 9.28 (5.43) | 0.10 | 1.18 (2.77) | 1.04 (2.36) | 0.05 | 4.57 (4.39) | 3.61 (3.61) | 0.24 |
| median [IQR] | 9.00 [6.00, 13.00] | 8.00 [6.00, 12.00] | 0.17 | 0.00 [0.00, 1.00] | 0.00 [0.00, 1.00] | 0.00 | 3.52 (4.39) | 2.49 (3.61) | 0.26 |
| Number electrocardiograms received | | . , . | | . , , | . , , | | , , | , , | |
| mean (sd) | 3.53 (2.68) | 3.19 (2.39) | 0.13 | 1.15 (1.49) | 1.05 (1.41) | 0.07 | 2.08 (2.04) | 1.72 (1.77) | 0.19 |
| median [IQR] | 3.00 [2.00, 5.00] | 3.00 [1.00, 4.00] | 0.00 | 1.00 [0.00, 2.00] | 1.00 [0.00, 2.00] | 0.00 | 1.78 (2.04) | 1.62 (1.77) | 0.08 |
| Number of HbA1c tests ordered | | (=,) | | [,] | | | (, | , | |
| mean (sd) | 0.34 (0.67) | 0.31 (0.64) | 0.05 | 0.21 (0.53) | 0.23 (0.55) | -0.04 | 0.26 (0.59) | 0.25 (0.58) | 0.02 |
| median [IQR] | 0.00 [0.00, 1.00] | 0.00 [0.00, 0.00] | 0.00 | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 | 0.00 (0.59) | 0.00 (0.58) | 0.00 |
| Number of glucose tests ordered | 0.00 [0.00) 1.00] | 0.00 [0.00, 0.00] | 0.00 | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 | 0.00 (0.00) | 0.00 (0.00) | 0.00 |
| mean (sd) | 0.17 (0.86) | 0.15 (1.08) | 0.02 | 0.12 (0.71) | 0.12 (0.59) | 0.00 | 0.14 (0.77) | 0.13 (0.78) | 0.01 |
| median [IQR] | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 | 0.00 (0.77) | 0.00 (0.78) | 0.00 |
| Number of lipid tests ordered | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 | 0.00 (0.77) | 0.00 (0.70) | 0.00 |
| mean (sd) | 0.50 (0.77) | 0.49 (0.76) | 0.01 | 0.37 (0.77) | 0.43 (0.75) | -0.08 | 0.42 (0.77) | 0.45 (0.75) | -0.04 |
| median [IQR] | 0.00 [0.00, 1.00] | 0.00 [0.00, 1.00] | 0.00 | 0.00 [0.00, 1.00] | 0.00 [0.00, 1.00] | 0.00 | 0.00 (0.77) | 0.43 (0.75) | 0.00 |
| Number of creatinine tests ordered | 0.00 [0.00, 1.00] | 0.00 [0.00, 1.00] | 0.00 | 0.00 [0.00, 1.00] | 0.00 [0.00, 1.00] | 0.00 | 0.00 (0.77) | 0.00 (0.73) | 0.00 |
| mean (sd) | 0.06 (0.32) | 0.03 (0.24) | 0.11 | 0.06 (0.37) | 0.04 (0.34) | 0.06 | 0.06 (0.35) | 0.04 (0.31) | 0.06 |
| median [IQR] | 0.00 (0.32) | 0.03 (0.24) | 0.00 | 0.00 [0.00, 0.00] | 0.04 (0.34) | 0.00 | 0.00 (0.35) | 0.04 (0.31) | 0.00 |
| Number of BUN tests ordered | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 | 0.00 (0.33) | 0.00 (0.31) | 0.00 |
| | 0.03 (0.30) | 0.02 (0.38) | 0.03 | 0.04 (0.36) | 0.03 (0.25) | 0.03 | 0.04 (0.34) | 0.03 (0.30) | 0.03 |
| mean (sd) | ` ′ | ` ' | 0.03 | , , | ` ' | 0.03 | ` ' | ` ' | 0.03 |
| median [IQR] Number of tests for microalbuminuria | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 | 0.00 (0.34) | 0.00 (0.30) | 0.00 |
| | 0.10 (0.64) | 0.17/0.63\ | 0.02 | 0.10 (0.46) | 0.13 (0.40) | 0.04 | 0.14(0.54) | 0.14(0.54) | 0.00 |
| mean (sd) | 0.19 (0.64) | 0.17 (0.63) | 0.03 | 0.10 (0.46) | 0.12 (0.49) | -0.04 | 0.14 (0.54) | 0.14 (0.54) | 0.00 |
| median [IQR] | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 | 0.00 (0.54) | 0.00 (0.54) | 0.00 |
| Total N distinct ICD9/ICD10 diagnoses at the 3rd digit level | | | | | | | | | |
| mean (sd) | 7.74 (9.49) | 5.68 (8.22) | 0.23 | 4.21 (7.22) | 3.52 (6.47) | 0.10 | 5.59 (8.18) | 4.19 (7.06) | 0.18 |
| median [IQR] | 5.00 [0.00, 13.00] | 0.00 [0.00, 9.00] | 0.56 | 0.00 [0.00, 7.00] | 0.00 [0.00, 4.00] | 0.00 | 1.95 (8.18) | 0.00 (7.06) | 0.26 |
| For PS | | | | | | | | | |
| Hemorrhagic stroke+Other<br>cerebrovascular disease+Cerebrovascular<br>procedure (for PS); n (%) | 465 (1.4%) | 44 (0.6%) | 0.08 | 420 (0.8%) | 47 (0.3%) | 0.07 | 885 (1.1%) | 91 (0.4%) | 0.08 |

Table 1: Prasugrel 10 mg vs Clopidogrel 75 mg

| Occurrence of creatinine tests ordered (for PS); n (%) | 1,365 (4.2%) | 160 (2.3%) | 0.11 | 2,291 (4.5%) | 467 (3.1%) | 0.07 | 3,656 (4.4%) | 0,627 (2.8%) | 0.09 |
|---|---|---|---|---|---|---|---|---|---|
| Occurrence of BUN tests ordered (for PS); n (%) | 761 (2.3%) | 85 (1.2%) | 0.08 | 1,388 (2.7%) | 311 (2.0%) | 0.05 | 2,149 (2.6%) | 0,396 (1.8%) | 0.05 |
| Occurrence of chronic renal insufficiency w/o CKD (for PS); n (%) | 2,591 (8.0%) | 320 (4.7%) | 0.14 | 1,642 (3.2%) | 301 (2.0%) | 0.08 | 4,233 (5.1%) | 0,621 (2.8%) | 0.12 |
| Chronic kidney disease Stage 1-2 (for PS); n (%) | 668 (2.1%) | 86 (1.3%) | 0.06 | 418 (0.8%) | 101 (0.7%) | 0.01 | 1086 (1.3%) | 187 (0.8%) | 0.05 |
| Chronic kidney disease Stage 3-6 (for PS); n (%) | 3,066 (9.4%) | 323 (4.7%) | 0.18 | 2,086 (4.1%) | 312 (2.1%) | 0.12 | 5,152 (6.2%) | 0,635 (2.9%) | 0.16 |
| Bladder stones+Kidney stones (for PS); n (%) | 744 (2.3%) | 148 (2.2%) | 0.01 | 879 (1.7%) | 263 (1.7%) | 0.00 | 1,623 (1.9%) | 0,411 (1.9%) | 0.00 |
| Diabetes with peripheral circulatory disorders+Gangrene+Osteomyelitis(for PS) with ICD10; n (%) | 1,023 (3.1%) | 115 (1.7%) | 0.09 | 646 (1.3%) | 144 (0.9%) | 0.04 | 1,669 (2.0%) | 0,259 (1.2%) | 0.06 |
| Alcohol abuse or dependence+Drug abuse or dependence (for PS); n (%) | 11 (0.0%) | 2 (0.0%) | #DIV/0! | 505 (1.0%) | 170 (1.1%) | -0.01 | 516 (0.6%) | 172 (0.8%) | -0.02 |
| Diabetes with other ophthalmic<br>manifestations+Retinal detachment,<br>vitreous hemorrhage, vitrectomy+Retinal<br>laser coagulation therapy (for PS); n (%) | 138 (0.4%) | 18 (0.3%) | 0.02 | 511 (1.0%) | 129 (0.8%) | 0.02 | 0,649 (0.8%) | 0,147 (0.7%) | 0.01 |
| Other atherosclerosis+Cardiac conduction disorders+Other CVD (for PS); n (%) | 14,046 (43.1%) | 2,369 (34.5%) | 0.18 | 15,374 (30.3%) | 3,959 (26.1%) | 0.09 | 29,420 (35.3%) | 6,328 (28.7%) | 0.14 |
| Previous cardiac procedure (CABG or PTCA or Stent) + History of CABG or PTCA (for PS) ; n (%) | 32,053 (98.5%) | 6,809 (99.1%) | -0.06 | 49,901 (98.2%) | 14,978 (98.6%) | -0.03 | 81,954 (98.3%) | 21,787 (98.8%) | -0.04 |
| Hyperthyroidism + Hypothyroidism + Other disorders of thyroid gland (for PS); n (%) | 4,843 (14.9%) | 758 (11.0%) | 0.12 | 4,841 (9.5%) | 1,139 (7.5%) | 0.07 | 9,684 (11.6%) | 1,897 (8.6%) | 0.10 |
| Delirium + Psychosis (for PS); n (%) | 215 (0.7%) | 22 (0.3%) | 0.06 | 162 (0.3%) | 25 (0.2%) | 0.02 | 377 (0.5%) | 47 (0.2%) | 0.05 |
| Any use of Meglitinides (for PS); n (%) | 63 (0.2%) | 16 (0.2%) | 0.00 | 146 (0.3%) | 37 (0.2%) | 0.02 | 209 (0.3%) | 53 (0.2%) | 0.02 |
| Any use of AGIs (for PS); n (%) | 21 (0.1%) | 3 (0.0%) | 0.04 | 36 (0.1%) | 5 (0.0%) | 0.04 | 29,420 (35.3%) | 6,328 (28.7%) | 0.14 |
| CKD stage 3-6 + dialysis (for PS); n (%) | 3,070 (9.4%) | 324 (4.7%) | 0.18 | 2,095 (4.1%) | 314 (2.1%) | 0.12 | 5,165 (6.2%) | 0,638 (2.9%) | 0.16 |
| Use of thiazide; n (%) | 2,836 (8.7%) | 460 (6.7%) | 0.08 | 3,685 (7.3%) | 913 (6.0%) | 0.05 | 73,405 (88.1%) | 19,556 (88.7%) | -0.02 |
| Use of beta blockers; n (%) | 28,402 (87.2%) | 5,986 (87.1%) | 0.00 | 45,003 (88.6%) | 13,570 (89.4%) | -0.03 | 17,365 (20.8%) | 3,512 (15.9%) | 0.13 |
| Use of calcium channel blockers; n (%) | 7,523 (23.1%) | 1,165 (17.0%) | 0.15 | 9,842 (19.4%) | 2,347 (15.5%) | 0.10 | 16,281 (19.5%) | 4,174 (18.9%) | 0.02 |
| All antidiabetic medications except Insulin; n (%) | 6,890 (21.2%) | 1,389 (20.2%) | 0.02 | 9,391 (18.5%) | 2,785 (18.3%) | 0.01 | 6,521 (7.8%) | 1,373 (6.2%) | 0.06 |
| DM Medications - Insulin ; n (%) | 2,879 (8.8%) | 621 (9.0%) | -0.01 | 3,775 (7.4%) | 1,127 (7.4%) | 0.00 | 6,654 (8.0%) | 1,748 (7.9%) | 0.00 |
| Use of Low Intensity Statins; n (%) | 12,186 (37.4%) | 2,249 (32.7%) | 0.10 | 20,920 (41.2%) | 5,246 (34.5%) | 0.14 | 33106 (39.7%) | 7,495 (34.0%) | 0.12 |
| Use of High Intensity Statins; n (%) | 19,933 (61.2%) | 4,628 (67.3%) | -0.13 | 28,101 (55.3%) | 9,643 (63.5%) | -0.17 | 48034 (57.6%) | 14,271 (64.7%) | -0.15 |
| Malignant hypertension; n (%) | 2,535 (7.8%) | 300 (4.4%) | 0.14 | 26,315 (51.8%) | 7,468 (49.2%) | 0.05 | 28850 (34.6%) | 7,768 (35.2%) | -0.01 |
| Cardiovascular stress test; n (%) | 92 (0.3%) | 7 (0.1%) | 0.04 | 93 (0.2%) | 21 (0.1%) | 0.03 | 0,185 (0.2%) | 28 (0.1%) | 0.03 |
| Echocardiogram; n (%) | 22,726 (69.8%) | 4,521 (65.8%) | 0.09 | 31,917 (62.8%) | 9,448 (62.2%) | 0.01 | 54,643 (65.6%) | 13969 (63.3%) | 0.05 |
| Number of BNP tests<br>mean (sd) | 0.09 (0.38) | 0.06 (0.29) | 0.09 | 0.11 (0.37) | 0.12 (0.37) | -0.03 | 0.10 (0.37) | 0.10 (0.35) | 0.00 |

Table 1: Prasugrel 10 mg vs Clopidogrel 75 mg

| median [IQR] | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 | 0.00 (0.37) | 0.00 (0.35) | 0.00 |
|---|---|---|---|---|---|---|---|---|---|
| Number of Cardiac biomarkers tests | | | | | | | | | |
| (tropnin, CK-MBs, Myoglobin, CPK) | | | | | | | | | |
| mean (sd) | 0.54 (1.57) | 0.41 (1.70) | 0.08 | 0.73 (1.62) | 0.80 (1.75) | -0.04 | 0.66 (1.60) | 0.68 (1.73) | -0.01 |
| median [IQR] | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 | 0.00 [0.00, 1.00] | 0.00 [0.00, 1.00] | 0.00 | 0.00 (1.60) | 0.00 (1.73) | 0.00 |
| Number of Ambulatory Blood pressure | | | | | | | | | |
| monitoring tests | | | | | | | | | |
| mean (sd) | 0.00 (0.03) | 0.00 (0.02) | 0.00 | 0.00 (0.03) | 0.00 (0.02) | 0.00 | 0.00 (0.03) | 0.00 (0.02) | 0.00 |
| median [IQR] | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 | 0.00 (0.03) | 0.00 (0.02) | 0.00 |
| N of days on antihypertensive medications | | | | | | | | | |
| during baseline | | | | | | | | | |
| mean (sd) | 85.76 (79.72) | 67.64 (76.90) | 0.23 | 75.26 (78.87) | 62.73 (75.55) | 0.16 | 79.36 (79.20) | 64.26 (75.97) | 0.19 |
| median [IQR] | 88.00 [1.00, 174.00] | | 1.03 | 31.00 [1.00, 168.00] | 2.00 [1.00, 153.00] | 0.38 | 53.26 (79.20) | 3.56 (75.97) | 0.64 |
| N of days in database anytime prior | | , | | | | | | , | |
| mean (sd) | 1,683.97 (1,295.93) | 1.631.68 (1.231.18) | 0.04 | 1,749.68 (1,252.71) | 1,712.87 (1,215.17) | 0.03 | 1724.01 (1269.77) | 1687.58 (1220.18) | 0.03 |
| median [IQR] | 1,324.00 [651.25, | 1,300.50 [633.00, | 0.02 | 1,412.00 [682.00, | 1,374.00 [702.00, | 0.03 | 1377.63 (1269.77) | , , | 0.02 |
| rearan part | 2,398.00] | 2,373.75] | 0.02 | 2,626.00] | 2,607.00] | 0.03 | 13.7.03 (1203.77) | 1331.10 (1220.10) | 0.02 |
| Mean Copay for per prescription cost | 2,330.00] | 2,373.73] | | 2,020.00] | 2,007.00] | | | | |
| (charges in U.S. \$) (180-1 day prior) | | | | | | | | | |
| mean (sd) | 23.49 (30.72) | 25.23 (27.71) | -0.06 | 19.47 (32.84) | 19.60 (23.87) | 0.00 | 21.04 (32.03) | 21.35 (25.13) | -0.01 |
| median [IQR] | 15.00 [6.31, 30.00] | 18.00 [8.00, 33.46] | -0.10 | 13.45 [5.38, 25.57] | 13.28 [5.00, 26.50] | 0.01 | 14.06 (32.03) | 14.75 (25.13) | -0.01 |
| Missing; n (%) | 4,763 (14.6%) | 1,189 (17.3%) | -0.10 | 8,729 (17.2%) | 2,756 (18.1%) | -0.02 | 13,492 (16.2%) | 3945 (17.9%) | -0.02 |
| | | | 0.00 | | | 0.02 | | , , | -0.03<br>-0.01 |
| Colonos; n (%) | 1,036 (3.2%) | 221 (3.2%) | | 1,556 (3.1%) | 476 (3.1%) | | 2,592 (3.1%) | 697 (3.2%) | |
| Fecal occult blood (FOB) test; n (%) | 892 (2.7%) | 216 (3.1%) | -0.02 | 1,516 (3.0%) | 405 (2.7%) | 0.02 | 2,408 (2.9%) | 621 (2.8%) | 0.01 |
| Flu vaccine; n (%) | 4,380 (13.5%) | 793 (11.5%) | 0.06 | 4,052 (8.0%) | 1,152 (7.6%) | 0.01 | 8,432 (10.1%) | 1945 (8.8%) | 0.04 |
| Mammogram; n (%) | 1,884 (5.8%) | 312 (4.5%) | 0.06 | 2,318 (4.6%) | 545 (3.6%) | 0.05 | 4,202 (5.0%) | 857 (3.9%) | 0.05 |
| Pap smear; n (%) | 580 (1.8%) | 141 (2.1%) | -0.02 | 1,171 (2.3%) | 348 (2.3%) | 0.00 | 1,751 (2.1%) | 489 (2.2%) | -0.01 |
| Pneumonia vaccine; n (%) | 3,945 (12.1%) | 725 (10.6%) | 0.05 | 2,330 (4.6%) | 656 (4.3%) | 0.01 | 6,275 (7.5%) | 1381 (6.3%) | 0.05 |
| PSA test or Prostate exam for DRE; n (%) | 4,334 (13.3%) | 1,050 (15.3%) | -0.06 | 5,608 (11.0%) | 2,061 (13.6%) | -0.08 | 9,942 (11.9%) | 3111 (14.1%) | -0.07 |
| Bone mineral density; n (%) | 686 (2.1%) | 105 (1.5%) | 0.05 | 594 (1.2%) | 103 (0.7%) | 0.05 | 1,280 (1.5%) | 208 (0.9%) | 0.06 |
| Use of Sympatomimetic agents; n (%) | 261 (0.8%) | 72 (1.0%) | -0.02 | 542 (1.1%) | 186 (1.2%) | -0.01 | 0,803 (1.0%) | 258 (1.2%) | -0.02 |
| Use of CNS stimulants; n (%) | 101 (0.3%) | 29 (0.4%) | -0.02 | 267 (0.5%) | 76 (0.5%) | 0.00 | 0,368 (0.4%) | 105 (0.5%) | -0.01 |
| Use of estrogens, progestins, androgens; n (%) | 946 (2.9%) | 268 (3.9%) | -0.06 | 2,000 (3.9%) | 656 (4.3%) | -0.02 | 2,946 (3.5%) | 924 (4.2%) | -0.04 |
| Use of Angiogenesis inhibitors; n (%) | 14 (0.0%) | 0 (0.0%) | #DIV/0! | 29 (0.1%) | 2 (0.0%) | 0.04 | 0,043 (0.1%) | 2 (0.0%) | 0.04 |
| Use of Oral Immunosuppressants; n (%) | 63 (0.2%) | 6 (0.1%) | 0.03 | 128 (0.3%) | 29 (0.2%) | 0.02 | 0,191 (0.2%) | 35 (0.2%) | 0.00 |
| Use of fondaparinux or Bivalirudin; n (%) | 11 (0.0%) | 3 (0.0%) | #DIV/0! | 20 (0.0%) | 2 (0.0%) | #DIV/0! | 0,031 (0.0%) | 5 (0.0%) | #DIV/0! |
| Use of other direct thrombin inhibitors<br>(lepirudin, desirudin, argatroban); n (%) | 0 (0.0%) | 0 (0.0%) | #DIV/0! | 0 (0.0%) | 0 (0.0%) | #DIV/0! | 0,000 (0.0%) | 0 (0.0%) | #DIV/0! |
| | 440 /4 20/1 | 02/4 22/ | 0.04 | 430 (2.22/) | 122 (0.000) | 0.00 | 0.046 (4.000) | 205 (0.00/) | 0.04 |
| Use of Prasugrel ON CED; n (%) | 418 (1.3%) | 82 (1.2%) | 0.01 | 428 (0.8%) | 123 (0.8%) | 0.00 | 0,846 (1.0%) | 205 (0.9%) | 0.01 |
| Use of Prasugrel 180 to 1 day prior; n (%) | 417 (1.3%) | 90 (1.3%) | 0.00 | 423 (0.8%) | 135 (0.9%) | -0.01 | 0,840 (1.0%) | 225 (1.0%) | 0.00 |
| Duration of index hospitalization (i.e. anchor hospitalization LOS) | | | | | | | | | |

Table 1: Prasugrel 10 mg vs Clopidogrel 75 mg

| mean (sd) | 3.61 (2.82) | 3.37 (1.49) | 0.11 | 3.58 (1.67) | 3.38 (1.34) | 0.13 | 3.59 (2.19) | 3.38 (1.39) | 0.11 |
|---|---|---|---|---|---|---|---|---|---|
| median [IQR] | 3.00 [3.00, 4.00] | 3.00 [3.00, 4.00] | 0.00 | 3.00 [3.00, 4.00] | 3.00 [3.00, 4.00] | 0.00 | 3.00 (2.19) | 3.00 (1.39) | 0.00 |
| Number of D-dimer tests | | | | | | | | | |
| mean (sd) | 0.04 (0.21) | 0.02 (0.17) | 0.10 | 0.05 (0.24) | 0.06 (0.26) | -0.04 | 0.05 (0.23) | 0.05 (0.24) | 0.00 |
| median [IQR] | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 | 0.00 (0.23) | 0.00 (0.24) | 0.00 |
| Numbe of CRP, high-sensitivity CRP tests | | | | | | | | | |
| mean (sd) | 0.05 (0.30) | 0.04 (0.24) | 0.04 | 0.04 (0.28) | 0.04 (0.28) | 0.00 | 0.04 (0.29) | 0.04 (0.27) | 0.00 |
| median [IQR] | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 | 0.00 (0.29) | 0.00 (0.27) | 0.00 |
| Number of PT or aPTTt tests | | | | | | | ( , | , | |
| mean (sd) | 0.46 (1.66) | 0.21 (0.99) | 0.18 | 0.47 (1.28) | 0.43 (1.01) | 0.03 | 0.47 (1.44) | 0.36 (1.00) | 0.09 |
| median [IQR] | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 | 0.00 [0.00, 0.00] | 0.00 [0.00, 1.00] | 0.00 | 0.00 (1.44) | 0.00 (1.00) | 0.00 |
| Number of Bleeding time tests | . , , | . , , | | . , . | . , . | | , , | , , | |
| mean (sd) | 0.00 (0.02) | 0.00 (0.01) | 0.00 | 0.00 (0.02) | 0.00 (0.01) | 0.00 | 0.00 (0.02) | 0.00 (0.01) | 0.00 |
| median [IQR] | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 | 0.00 (0.02) | 0.00 (0.01) | 0.00 |
| HAS-BLED Score (ICD-9 and ICD-10), 180 | | | | | | | , | , | |
| days | | | | | | | | | |
| mean (sd) | 3.74 (0.76) | 3.42 (0.67) | 0.45 | 3.38 (0.65) | 3.16 (0.50) | 0.38 | 3.52 (0.70) | 3.24 (0.56) | 0.44 |
| median [IQR] | 4.00 [3.00, 4.00] | 3.00 [3.00, 4.00] | 1.40 | 3.00 [3.00, 4.00] | 3.00 [3.00, 3.00] | 0.00 | 3.39 (0.70) | 3.00 (0.56) | 0.62 |
| Drug eluting stent; n (%) | 14,767 (45.4%) | 3,976 (57.9%) | -0.25 | 21,794 (42.9%) | 7,216 (47.5%) | -0.09 | 36,561 (43.9%) | 11192 (50.7%) | -0.14 |
| Bare metal stent; n (%) | 21,714 (66.7%) | 4,304 (62.6%) | 0.09 | 23,619 (46.5%) | 7,240 (47.7%) | -0.02 | 45,333 (54.4%) | 11544 (52.3%) | 0.04 |
| Use of CYP inhibitors; n (%) | 5,868 (18.0%) | 1,035 (15.1%) | 0.08 | 8,155 (16.1%) | 2,209 (14.5%) | 0.04 | 14,023 (16.8%) | 3244 (14.7%) | 0.06 |
| Use of CYP inducers; n (%) | 237 (0.7%) | 32 (0.5%) | 0.03 | 363 (0.7%) | 83 (0.5%) | 0.03 | 0,600 (0.7%) | 115 (0.5%) | 0.03 |
| Commercial vs Medicare Advantage- | - ( , | (- ( ) | | , | , | | -, ( , | - ( / | |
| Business Type Code - CORRECT ONE - | | | | | | | | | |
| TRUVEN | | | | | | | | | |
| Commercial; n (%) | 14,856 (45.6%) | 4,721 (68.7%) | -0.48 | 15,837 (31.2%) | 2,186 (14.4%) | 0.41 | 30,693 (36.8%) | 6907 (31.3%) | 0.12 |
| Medicare Advantage; n (%) | 17,700 (54.4%) | 2,151 (31.3%) | 0.48 | 34,958 (68.8%) | 13,001 (85.6%) | -0.41 | 52,658 (63.2%) | 15152 (68.7%) | -0.12 |
| Commercial vs Medicare Advantage- | | | | | | | | | |
| Business Type Code | 14.056 (45.60/) | 4 724 (60 70/) | 0.40 | | | 40.401.1151 | 14 056 (45 60/) | 4 724 (60 70/) | 0.40 |
| COM = COMMERCIAL; n (%) | 14,856 (45.6%) | 4,721 (68.7%) | -0.48 | - | - | #VALUE! | 14,856 (45.6%) | 4,721 (68.7%) | -0.48 |
| MCR = MEDICARE; n (%) | 17,700 (54.4%) | 2,151 (31.3%) | 0.48 | - | - | #VALUE! | 17,700 (54.4%) | 2,151 (31.3%) | 0.48 |
| MCD = MEDICAID; n (%) | 0 (0.0%) | 0 (0.0%) | #DIV/0! | - | - | #VALUE! | 0 (0.0%) | 0 (0.0%) | #DIV/0! |
| NONE = NO BUSINESS LINE CODE (added | 0 (0.0%) | 0 (0.0%) | #DIV/0! | - | - | #VALUE! | 0 (0.0%) | 0 (0.0%) | #DIV/0! |
| in 2015); n (%)<br>UNK = UNKNOWN (added in 2015); n (%) | 0 (0.0%) | 0 (0.0%) | #DIV/0! | - | - | #VALUE! | 0 (0.0%) | 0 (0.0%) | #DIV/0! |
| Commercial vs Medicare Advantage- Data | | | | | | | | | |
| Type<br>1 - Fee For Service; n (%) | | | #VALUE! | 30,527 (60.1%) | 11,547 (76.0%) | -0.35 | 30,527 (60.1%) | 11,547 (76.0%) | -0.35 |
| ' ' ' | - | - | #VALUE! | | | -0.35<br>-0.03 | | | -0.35<br>-0.03 |
| 2 - Encounter; n (%) | - | - | #VALUE! | 4,431 (8.7%)<br>13,608 (26.8%) | 1,454 (9.6%) | -0.03<br>0.36 | 4,431 (8.7%) | 1,454 (9.6%) | -0.03<br>0.36 |
| 3 - Medicare; n (%)<br>4 - Medicare Encounter; n (%) | - | - | #VALUE! | 2,229 (4.4%) | 1,922 (12.7%)<br>264 (1.7%) | 0.36 | 13,608 (26.8%)<br>2,229 (4.4%) | 1,922 (12.7%)<br>264 (1.7%) | 0.36 |
| , | - | - | #VALUE! | ۷,225 (4.4%) | 204 (1.7%) | 0.10 | ۷,۷۷۶ (4.4%) | 204 (1./%) | 0.16 |
| Metropolitan Statistical Area - Urban (any<br>MSA) vs Rural (non-MSA) | | | | | | | | | |
| Urban; n (%) | - | - | #VALUE! | 38,125 (75.1%) | 11,909 (78.4%) | -0.08 | 38,125 (75.1%) | 11,909 (78.4%) | -0.08 |
| Rural; n (%) | - | - | #VALUE! | 1,177 (2.3%) | 269 (1.8%) | 0.04 | 1,177 (2.3%) | 269 (1.8%) | 0.04 |

Table 1: Prasugrel 10 mg vs Clopidogrel 75 mg

| N of Generic name drugs | | | | 0 | 0 | | 0 | 0 | |
|---|---|---|---|---|---|---|---|---|---|
| mean (sd) | 13.63 (11.66) | 11.15 (10.53) | 0.22 | 11.00 (9.22) | 9.50 (8.53) | 0.17 | 12.03 (10.24) | 10.01 (9.20) | 0.21 |
| median [IQR] | 10.00 [5.00, 18.00] | 8.00 [4.00, 15.00] | 0.18 | 8.00 [5.00, 15.00] | 7.00 [4.00, 12.00] | 0.11 | 8.78 (10.24) | 7.31 (9.20) | 0.15 |
| N of Brand name drugs | | | | 0 | 0 | | 0 | 0 | |
| mean (sd) | 3.10 (4.35) | 3.81 (4.42) | -0.16 | 3.61 (4.23) | 3.98 (4.17) | -0.09 | 3.41 (4.28) | 3.93 (4.25) | -0.12 |
| median [IQR] | 2.00 [0.00, 4.00] | 2.00 [1.00, 5.00] | 0 | 2.00 [1.00, 5.00] | 2.00 [2.00, 5.00] | 0 | 2.00 (4.28) | 2.00 (4.25) | 0.00 |

Table 1: Prasugrel 10 mg vs Clopidogrel 75 mg

| | | | Р | S-matched | | | | | |
|---|---|---|---|---|---|---|---|---|---|
| | Ор | tum | | 1 | iven | | POO | LED | |
| Variable | Clopidogrel 75mg | Prasugrel 10mg | St. Diff. | Clopidogrel 75mg | Prasugrel 10mg | St. Diff. | Clopidogrel 75mg | Ticagrelor 90mg | St. Diff. |
| Number of patients | 6,835 | 6,835 | | 15,097 | 15,097 | | 21,932 | 21,932 | |
| Age | | | | | | | | | |
| mean (sd) | 58.80 (11.42) | 59.02 (10.25) | -0.02 | 55.93 (10.14) | 56.12 (8.94) | -0.02 | 56.82 (10.56) | 57.02 (9.37) | -0.02 |
| median [IQR] | 58.00 [51.00, 67.00] | 59.00 [52.00, 67.00] | -0.09 | 56.00 [49.00, 62.00] | 57.00 [50.00, 62.00] | -0.10 | 56.62 (10.56) | 57.62 (9.37) | -0.10 |
| Age categories | | | | | | | | | |
| 18 - 54; n (%) | 2,525 (36.9%) | 2,314 (33.9%) | 0.06 | 6,689 (44.3%) | 6,235 (41.3%) | 0.06 | 9,214 (42.0%) | 8,549 (39.0%) | 0.06 |
| 55 - 64; n (%) | 2,191 (32.1%) | 2,291 (33.5%) | -0.03 | 6,340 (42.0%) | 6,718 (44.5%) | -0.05 | 8,531 (38.9%) | 9,009 (41.1%) | -0.04 |
| 65 - 74; n (%) | 1,458 (21.3%) | 1,861 (27.2%) | -0.14 | 1,285 (8.5%) | 1,832 (12.1%) | -0.12 | 2,743 (12.5%) | 3,693 (16.8%) | -0.12 |
| >= 75; n (%) | 661 (9.7%) | 369 (5.4%) | 0.16 | 783 (5.2%) | 312 (2.1%) | 0.17 | 1,444 (6.6%) | 0,681 (3.1%) | 0.16 |
| Gender- United | (* ', | , | | , | - ( - , | | , (, | -, ( , | |
| Males; n (%) | 5,252 (76.8%) | 5,251 (76.8%) | 0.00 | 12,060 (79.9%) | 12,032 (79.7%) | 0.00 | 17,312 (78.9%) | 17,283 (78.8%) | 0.00 |
| Females; n (%) | 1,583 (23.2%) | 1,584 (23.2%) | 0.00 | 3,037 (20.1%) | 3,065 (20.3%) | 0.00 | 4,620 (21.1%) | 4,649 (21.2%) | 0.00 |
| Region | ,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,, | , ( , | | -, ( , | ,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,, | | , ( | , , , | |
| Northeast; n (%) | 516 (7.5%) | 519 (7.6%) | 0.00 | 2,390 (15.8%) | 2,403 (15.9%) | 0.00 | 2,906 (13.3%) | 2,922 (13.3%) | 0.00 |
| South; n (%) | 3,490 (51.1%) | 3,498 (51.2%) | 0.00 | 3,829 (25.4%) | 3,783 (25.1%) | 0.01 | 7,319 (33.4%) | 7,281 (33.2%) | 0.00 |
| Midwest; n (%) | 1,676 (24.5%) | 1,655 (24.2%) | 0.01 | 6,469 (42.8%) | 6,518 (43.2%) | -0.01 | 8,145 (37.1%) | 8,173 (37.3%) | 0.00 |
| West; n (%) | 1,153 (16.9%) | 1,163 (17.0%) | 0.00 | 2,181 (14.4%) | 2,174 (14.4%) | 0.00 | 3,334 (15.2%) | 3,337 (15.2%) | 0.00 |
| Unknown+missing; n (%) | N/A | N/A | #VALUE! | 228 (1.5%) | 219 (1.5%) | 0.00 | 228 (1.0%) | 219 (1.0%) | 0.00 |
| CV Covariates | | | | | | | | | |
| Ischemic heart disease; n (%) | 6,835 (100.0%) | 6,835 (100.0%) | #DIV/0! | 15,097 (100.0%) | 15,097 (100.0%) | #DIV/0! | 21,932 (100.0%) | 21,932 (100.0%) | #DIV/0! |
| Acute MI; n (%) | 6,541 (95.7%) | 6,548 (95.8%) | 0.00 | 14,764 (97.8%) | 14,756 (97.7%) | 0.01 | 21305 (97.1%) | 21304 (97.1%) | 0.00 |
| ACS/unstable angina; n (%) | 2,496 (36.5%) | 2,482 (36.3%) | 0.00 | 4,708 (31.2%) | 4,681 (31.0%) | 0.00 | 7204 (32.8%) | 7163 (32.7%) | 0.00 |
| Old MI; n (%) | 711 (10.4%) | 737 (10.8%) | -0.01 | 991 (6.6%) | 1,009 (6.7%) | 0.00 | 1702 (7.8%) | 1746 (8.0%) | -0.01 |
| Stable angina; n (%) | 1,083 (15.8%) | 1,064 (15.6%) | 0.01 | 1,637 (10.8%) | 1,655 (11.0%) | -0.01 | 2,720 (12.4%) | 2,719 (12.4%) | 0.00 |
| Coronary atherosclerosis and other<br>forms of chronic ischemic heart<br>disease; n (%) | 6,630 (97.0%) | 6,627 (97.0%) | 0.00 | 13,761 (91.2%) | 13,777 (91.3%) | 0.00 | 20,391 (93.0%) | 20,404 (93.0%) | 0.00 |
| Other atherosclerosis with ICD10; n | 115 (1.7%) | 96 (1.4%) | 0.02 | 185 (1.2%) | 156 (1.0%) | 0.02 | 300 (1.4%) | 252 (1.1%) | 0.03 |
| (%) | | | | | | | | | |
| Previous cardiac procedure (CABG or PTCA or Stent) ; n (%) | 6,755 (98.8%) | 6,749 (98.7%) | 0.01 | 14,848 (98.4%) | 14,847 (98.3%) | 0.01 | 21603 (98.5%) | 21596 (98.5%) | 0.00 |
| History of CABG or PTCA; n (%) | 1,761 (25.8%) | 1,624 (23.8%) | 0.05 | 2,106 (13.9%) | 1,980 (13.1%) | 0.02 | 3,867 (17.6%) | 3,604 (16.4%) | 0.03 |
| Any stroke; n (%) | 298 (4.4%) | 287 (4.2%) | 0.01 | 369 (2.4%) | 390 (2.6%) | -0.01 | 0,667 (3.0%) | 0,677 (3.1%) | -0.01 |
| Ischemic stroke (w and w/o mention of | 297 (4.3%) | 287 (4.2%) | 0.00 | 369 (2.4%) | 390 (2.6%) | -0.01 | 0,666 (3.0%) | 0,677 (3.1%) | -0.01 |
| cerebral infarction); n (%) | | | | | | | | | |
| Hemorrhagic stroke; n (%) | 1 (0.0%) | 0 (0.0%) | #DIV/0! | 1 (0.0%) | 0 (0.0%) | #DIV/0! | 2 (0.0%) | 0 (0.0%) | #DIV/0! |
| TIA; n (%) | 53 (0.8%) | 46 (0.7%) | 0.01 | 64 (0.4%) | 63 (0.4%) | 0.00 | 117 (0.5%) | 109 (0.5%) | 0.00 |
| Other cerebrovascular disease; n (%) | 48 (0.7%) | 43 (0.6%) | 0.01 | 39 (0.3%) | 46 (0.3%) | 0.00 | 87 (0.4%) | 89 (0.4%) | 0.00 |
| Late effects of cerebrovascular disease;<br>n (%) | 29 (0.4%) | 28 (0.4%) | 0.00 | 20 (0.1%) | 21 (0.1%) | 0.00 | 49 (0.2%) | 49 (0.2%) | 0.00 |
| Cerebrovascular procedure; n (%) | 3 (0.0%) | 1 (0.0%) | #DIV/0! | 7 (0.0%) | 1 (0.0%) | #DIV/0! | 10 (0.0%) | 2 (0.0%) | #DIV/0! |
| Heart failure (CHF); n (%) | 917 (13.4%) | 939 (13.7%) | -0.01 | 1,558 (10.3%) | 1,623 (10.8%) | -0.02 | 2,475 (11.3%) | 2,562 (11.7%) | -0.01 |
| Peripheral Vascular Disease (PVD) or<br>PVD Surgery ; n (%) | 336 (4.9%) | 359 (5.3%) | -0.02 | 410 (2.7%) | 413 (2.7%) | 0.00 | 0,746 (3.4%) | 0,772 (3.5%) | -0.01 |

Table 1: Prasugrel 10 mg vs Clopidogrel 75 mg

| Ī | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|
| Atrial fibrillation; n (%) | 404 (5.9%) | 412 (6.0%) | 0.00 | 543 (3.6%) | 573 (3.8%) | -0.01 | 0,947 (4.3%) | 0,985 (4.5%) | -0.01 |
| Other cardiac dysrhythmia; n (%) | 1,605 (23.5%) | 1,626 (23.8%) | -0.01 | 2,685 (17.8%) | 2,644 (17.5%) | 0.01 | 4,290 (19.6%) | 4,270 (19.5%) | 0.00 |
| Cardiac conduction disorders; n (%) | 628 (9.2%) | 638 (9.3%) | 0.00 | 1,033 (6.8%) | 957 (6.3%) | 0.02 | 1661 (7.6%) | 1595 (7.3%) | 0.01 |
| Other CVD; n (%) | 1,884 (27.6%) | 1,884 (27.6%) | 0.00 | 3,058 (20.3%) | 3,144 (20.8%) | -0.01 | 4,942 (22.5%) | 5,028 (22.9%) | -0.01 |
| Diabetes-related complications | | | | | | | | | |
| Diabetic retinopathy; n (%) | 125 (1.8%) | 139 (2.0%) | -0.01 | 139 (0.9%) | 152 (1.0%) | -0.01 | 0,264 (1.2%) | 0,291 (1.3%) | -0.01 |
| Diabetes with other ophthalmic | 0 (0.0%) | 6 (0.1%) | -0.04 | 90 (0.6%) | 108 (0.7%) | -0.01 | 0,090 (0.4%) | 0,114 (0.5%) | -0.01 |
| manifestations; n (%) | | | | | | | | | |
| Retinal detachment, vitreous | 4 (0.1%) | 1 (0.0%) | 0.04 | 3 (0.0%) | 4 (0.0%) | #DIV/0! | 7 (0.0%) | 5 (0.0%) | #DIV/0! |
| hemorrhage, vitrectomy; n (%) | | | | | | | | | |
| Retinal laser coagulation therapy; n (%) | 14 (0.2%) | 11 (0.2%) | 0.00 | 25 (0.2%) | 28 (0.2%) | 0.00 | 39 (0.2%) | 39 (0.2%) | 0.00 |
| Occurrence of Diabetic Neuropathy; n<br>(%) | 355 (5.2%) | 329 (4.8%) | 0.02 | 326 (2.2%) | 351 (2.3%) | -0.01 | 0,681 (3.1%) | 0,680 (3.1%) | 0.00 |
| Occurrence of diabetic nephropathy with ICD10 ; n (%) | 231 (3.4%) | 237 (3.5%) | -0.01 | 196 (1.3%) | 199 (1.3%) | 0.00 | 0,427 (1.9%) | 0,436 (2.0%) | -0.01 |
| Hypoglycemia ; n (%) | 66 (1.0%) | 70 (1.0%) | 0.00 | 129 (0.9%) | 137 (0.9%) | 0.00 | 0,195 (0.9%) | 0,207 (0.9%) | 0.00 |
| Hyperglycemia; n (%) | 537 (7.9%) | 517 (7.6%) | 0.01 | 693 (4.6%) | 692 (4.6%) | 0.00 | 1,230 (5.6%) | 1,209 (5.5%) | 0.00 |
| Disorders of fluid electrolyte and acidbase balance; n (%) | 797 (11.7%) | 802 (11.7%) | 0.00 | 1,038 (6.9%) | 1,067 (7.1%) | -0.01 | 1,835 (8.4%) | 1,869 (8.5%) | 0.00 |
| Diabetic ketoacidosis; n (%) | 32 (0.5%) | 21 (0.3%) | 0.03 | 46 (0.3%) | 53 (0.4%) | -0.02 | 78 (0.4%) | 74 (0.3%) | 0.02 |
| Hyperosmolar hyperglycemic nonketotic syndrome (HONK); n (%) | 16 (0.2%) | 18 (0.3%) | -0.02 | 13 (0.1%) | 14 (0.1%) | 0.00 | 29 (0.1%) | 32 (0.1%) | 0.00 |
| Diabetes with peripheral circulatory | 114 (1.7%) | 101 (1.5%) | 0.02 | 111 (0.7%) | 124 (0.8%) | -0.01 | 0,225 (1.0%) | 0,225 (1.0%) | 0.00 |
| disorders with ICD-10; n (%) | 50 (0.00() | 5.4.(0.00() | 0.04 | 402 (0.70() | 04 (0.60() | 0.04 | 4.62 (0.70() | 4.45 (0.70() | 0.00 |
| Diabetic Foot; n (%) | 59 (0.9%) | 54 (0.8%) | 0.01 | 103 (0.7%) | 91 (0.6%) | 0.01 | 162 (0.7%) | 145 (0.7%) | 0.00 |
| Gangrene ; n (%) | 6 (0.1%) | 4 (0.1%) | 0.00 | 5 (0.0%) | 9 (0.1%) | -0.04 | 11 (0.1%) | 13 (0.1%) | 0.00 |
| Lower extremity amputation; n (%) | 16 (0.2%) | 22 (0.3%) | -0.02 | 18 (0.1%) | 23 (0.2%) | -0.03 | 34 (0.2%) | 45 (0.2%) | 0.00 |
| Osteomyelitis; n (%) | 17 (0.2%) | 16 (0.2%) | 0.00 | 36 (0.2%) | 21 (0.1%) | 0.03 | 53 (0.2%) | 37 (0.2%) | 0.00 |
| Skin infections; n (%) | 200 (2.9%) | 239 (3.5%) | -0.03 | 402 (2.7%) | 436 (2.9%) | -0.01 | 0,602 (2.7%) | 0,675 (3.1%) | -0.02 |
| Erectile dysfunction; n (%) | 217 (3.2%) | 238 (3.5%) | -0.02 | 334 (2.2%) | 326 (2.2%) | 0.00 | 0,551 (2.5%) | 0,564 (2.6%) | -0.01 |
| Diabetes with unspecified complication; n (%) | 138 (2.0%) | 147 (2.2%) | -0.01 | 245 (1.6%) | 244 (1.6%) | 0.00 | 0,383 (1.7%) | 0,391 (1.8%) | -0.01 |
| Diabetes mellitus without mention of complications; n (%) | 2,146 (31.4%) | 2,128 (31.1%) | 0.01 | 3,904 (25.9%) | 3,932 (26.0%) | 0.00 | 6,050 (27.6%) | 6,060 (27.6%) | 0.00 |
| Hypertension: 1 inpatient or 2<br>outpatient claims within 365 days; n<br>(%) | 4,975 (72.8%) | 4,998 (73.1%) | -0.01 | 9,576 (63.4%) | 9,586 (63.5%) | 0.00 | 14,551 (66.3%) | 14,584 (66.5%) | 0.00 |
| Hyperlipidemia ; n (%) | 5,523 (80.8%) | 5,550 (81.2%) | -0.01 | 9,909 (65.6%) | 9,936 (65.8%) | 0.00 | 15,432 (70.4%) | 15,486 (70.6%) | 0.00 |
| Edema; n (%) | 188 (2.8%) | 182 (2.7%) | 0.01 | 255 (1.7%) | 260 (1.7%) | 0.00 | 0,443 (2.0%) | 0,442 (2.0%) | 0.00 |
| Renal Dysfunction (non-diabetic) ; n (%) | 910 (13.3%) | 933 (13.7%) | -0.01 | 1,193 (7.9%) | 1,157 (7.7%) | 0.01 | 2,103 (9.6%) | 2,090 (9.5%) | 0.00 |
| Occurrence of acute renal disease ; n (%) | 381 (5.6%) | 403 (5.9%) | -0.01 | 474 (3.1%) | 485 (3.2%) | -0.01 | 855 (3.9%) | 888 (4.0%) | -0.01 |
| Occurrence of chronic renal insufficiency; n (%) | 523 (7.7%) | 547 (8.0%) | -0.01 | 557 (3.7%) | 553 (3.7%) | 0.00 | 1,080 (4.9%) | 1,100 (5.0%) | 0.00 |
| Chronic kidney disease ; n (%) | 500 (7.3%) | 524 (7.7%) | -0.02 | 533 (3.5%) | 533 (3.5%) | 0.00 | 1,033 (4.7%) | 1,057 (4.8%) | 0.00 |
| , | , , | , | - | ,· , | \· / | | , , , | , , , , , , , | -0.01 |

Table 1: Prasugrel 10 mg vs Clopidogrel 75 mg

| Occurrence of hypertensive | 397 (5.8%) | 411 (6.0%) | -0.01 | 391 (2.6%) | 410 (2.7%) | -0.01 | 788 (3.6%) | 821 (3.7%) | -0.01 |
|---|---|---|---|---|---|---|---|---|---|
| nephropathy; n (%) | | / | | | | | / | () | |
| Occurrence of miscellaneous renal | 348 (5.1%) | 358 (5.2%) | 0.00 | 422 (2.8%) | 412 (2.7%) | 0.01 | 0,770 (3.5%) | 0,770 (3.5%) | 0.00 |
| insufficiency; n (%) | 624 (0.20() | F72 (0, 40() | 0.00 | 040 (0 40() | 005 (5.00() | 0.04 | 4.550/7.40/\ | 4 460 (6 70() | 0.00 |
| Glaucoma or cataracts; n (%) | 631 (9.2%) | 573 (8.4%) | 0.03 | 919 (6.1%) | 896 (5.9%) | 0.01 | 1,550 (7.1%) | 1,469 (6.7%) | 0.02 |
| Cellulitis or abscess of toe; n (%) | 36 (0.5%) | 33 (0.5%) | 0.00 | 41 (0.3%) | 48 (0.3%) | 0.00 | 77 (0.4%) | 81 (0.4%) | 0.00 |
| Foot ulcer; n (%) | 58 (0.8%) | 52 (0.8%) | 0.00 | 103 (0.7%) | 91 (0.6%) | 0.01 | 161 (0.7%) | 143 (0.7%) | 0.00 |
| Bladder stones; n (%) | 9 (0.1%) | 7 (0.1%) | 0.00 | 8 (0.1%) | 8 (0.1%) | 0.00 | 17 (0.1%) | 15 (0.1%) | 0.00 |
| Kidney stones; n (%) | 137 (2.0%) | 143 (2.1%) | -0.01 | 271 (1.8%) | 255 (1.7%) | 0.01 | 0,408 (1.9%) | 0,398 (1.8%) | 0.01 |
| Urinary tract infections (UTIs); n (%) | 314 (4.6%) | 303 (4.4%) | 0.01 | 400 (2.6%) | 439 (2.9%) | -0.02 | 0,714 (3.3%) | 0,742 (3.4%) | -0.01 |
| Dipstick urinalysis; n (%) | 1,338 (19.6%) | 1,363 (19.9%) | -0.01 | 3,037 (20.1%) | 3,034 (20.1%) | 0.00 | 4,375 (19.9%) | 4,397 (20.0%) | 0.00 |
| Non-dipstick urinalysis; n (%) | 653 (9.6%) | 659 (9.6%) | 0.00 | 1,171 (7.8%) | 1,211 (8.0%) | -0.01 | 1,824 (8.3%) | 1,870 (8.5%) | -0.01 |
| Urine function test; n (%) | 114 (1.7%) | 105 (1.5%) | 0.02 | 186 (1.2%) | 189 (1.3%) | -0.01 | 0,300 (1.4%) | 0,294 (1.3%) | 0.01 |
| Cytology; n (%) | 50 (0.7%) | 45 (0.7%) | 0.00 | 98 (0.6%) | 85 (0.6%) | 0.00 | 148 (0.7%) | 130 (0.6%) | 0.01 |
| Cystos; n (%) | 66 (1.0%) | 60 (0.9%) | 0.01 | 121 (0.8%) | 112 (0.7%) | 0.01 | 187 (0.9%) | 172 (0.8%) | 0.01 |
| Other Covariates | | | | | | | | | |
| Liver disease; n (%) | 4 (0.1%) | 2 (0.0%) | 0.04 | 6 (0.0%) | 5 (0.0%) | #DIV/0! | 0,010 (0.0%) | 0,007 (0.0%) | #DIV/0! |
| Osteoarthritis; n (%) | 790 (11.6%) | 793 (11.6%) | 0.00 | 1,138 (7.5%) | 1,162 (7.7%) | -0.01 | 1,928 (8.8%) | 1,955 (8.9%) | 0.00 |
| Other arthritis, arthropathies and | 2,079 (30.4%) | 2,059 (30.1%) | 0.01 | 3,709 (24.6%) | 3,698 (24.5%) | 0.00 | 5,788 (26.4%) | 5,757 (26.2%) | 0.00 |
| musculoskeletal pain; n (%) | | | | | | | | | |
| Dorsopathies; n (%) | 1,460 (21.4%) | 1,456 (21.3%) | 0.00 | 2,421 (16.0%) | 2,477 (16.4%) | -0.01 | 3,881 (17.7%) | 3,933 (17.9%) | -0.01 |
| Fractures; n (%) | 110 (1.6%) | 115 (1.7%) | -0.01 | 209 (1.4%) | 208 (1.4%) | 0.00 | 0,319 (1.5%) | 0,323 (1.5%) | 0.00 |
| Falls ; n (%) | 72 (1.1%) | 85 (1.2%) | -0.01 | 53 (0.4%) | 54 (0.4%) | 0.00 | 125 (0.6%) | 139 (0.6%) | 0.00 |
| Osteoporosis; n (%) | 127 (1.9%) | 137 (2.0%) | -0.01 | 141 (0.9%) | 149 (1.0%) | -0.01 | 0,268 (1.2%) | 0,286 (1.3%) | -0.01 |
| Hyperthyroidism; n (%) | 32 (0.5%) | 34 (0.5%) | 0.00 | 55 (0.4%) | 37 (0.2%) | 0.04 | 87 (0.4%) | 71 (0.3%) | 0.02 |
| Hypothyroidism; n (%) | 653 (9.6%) | 674 (9.9%) | -0.01 | 1,002 (6.6%) | 986 (6.5%) | 0.00 | 1,655 (7.5%) | 1,660 (7.6%) | 0.00 |
| Other disorders of thyroid gland; n (%) | 136 (2.0%) | 131 (1.9%) | 0.01 | 208 (1.4%) | 222 (1.5%) | -0.01 | 0,344 (1.6%) | 0,353 (1.6%) | 0.00 |
| Depression; n (%) | 635 (9.3%) | 631 (9.2%) | 0.00 | 899 (6.0%) | 903 (6.0%) | 0.00 | 1,534 (7.0%) | 1,534 (7.0%) | 0.00 |
| Anxiety; n (%) | 726 (10.6%) | 716 (10.5%) | 0.00 | 988 (6.5%) | 993 (6.6%) | 0.00 | 1,714 (7.8%) | 1,709 (7.8%) | 0.00 |
| Sleep_Disorder; n (%) | 566 (8.3%) | 590 (8.6%) | -0.01 | 1,245 (8.2%) | 1,207 (8.0%) | 0.01 | 1,811 (8.3%) | 1,797 (8.2%) | 0.00 |
| Dementia; n (%) | 21 (0.3%) | 22 (0.3%) | 0.00 | 41 (0.3%) | 38 (0.3%) | 0.00 | 62 (0.3%) | 60 (0.3%) | 0.00 |
| Delirium; n (%) | 19 (0.3%) | 20 (0.3%) | 0.00 | 20 (0.1%) | 23 (0.2%) | -0.03 | 39 (0.2%) | 43 (0.2%) | 0.00 |
| Psychosis; n (%) | 2 (0.0%) | 2 (0.0%) | #DIV/0! | 2 (0.0%) | 2 (0.0%) | #DIV/0! | 4 (0.0%) | 4 (0.0%) | #DIV/0! |
| Obesity; n (%) | 1,558 (22.8%) | 1,593 (23.3%) | -0.01 | 2,340 (15.5%) | 2,314 (15.3%) | 0.01 | 3,898 (17.8%) | 3,907 (17.8%) | 0.00 |
| Overweight; n (%) | 239 (3.5%) | 254 (3.7%) | -0.01 | 274 (1.8%) | 257 (1.7%) | 0.01 | 0,513 (2.3%) | 0,511 (2.3%) | 0.00 |
| Smoking; n (%) | 3,226 (47.2%) | 3,191 (46.7%) | 0.01 | 4,904 (32.5%) | 4,789 (31.7%) | 0.02 | 8,130 (37.1%) | 7,980 (36.4%) | 0.01 |
| Alcohol abuse or dependence; n (%) | 0 (0.0%) | 0 (0.0%) | #DIV/0! | 176 (1.2%) | 169 (1.1%) | 0.01 | 176 (0.8%) | 169 (0.8%) | 0.00 |
| Drug abuse or dependence; n (%) | 1 (0.0%) | 2 (0.0%) | #DIV/0! | 1 (0.0%) | 0 (0.0%) | #DIV/0! | 2 (0.0%) | 2 (0.0%) | #DIV/0! |
| COPD; n (%) | 630 (9.2%) | 673 (9.8%) | -0.02 | 953 (6.3%) | 958 (6.3%) | 0.00 | 1,583 (7.2%) | 1,631 (7.4%) | -0.01 |
| Asthma; n (%) | 391 (5.7%) | 397 (5.8%) | 0.02 | 620 (4.1%) | 616 (4.1%) | 0.00 | 1,011 (4.6%) | 1,013 (4.6%) | 0.00 |
| ' ' ' | 645 (9.4%) | 628 (9.2%) | 0.00 | | | 0.00 | | 1,666 (7.6%) | 0.00 |
| Obstructive sleep apnea; n (%) | , , | , , | -0.02 | 1,057 (7.0%) | 1,038 (6.9%) | -0.01 | 1,702 (7.8%) | 0,594 (2.7%) | -0.01 |
| Pneumonia; n (%) | 210 (3.1%) | 237 (3.5%) | | 328 (2.2%) | 357 (2.4%) | | 0,538 (2.5%) | | |
| Imaging; n (%) | 126 (1.8%) | 132 (1.9%) | -0.01 | 137 (0.9%) | 131 (0.9%) | 0.00 | 263 (1.2%) | 263 (1.2%) | 0.00 |
| Other Medications | 2.740 (5.4.46) | 2 724 (54 504) | 0.00 | 0.447/60.46() | 0.024 (50.004) | 0.01 | 42.025 (50.5%) | 42.755 (50.22() | 0.01 |
| Use of ACE inhibitors; n (%) | 3,718 (54.4%) | 3,724 (54.5%) | 0.00 | 9,117 (60.4%) | 9,031 (59.8%) | 0.01 | 12,835 (58.5%) | 12,755 (58.2%) | 0.01 |
| Use of ARBs; n (%) | 1,134 (16.6%) | 1,169 (17.1%) | -0.01 | 2,308 (15.3%) | 2,326 (15.4%) | 0.00 | 3,442 (15.7%) | 3,495 (15.9%) | -0.01 |
| Use of Loop Diuretics - United; n (%) | 434 (6.3%) | 448 (6.6%) | -0.01 | 690 (4.6%) | 715 (4.7%) | 0.00 | 1,124 (5.1%) | 1,163 (5.3%) | -0.01 |
| Use of other diuretics- United; n (%) | 215 (3.1%) | 249 (3.6%) | -0.03 | 488 (3.2%) | 516 (3.4%) | -0.01 | 0,703 (3.2%) | 0,765 (3.5%) | -0.02 |

Table 1: Prasugrel 10 mg vs Clopidogrel 75 mg

| Use of nitrates-United; n (%) | 3,016 (44.1%) | 2,968 (43.4%) | 0.01 | 6,873 (45.5%) | 6,878 (45.6%) | 0.00 | 9,889 (45.1%) | 9,846 (44.9%) | 0.00 |
|---|---|---|---|---|---|---|---|---|---|
| Use of other hypertension drugs; n (%) | 239 (3.5%) | 270 (4.0%) | -0.03 | 514 (3.4%) | 512 (3.4%) | 0.00 | 0,753 (3.4%) | 0,782 (3.6%) | -0.01 |
| Use of digoxin- United; n (%) | 58 (0.8%) | 49 (0.7%) | 0.01 | 95 (0.6%) | 94 (0.6%) | 0.00 | 153 (0.7%) | 143 (0.7%) | 0.00 |
| Use of Anti-arrhythmics; n (%) | 84 (1.2%) | 88 (1.3%) | -0.01 | 178 (1.2%) | 170 (1.1%) | 0.01 | 262 (1.2%) | 258 (1.2%) | 0.00 |
| Use of COPD/asthma meds- United; n<br>(%) | 737 (10.8%) | 744 (10.9%) | 0.00 | 1,626 (10.8%) | 1,640 (10.9%) | 0.00 | 2,363 (10.8%) | 2,384 (10.9%) | 0.00 |
| Use of statins; n (%) | 6,235 (91.2%) | 6,239 (91.3%) | 0.00 | 13,750 (91.1%) | 13,729 (90.9%) | 0.01 | 19,985 (91.1%) | 19,968 (91.0%) | 0.00 |
| Use of other lipid-lowering drugs; n (%) | 578 (8.5%) | 598 (8.7%) | -0.01 | 1,382 (9.2%) | 1,425 (9.4%) | -0.01 | 1,960 (8.9%) | 2,023 (9.2%) | -0.01 |
| Use of oral anticoagulants (Dabigatran,<br>Rivaroxaban, Apixaban, Warfarin); n (%) | 167 (2.4%) | 171 (2.5%) | -0.01 | 405 (2.7%) | 393 (2.6%) | 0.01 | 0,572 (2.6%) | 0,564 (2.6%) | 0.00 |
| Use of heparin and other low-molecular weight heparins; n (%) | 31 (0.5%) | 29 (0.4%) | 0.01 | 2 (0.0%) | 2 (0.0%) | #DIV/0! | 33 (0.2%) | 31 (0.1%) | 0.03 |
| Use of NSAIDs; n (%) | 868 (12.7%) | 891 (13.0%) | -0.01 | 1,920 (12.7%) | 1,952 (12.9%) | -0.01 | 2,788 (12.7%) | 2,843 (13.0%) | -0.01 |
| Use of oral corticosteroids; n (%) | 936 (13.7%) | 946 (13.8%) | 0.00 | 1,934 (12.8%) | 2,015 (13.3%) | -0.01 | 2,870 (13.1%) | 2,961 (13.5%) | -0.01 |
| Use of bisphosphonate (United); n (%) | 45 (0.7%) | 58 (0.8%) | -0.01 | 72 (0.5%) | 82 (0.5%) | 0.00 | 117 (0.5%) | 140 (0.6%) | -0.01 |
| Use of opioids- United; n (%) | 1,585 (23.2%) | 1,555 (22.8%) | 0.01 | 3,186 (21.1%) | 3,248 (21.5%) | -0.01 | 4,771 (21.8%) | 4,803 (21.9%) | 0.00 |
| Use of antidepressants; n (%) | 1,047 (15.3%) | 1,049 (15.3%) | 0.00 | 2,039 (13.5%) | 2,076 (13.8%) | -0.01 | 3,086 (14.1%) | 3,125 (14.2%) | 0.00 |
| Use of antipsychotics; n (%) | 45 (0.7%) | 44 (0.6%) | 0.01 | 104 (0.7%) | 107 (0.7%) | 0.00 | 0,149 (0.7%) | 0,151 (0.7%) | 0.00 |
| Use of anticonvulsants; n (%) | 503 (7.4%) | 494 (7.2%) | 0.01 | 775 (5.1%) | 783 (5.2%) | 0.00 | 1,278 (5.8%) | 1,277 (5.8%) | 0.00 |
| Use of lithium- United; n (%) | 9 (0.1%) | 7 (0.1%) | 0.00 | 16 (0.1%) | 17 (0.1%) | 0.00 | 25 (0.1%) | 24 (0.1%) | 0.00 |
| Use of Benzos- United; n (%) | 646 (9.5%) | 660 (9.7%) | -0.01 | 1,460 (9.7%) | 1,411 (9.3%) | 0.01 | 2,106 (9.6%) | 2,071 (9.4%) | 0.01 |
| Use of anxiolytics/hypnotics- United; n<br>(%) | 334 (4.9%) | 351 (5.1%) | -0.01 | 798 (5.3%) | 809 (5.4%) | 0.00 | 1,132 (5.2%) | 1,160 (5.3%) | 0.00 |
| Use of dementia meds- United; n (%) | 14 (0.2%) | 14 (0.2%) | 0.00 | 15 (0.1%) | 13 (0.1%) | 0.00 | 29 (0.1%) | 27 (0.1%) | 0.00 |
| Use of antiparkinsonian meds- United;<br>n (%) | 60 (0.9%) | 63 (0.9%) | 0.00 | 122 (0.8%) | 118 (0.8%) | 0.00 | 0,182 (0.8%) | 0,181 (0.8%) | 0.00 |
| Entresto (sacubitril/valsartan); n (%)<br>Labs | 1 (0.0%) | 2 (0.0%) | #DIV/0! | 1 (0.0%) | 2 (0.0%) | #DIV/0! | 2 (0.0%) | 4 (0.0%) | #DIV/0! |
| Lab values- HbA1c (%) ; n (%) | 709 (10.4%) | 663 (9.7%) | 0.02 | 156 (1.0%) | 129 (0.9%) | 0.01 | 0,865 (3.9%) | 0,792 (3.6%) | 0.02 |
| Lab values- HbA1c (%) (within 3<br>months) ; n (%) | 447 (6.5%) | 413 (6.0%) | 0.02 | 105 (0.7%) | 78 (0.5%) | 0.03 | 0,552 (2.5%) | 0,491 (2.2%) | 0.02 |
| Lab values- HbA1c (%) (within 6<br>months) ; n (%) | 709 (10.4%) | 663 (9.7%) | 0.02 | 156 (1.0%) | 129 (0.9%) | 0.01 | 0,865 (3.9%) | 0,792 (3.6%) | 0.02 |
| Lab values- BNP; n (%) | 39 (0.6%) | 31 (0.5%) | 0.01 | 7 (0.0%) | 6 (0.0%) | #DIV/0! | 46 (0.2%) | 37 (0.2%) | 0.00 |
| Lab values- BNP (within 3 months); n<br>(%) | 33 (0.5%) | 26 (0.4%) | 0.01 | 7 (0.0%) | 5 (0.0%) | #DIV/0! | 40 (0.2%) | 31 (0.1%) | 0.03 |
| Lab values- BNP (within 6 months); n<br>(%) | 39 (0.6%) | 31 (0.5%) | 0.01 | 7 (0.0%) | 6 (0.0%) | #DIV/0! | 46 (0.2%) | 37 (0.2%) | 0.00 |
| Lab values- BUN (mg/dl); n (%) | 1,233 (18.0%) | 1,236 (18.1%) | 0.00 | 142 (0.9%) | 143 (0.9%) | 0.00 | 1,375 (6.3%) | 1,379 (6.3%) | 0.00 |
| Lab values- BUN (mg/dl) (within 3 months); n (%) | 769 (11.3%) | 749 (11.0%) | 0.01 | 98 (0.6%) | 94 (0.6%) | 0.00 | 0,867 (4.0%) | 0,843 (3.8%) | 0.01 |
| Lab values- BUN (mg/dl) (within 6<br>months); n (%) | 1,233 (18.0%) | 1,236 (18.1%) | 0.00 | 142 (0.9%) | 143 (0.9%) | 0.00 | 1,375 (6.3%) | 1,379 (6.3%) | 0.00 |
| Lab values- Creatinine (mg/dl); n (%) | 1,265 (18.5%) | 1,267 (18.5%) | 0.00 | 152 (1.0%) | 152 (1.0%) | 0.00 | 1,417 (6.5%) | 1,419 (6.5%) | 0.00 |
| Lab values- Creatinine (mg/dl) (within 3 months); n (%) | 789 (11.5%) | 769 (11.3%) | 0.01 | 103 (0.7%) | 99 (0.7%) | 0.00 | 0,892 (4.1%) | 0,868 (4.0%) | 0.01 |

Table 1: Prasugrel 10 mg vs Clopidogrel 75 mg

| Lab values- Creatinine (mg/dl) (within 6 months); n (%) | 1,265 (18.5%) | 1,267 (18.5%) | 0.00 | 152 (1.0%) | 152 (1.0%) | 0.00 | 1,417 (6.5%) | 1,419 (6.5%) | 0.00 |
|---|---|---|---|---|---|---|---|---|---|
| Lab values- HDL level (mg/dl); n (%) | 1,020 (14.9%) | 1,056 (15.4%) | -0.01 | 154 (1.0%) | 129 (0.9%) | 0.01 | 1,174 (5.4%) | 1,185 (5.4%) | 0.00 |
| Lab values- HDL level (mg/dl) (within 3 | 596 (8.7%) | 620 (9.1%) | -0.01 | 100 (0.7%) | 84 (0.6%) | 0.01 | 0,696 (3.2%) | 0,704 (3.2%) | 0.00 |
| months); n (%) | 330 (8.770) | 020 (3.170) | 0.01 | 100 (0.770) | 04 (0.070) | 0.01 | 0,030 (3.270) | 0,704 (3.270) | 0.00 |
| Lab values- HDL level (mg/dl) (within 6 | 1,020 (14.9%) | 1,056 (15.4%) | -0.01 | 154 (1.0%) | 129 (0.9%) | 0.01 | 1,174 (5.4%) | 1,185 (5.4%) | 0.00 |
| months); n (%) | 2,020 (2576) | 2,000 (2011/0) | 0.01 | 25 . (2.070) | 123 (0.370) | 0.01 | 2)27 . (5.175) | 1)100 (5.170) | 0.00 |
| Lab values- LDL level (mg/dl); n (%) | 1,035 (15.1%) | 1,065 (15.6%) | -0.01 | 163 (1.1%) | 134 (0.9%) | 0.02 | 1,198 (5.5%) | 1,199 (5.5%) | 0.00 |
| Lab values- LDL level (mg/dl) (within 3 | 601 (8.8%) | 622 (9.1%) | -0.01 | 109 (0.7%) | 86 (0.6%) | 0.01 | 0,710 (3.2%) | 0,708 (3.2%) | 0.00 |
| months); n (%) | ( , | (- , | | , | , | | -, - ( , | -, ( , | |
| Lab values- LDL level (mg/dl) (within 6 | 1,035 (15.1%) | 1,065 (15.6%) | -0.01 | 163 (1.1%) | 134 (0.9%) | 0.02 | 1,198 (5.5%) | 1,199 (5.5%) | 0.00 |
| months); n (%) | | | | | | | | | |
| Lab values- NT-proBNP; n (%) | 6 (0.1%) | 7 (0.1%) | 0.00 | 1 (0.0%) | 0 (0.0%) | #DIV/0! | 7 (0.0%) | 7 (0.0%) | #DIV/0! |
| Lab values- NT-proBNP (within 3 | 3 (0.0%) | 6 (0.1%) | -0.04 | 1 (0.0%) | 0 (0.0%) | #DIV/0! | 4 (0.0%) | 6 (0.0%) | #DIV/0! |
| months); n (%) | | | | | | | | | |
| Lab values- NT-proBNP (within 6 | 6 (0.1%) | 7 (0.1%) | 0.00 | 1 (0.0%) | 0 (0.0%) | #DIV/0! | 7 (0.0%) | 7 (0.0%) | #DIV/0! |
| months); n (%) | | | | | | | | | |
| Lab values- Total cholesterol (mg/dl); n<br>(%) | 1,040 (15.2%) | 1,059 (15.5%) | -0.01 | 158 (1.0%) | 130 (0.9%) | 0.01 | 1,198 (5.5%) | 1,189 (5.4%) | 0.00 |
| Lab values-Total cholesterol (mg/dl) | 608 (8.9%) | 617 (9.0%) | 0.00 | 104 (0.7%) | 84 (0.6%) | 0.01 | 0,712 (3.2%) | 0,701 (3.2%) | 0.00 |
| (within 3 months); n (%) | | | | | | | | | |
| Lab values-Total cholesterol (mg/dl) | 1,040 (15.2%) | 1,059 (15.5%) | -0.01 | 158 (1.0%) | 130 (0.9%) | 0.01 | 1,198 (5.5%) | 1,189 (5.4%) | 0.00 |
| (within 6 months); n (%) | | | | | | | | | |
| Lab values- Triglyceride level (mg/dl); n (%) | 1,024 (15.0%) | 1,061 (15.5%) | -0.01 | 149 (1.0%) | 128 (0.8%) | 0.02 | 1,173 (5.3%) | 1,189 (5.4%) | 0.00 |
| Lab values- Triglyceride level (mg/dl) | 596 (8.7%) | 619 (9.1%) | -0.01 | 96 (0.6%) | 83 (0.5%) | 0.01 | 0,692 (3.2%) | 0,702 (3.2%) | 0.00 |
| (within 3 months); n (%) | | | | | | | | | |
| Lab values-Triglyceride level (mg/dl)<br>(within 6 months); n (%) | 1,024 (15.0%) | 1,061 (15.5%) | -0.01 | 149 (1.0%) | 128 (0.8%) | 0.02 | 1,173 (5.3%) | 1,189 (5.4%) | 0.00 |
| Lab result number- HbA1c (%) mean (only 2 to 20 included) | 705 | 659 | | 134 | 117 | | 0 | 0 | |
| mean (sd) | 7.42 (1.91) | 7.18 (1.76) | 0.13 | 8.30 (1.99) | 8.21 (1.99) | 0.05 | 8.03 (1.97) | 7.89 (1.92) | 0.07 |
| median [IQR] | 6.80 [6.00, 8.50] | 6.60 [5.90, 8.00] | 0.11 | 7.80 [6.70, 9.72] | 7.60 [6.85, 9.45] | 0.10 | 7.49 (1.97) | 7.29 (1.92) | 0.10 |
| Missing; n (%) | 6,130 (89.7%) | 6,176 (90.4%) | -0.02 | 14,963 (99.1%) | 14,980 (99.2%) | -0.01 | 21,093 (96.2%) | 21,156 (96.5%) | -0.02 |
| Lab result number- BNP mean | 39 | 31 | | 7 | 6 | | 0 | 0 | |
| mean (sd) | 141.44 (237.21) | 181.63 (295.19) | -0.15 | 149.07 (138.05) | 98.17 (120.28) | 0.39 | 146.69 (175.08) | 124.18 (192.65) | 0.12 |
| median [IQR] | 41.00 [13.00, | 66.10 [31.00, | -0.09 | 113.00 [42.50, | 55.00 [30.75, | 0.45 | 90.56 (175.08) | 58.46 (192.65) | 0.17 |
| | 131.00] | 164.33] | | 178.00] | 161.50] | | | | |
| Missing; n (%) | 6,796 (99.4%) | 6,804 (99.5%) | -0.01 | 15,090 (100.0%) | 15,091 (100.0%) | #DIV/0! | 21,886 (99.8%) | 21,895 (99.8%) | 0.00 |
| Lab result number- BUN (mg/dl) mean | 1,233 | 1,236 | | 142 | 143 | | 0 | 0 | |
| mean (sd) | 16.90 (6.75) | 17.50 (7.03) | -0.09 | 16.04 (4.95) | 1,696.39 | -0.17 | 16.31 (5.57) | 1173.17 | -0.14 |
| | | | | | (14,189.00) | | | (11772.36) | |
| median [IQR] | 16.00 [13.00, 19.00] | 16.00 [13.00, 20.00] | 0.00 | 15.50 [13.00, 18.62] | 16.50 [13.00, 21.00] | 0.00 | 15.66 (5.57) | 16.34 (11772.36) | 0.00 |
| Missing; n (%) | 5,602 (82.0%) | 5,599 (81.9%) | 0.00 | 14,955 (99.1%) | 14,954 (99.1%) | 0.00 | 20,557 (93.7%) | 20,553 (93.7%) | 0.00 |
| Lab result number- Creatinine (mg/dl) | 1,250 | 1,258 | | 145 | 136 | | 1,395 | 1,394 | |
| mean (only 0.1 to 15 included) | | | | | | | | | |
| mean (sd) | 1.01 (0.33) | 1.04 (0.43) | -0.08 | 0.97 (0.26) | 1.06 (0.53) | -0.22 | 0.98 (0.28) | 1.05 (0.50) | -0.17 |
| median [IQR] | 0.96 [0.82, 1.12] | 0.98 [0.83, 1.14] | -0.05 | 0.93 [0.83, 1.04] | 1.00 [0.82, 1.19] | -0.17 | 0.94 (0.28) | 0.99 (0.50) | -0.12 |
| • | • | | | | | | | | |

Table 1: Prasugrel 10 mg vs Clopidogrel 75 mg

| Missing; n (%) Lab result number- HDL level (mg/dl) | 5,585 (81.7%)<br>1,020 | 5,577 (81.6%)<br>1,056 | 0.00 | 14,952 (99.0%)<br>154 | 14,961 (99.1%)<br>127 | -0.01 | 20,537 (93.6%)<br>1,174 | 20,538 (93.6%)<br>1,183 | 0.00 |
|---|---|---|---|---|---|---|---|---|---|
| mean (only =<5000 included)mean (sd) | 44.94 (13.33) | 44.43 (12.73) | 0.04 | 40.24 (12.24) | 41.52 (11.98) | -0.11 | 41.70 (12.59) | 42.43 (12.22) | -0.06 |
| median [IQR] | ` ' | 43.00 [36.00, 51.00] | 0.04 | ` ' | 40.00 [33.00, 47.00] | -0.11<br>-0.11 | 40.02 (12.59) | 40.93 (12.22) | -0.06 |
| median [iQN] | 43.00 [30.00, 31.38] | 43.00 [30.00, 31.00] | 0.00 | 38.07 [32.00, 40.23] | 40.00 [55.00, 47.00] | -0.11 | 40.02 (12.39) | 40.93 (12.22) | -0.07 |
| Missing; n (%) | 5,815 (85.1%) | 5,779 (84.6%) | 0.01 | 14,943 (99.0%) | 14,970 (99.2%) | -0.02 | 20,758 (94.6%) | 20,749 (94.6%) | 0.00 |
| Lab result number- LDL level (mg/dl) | 1,022 | 1,047 | | 148 | 119 | | 1,170 | 1,166 | |
| mean (only =<5000 included) | | | | | | | | | |
| mean (sd) | 109.40 (47.20) | 108.64 (47.27) | 0.02 | 101.12 (49.66) | 99.27 (50.71) | 0.04 | 103.70 (48.91) | 102.19 (49.66) | 0.03 |
| median [IQR] | 107.00 [81.00,<br>138.00] | 110.00 [81.00,<br>136.00] | -0.06 | 100.50 [74.00,<br>134.00] | 100.00 [71.00,<br>134.00] | 0.01 | 102.53 (48.91) | 103.12 (49.66) | -0.01 |
| Missing; n (%) | 5,813 (85.0%) | 5,788 (84.7%) | 0.01 | 14,949 (99.0%) | 14,978 (99.2%) | -0.02 | 20,762 (94.7%) | 20,766 (94.7%) | 0.00 |
| Lab result number-Total cholesterol | 1,039 | 1,057 | | 158 | 128 | | 1,197 | 1,185 | |
| (mg/dl) mean (only =<5000 included) | | | | | | | | | |
| mean (sd) | 195.21 (53.28) | 195.39 (47.33) | 0.00 | 192.59 (52.95) | 191.62 (63.08) | 0.02 | 193.41 (53.05) | 192.79 (58.63) | 0.01 |
| median [IQR] | 190.00 [161.00,<br>222.00] | 192.00 [163.75,<br>224.00] | -0.04 | 192.50 [154.00,<br>224.25] | 187.00 [148.25,<br>223.00] | 0.09 | 191.72 (53.05) | 188.56 (58.63) | 0.06 |
| Missing; n (%) | 5,796 (84.8%) | 5,778 (84.5%) | 0.01 | 14,939 (99.0%) | 14,969 (99.2%) | -0.02 | 20,735 (94.5%) | 20,747 (94.6%) | 0.00 |
| Lab result number-Triglyceride level | 1,023 | 1,061 | | 149 | 126 | | 1,172 | 1,187 | |
| (mg/dl) mean (only =<5000 included) | | | | | | | | | |
| mean (sd) | 182.19 (149.91) | 185.54 (154.25) | -0.02 | 219.48 (160.86) | 215.70 (192.55) | 0.02 | 207.86 (157.53) | 206.30 (181.48) | 0.01 |
| median [IQR] | 147.00 [103.50,<br>216.00] | 149.00 [106.00,<br>214.00] | -0.01 | 184.00 [127.50,<br>248.00] | 162.25 [110.00,<br>232.00] | 0.12 | 172.47 (157.53) | 158.12 (181.48) | 0.08 |
| Missing; n (%) | 5,812 (85.0%) | 5,774 (84.5%) | 0.01 | 14,948 (99.0%) | 14,971 (99.2%) | -0.02 | 20,760 (94.7%) | 20,745 (94.6%) | 0.00 |
| Lab result number- Hemoglobin mean | 920 | 921 | | 100 | 89 | | 1,020 | 1,010 | |
| (only >0 included) | | | | | | | | | |
| mean (sd) | 14.50 (1.64) | 14.57 (1.65) | -0.04 | 1,394.12 | 14.31 (1.39) | 0.14 | 964.17 (11448.42) | 14.39 (1.48) | 0.12 |
| median [IQR] | 14.70 [13.50, 15.60] | 14.70 [13.60, 15.70] | 0.00 | 14.35 [13.20, 15.40] | 14.40 [13.65, 15.20] | 0.00 | 14.46 (11448.42) | 14.49 (1.48) | 0.00 |
| Missing; n (%) | 5,915 (86.5%) | 5,914 (86.5%) | 0.00 | 14,997 (99.3%) | 15,008 (99.4%) | -0.01 | 20,912 (95.3%) | 20,922 (95.4%) | 0.00 |
| Lab result number- Serum sodium | 1,213 | 1,237 | | 143 | 137 | | 1,356 | 1,374 | |
| mean (only > 90 and < 190 included) | | | | | | | | | |
| mean (sd) | 139.71 (2.67) | 139.76 (2.52) | -0.02 | 138.34 (2.60) | 138.76 (2.94) | -0.15 | 138.77 (2.62) | 139.07 (2.82) | -0.11 |
| median [IQR] | 140.00 [138.00,<br>141.00] | 140.00 [138.00,<br>141.00] | 0.00 | 138.40 [137.00,<br>140.00] | 139.00 [137.00,<br>141.00] | -0.22 | 138.90 (2.62) | 139.31 (2.82) | -0.15 |
| Missing; n (%) | 5,622 (82.3%) | 5,598 (81.9%) | 0.01 | 14,954 (99.1%) | 14,960 (99.1%) | 0.00 | 20,576 (93.8%) | 20,558 (93.7%) | 0.00 |
| Lab result number- Albumin mean (only >0 and <=10 included) | 1,136 | 1,167 | | 123 | 114 | | 1,259 | 1,281 | |
| mean (sd) | 4.29 (0.32) | 4.28 (0.32) | 0.03 | 4.18 (0.50) | 4.13 (0.53) | 0.10 | 4.21 (0.45) | 4.18 (0.47) | 0.07 |
| median [IQR] | 4.30 [4.10, 4.50] | 4.30 [4.10, 4.50] | 0.00 | 4.20 [4.00, 4.40] | 4.20 [4.00, 4.40] | 0.00 | 4.23 (0.45) | 4.23 (0.47) | 0.00 |
| Missing; n (%) | 5,699 (83.4%) | 5,668 (82.9%) | 0.01 | 14,974 (99.2%) | 14,983 (99.2%) | 0.00 | 20,673 (94.3%) | 20,651 (94.2%) | 0.00 |
| Lab result number- Glucose (fasting or random) mean (only 10-1000 included) | 1,198 | 1,230 | | 132 | 131 | | 1,330 | 1,361 | |
| mean (sd) | 128.66 (60.29) | 120.80 (51.79) | 0.14 | 171.15 (68.93) | 165.87 (78.57) | 0.07 | 157.91 (66.36) | 151.82 (71.31) | 0.09 |
| median [IQR] | 105.00 [92.50, | 103.00 [92.50, | 0.04 | 149.00 [118.25, | 144.00 [110.00, | 0.07 | 135.29 (66.36) | 131.22 (71.31) | 0.06 |
| | 141.00] | 129.25] | | 218.12] | 190.00] | | (00.00) | (, 2.02) | |

Table 1: Prasugrel 10 mg vs Clopidogrel 75 mg

| Missing; n (%) | 5,637 (82.5%) | 5,605 (82.0%) | 0.01 | 14,965 (99.1%) | 14,966 (99.1%) | 0.00 | 20,602 (93.9%) | 20,571 (93.8%) | 0.00 |
|---|---|---|---|---|---|---|---|---|---|
| Lab result number-Potassium mean | 1,240 | 1,265 | | 141 | 140 | | 1,381 | 1,405 | |
| (only 1-7 included) | | | | | | | | | |
| mean (sd) | 4.38 (0.42) | 4.40 (0.42) | -0.05 | 4.30 (0.43) | 4.31 (0.48) | -0.02 | 4.32 (0.43) | 4.34 (0.46) | -0.04 |
| median [IQR] | 4.40 [4.10, 4.60] | 4.40 [4.10, 4.70] | 0.00 | 4.30 [4.00, 4.59] | 4.30 [4.00, 4.67] | 0.00 | 4.33 (0.43) | 4.33 (0.46) | 0.00 |
| Missing; n (%) | 5,595 (81.9%) | 5,570 (81.5%) | 0.01 | 14,956 (99.1%) | 14,957 (99.1%) | 0.00 | 20,551 (93.7%) | 20,527 (93.6%) | 0.00 |
| Comorbidity Scores | | | | | | | | | |
| CCI (180 days)- ICD9 and ICD10 | | | | | | | | | |
| mean (sd) | 2.17 (1.78) | 2.20 (1.82) | -0.02 | 1.60 (1.45) | 1.61 (1.43) | -0.01 | 1.78 (1.56) | 1.79 (1.56) | -0.01 |
| median [IQR] | 2.00 [1.00, 3.00] | 2.00 [1.00, 3.00] | 0.00 | 1.00 [1.00, 2.00] | 1.00 [1.00, 2.00] | 0.00 | 1.31 (1.56) | 1.31 (1.56) | 0.00 |
| Frailty Score (mean): Empirical Version | | | | | | | | | |
| 365 days, | | | | | | | | | |
| mean (sd) | 0.17 (0.04) | 0.17 (0.04) | 0.00 | 0.16 (0.03) | 0.16 (0.03) | 0.00 | 0.16 (0.03) | 0.16 (0.03) | 0.00 |
| median [IQR] | 0.17 [0.15, 0.19] | 0.17 [0.15, 0.19] | 0.00 | 0.16 [0.14, 0.18] | 0.16 [0.14, 0.18] | 0.00 | 0.16 (0.03) | 0.16 (0.03) | 0.00 |
| Healthcare Utilization | | | | | | | | | |
| Any hospitalization; n (%) | 6,832 (100.0%) | 6,834 (100.0%) | #DIV/0! | 15,097 (100.0%) | 15,096 (100.0%) | #DIV/0! | 21,929 (100.0%) | 21,930 (100.0%) | #DIV/0! |
| Any hospitalization during prior 31-<br>180 days; n (%) | 178 (2.6%) | 210 (3.1%) | -0.03 | 278 (1.8%) | 351 (2.3%) | -0.04 | 0,456 (2.1%) | 0,561 (2.6%) | -0.03 |
| Endocrinologist Visit; n (%) | 319 (4.7%) | 323 (4.7%) | 0.00 | 500 (3.3%) | 556 (3.7%) | -0.02 | 0,819 (3.7%) | 0,879 (4.0%) | -0.02 |
| Endocrinologist Visit, (30 days prior); n | 151 (2.2%) | 173 (2.5%) | -0.02 | 275 (1.8%) | 315 (2.1%) | -0.02 | 0,426 (1.9%) | 0,488 (2.2%) | -0.02 |
| (%) | | | | | | | | | |
| Endocrinologist Visit (31 to 180 days prior); n (%) | 221 (3.2%) | 191 (2.8%) | 0.02 | 287 (1.9%) | 339 (2.2%) | -0.02 | 0,508 (2.3%) | 0,530 (2.4%) | -0.01 |
| Internal medicine/family medicine | 4,888 (71.5%) | 4,835 (70.7%) | 0.02 | 9,379 (62.1%) | 9,434 (62.5%) | -0.01 | 14,267 (65.1%) | 14,269 (65.1%) | 0.00 |
| visits; n (%) | , | , ( , | | -, ( , | -, - (, | | , - ( , | , ( , | |
| Internal medicine/family medicine | 4,019 (58.8%) | 3,918 (57.3%) | 0.03 | 5,587 (37.0%) | 5,685 (37.7%) | -0.01 | 9,606 (43.8%) | 9,603 (43.8%) | 0.00 |
| visits (30 days prior) ; n (%) | , , | | | | | | | | |
| Internal medicine/family medicine | 3,008 (44.0%) | 3,037 (44.4%) | -0.01 | 7,347 (48.7%) | 7,389 (48.9%) | 0.00 | 10,355 (47.2%) | 10,426 (47.5%) | -0.01 |
| visits (31 to 180 days prior); n (%) | | | | | | | | | |
| Cardiologist visit; n (%) | 6,637 (97.1%) | 6,586 (96.4%) | 0.04 | 4,991 (33.1%) | 4,966 (32.9%) | 0.00 | 11,628 (53.0%) | 11,552 (52.7%) | 0.01 |
| Number of Cardiologist visits (30 days | 6,615 (96.8%) | 6,567 (96.1%) | 0.04 | 4,217 (27.9%) | 4,234 (28.0%) | 0.00 | 10,832 (49.4%) | 10,801 (49.2%) | 0.00 |
| prior); n (%) | | | | | | | | | |
| Number of Cardiologist visits (31 to | 951 (13.9%) | 910 (13.3%) | 0.02 | 1,343 (8.9%) | 1,297 (8.6%) | 0.01 | 2,294 (10.5%) | 2,207 (10.1%) | 0.01 |
| 180 days prior); n (%) | | | | | | | | | |
| Electrocardiogram ; n (%) | 6,232 (91.2%) | 6,308 (92.3%) | -0.04 | 8,331 (55.2%) | 8,225 (54.5%) | 0.01 | 14,563 (66.4%) | 14,533 (66.3%) | 0.00 |
| Use of glucose test strips; n (%) | 73 (1.1%) | 67 (1.0%) | 0.01 | 140 (0.9%) | 157 (1.0%) | -0.01 | 0,213 (1.0%) | 0,224 (1.0%) | 0.00 |
| Dialysis; n (%) | 22 (0.3%) | 27 (0.4%) | -0.02 | 31 (0.2%) | 20 (0.1%) | 0.03 | 53 (0.2%) | 47 (0.2%) | 0.00 |
| number of different/distinct | | | | | | | | | |
| medication prescriptions | | | | | | | | | |
| mean (sd) | 8.41 (4.29) | 8.41 (4.40) | 0.00 | 8.17 (4.00) | 8.21 (4.09) | -0.01 | 8.24 (4.09) | 8.27 (4.19) | -0.01 |
| median [IQR] | 7.00 [5.00, 11.00] | 7.00 [5.00, 11.00] | 0.00 | 7.00 [5.00, 10.00] | 7.00 [5.00, 10.00] | 0.00 | 7.00 (4.09) | 7.00 (4.19) | 0.00 |
| Number of Hospitalizations | | | | | | | | | |
| mean (sd) | 1.08 (0.30) | 1.09 (0.31) | -0.03 | 1.07 (0.27) | 1.07 (0.28) | 0.00 | 1.07 (0.28) | 1.08 (0.29) | -0.04 |
| median [IQR] | 1.00 [1.00, 1.00] | 1.00 [1.00, 1.00] | 0.00 | 1.00 [1.00, 1.00] | 1.00 [1.00, 1.00] | 0.00 | 1.00 (0.28) | 1.00 (0.29) | 0.00 |
| Number of hospital days | | | | | | | | | |
| mean (sd) | 3.68 (2.09) | 3.71 (2.08) | -0.01 | 3.60 (2.07) | 3.60 (1.70) | 0.00 | 3.62 (2.08) | 3.63 (1.83) | -0.01 |
| median [IQR] | 3.00 [3.00, 4.00] | 3.00 [3.00, 4.00] | 0.00 | 3.00 [3.00, 4.00] | 3.00 [3.00, 4.00] | 0.00 | 3.00 (2.08) | 3.00 (1.83) | 0.00 |

Table 1: Prasugrel 10 mg vs Clopidogrel 75 mg

| visits mean (sd) 0.90 (1.06) 0.88 (1.13) 0.02 3.16 (5.52) 3.10 (5.67) 0.01 2.46 (4.62) 2.41 (4.75) median [lQR] 1.00 [0.00, 1.00] 1.00 [0.00, 1.00] 0.00 2.00 [0.00, 4.00] 2.00 [0.00, 4.00] 0.00 1.69 (4.62) 1.69 (4.75) Number of Office visits mean (sd) 2.95 (3.25) 2.94 (3.25) 0.00 2.59 (2.99) 2.64 (3.14) -0.02 2.70 (3.07) 2.73 (3.17) median [lQR] 2.00 [1.00, 4.00] 2.00 [1.00, 4.00] 0.00 [1.00, 4.00] 0.00 [1.00, 4.00] 0.00 [0.00, | 0.01<br>0.00<br>-0.01<br>0.00<br>-0.02<br>0.00<br>-0.10 |
|---|---|
| median [IQR] | 0.00<br>-0.01<br>0.00<br>-0.02<br>0.00 |
| Number of Office visitsmean (sd)median [IQR] Number of Endocrinologist visitsmean (sd) 0.21 (1.56) 0.19 (1.21) 0.00 [0.00, 0.00] 0.00 [0.00, 0 | -0.01<br>0.00<br>-0.02<br>0.00 |
| mean (sd) 2.95 (3.25) 2.94 (3.25) 0.00 2.59 (2.99) 2.64 (3.14) -0.02 2.70 (3.07) 2.73 (3.17) 2.00 [1.00, 4.00] 2.00 [1.00, 4.00] 0.00 2.00 [1.00, 4.00] 0.00 2.00 [1.00, 4.00] 0.00 2.00 (3.07) 2.00 (3.17) 2.00 [1.00, 4.00] 0.00 2.00 [1.00, 4.00] 0.00 2.00 [1.00, 4.00] 0.00 2.00 (3.07) 2.00 (3.17) 2.00 [3.17] 2.00 [ | 0.00<br>-0.02<br>0.00 |
| median [IQR] 2.00 [1.00, 4.00] 2.00 [1.00, 4.00] 0.00 2.00 [1.00, 4.00] 0.00 2.00 [3.07] 2.00 (3.17) Number of Endocrinologist visitsmean (sd) 0.21 (1.56) 0.19 (1.21) 0.01 0.14 (1.09) 0.18 (1.30) -0.03 0.38 (1.08) 0.40 (1.25) Number of internal medicine/family medicine visitsmean (sd) 5.36 (9.27) 5.39 (9.09) 0.00 3.48 (6.29) 3.51 (6.05) 0.00 4.07 (7.35) 4.10 (7.14)median [IQR] 3.00 [0.00, 7.00] 3.00 [0.00, 7.00] 0.00 1.00 [0.00, 5.00] 2.00 [0.00, 5.00] -0.16 1.62 (7.35) 2.31 (7.14) Number of Cardiologist visitsmean (sd) 9.25 (5.74) 9.28 (5.43) -0.01 1.02 (2.32) 1.03 (2.35) 0.00 3.58 (3.74) 3.60 (3.60) | 0.00<br>-0.02<br>0.00 |
| Number of Endocrinologist visitsmean (sd)median [IQR] Number of internal medicine/family medicine visitsmean (sd)mean (sd)mean (sd) 0.00 [0.00, 0.00] 0.00 | -0.02<br>0.00 |
| median [IQR] Number of internal medicine/family medicine visitsmedian [IQR] Number of Cardiologist visitsmean (sd) 0.21 (1.56) 0.19 (1.21) 0.01 0.00 [0.00, 0.00] 0 | 0.00 |
| median [IQR] 0.00 [0.00, 0.00] 0.00 0.31 (1.08) 0.31 (1.25) 0.00 0.00 [0.00, 0.00] 0.00 [0.00, 0.00] 0.00 0.00 [0.00, 0.00] 0.00 0.31 (1.08) 0.31 (1.25) 0.00 0.00 0.00 [0.00, 0.00] 0.00 0.00 [0.00, 0.00] 0.00 0.00 [0.00, 0.00] 0.00 0.31 (1.08) 0.31 (1.25) 0.31 (1.25) 0.00 0.31 (1.08) 0.31 (1.25) 0.31 ( | 0.00 |
| Number of internal medicine/family medicine visitsmean (sd)median [IQR] Number of Cardiologist visitsmean (sd) 9.25 (5.74) 9.28 (5.43) 5.39 (9.09) 0.00 3.48 (6.29) 3.51 (6.05) 0.00 4.07 (7.35) 4.10 (7.14) 2.00 [0.00, 5.00] 2.00 [0.00, 5.00] 2.00 [0.00, 5.00] 3.58 (3.74) 3.60 (3.60) | 0.00 |
| medicine visits 5.36 (9.27) 5.39 (9.09) 0.00 3.48 (6.29) 3.51 (6.05) 0.00 4.07 (7.35) 4.10 (7.14) median [IQR] 3.00 [0.00, 7.00] 3.00 [0.00, 7.00] 0.00 1.00 [0.00, 5.00] 2.00 [0.00, 5.00] -0.16 1.62 (7.35) 2.31 (7.14) Number of Cardiologist visits mean (sd) 9.25 (5.74) 9.28 (5.43) -0.01 1.02 (2.32) 1.03 (2.35) 0.00 3.58 (3.74) 3.60 (3.60) | |
| mean (sd) 5.36 (9.27) 5.39 (9.09) 0.00 3.48 (6.29) 3.51 (6.05) 0.00 4.07 (7.35) 4.10 (7.14)median [IQR] 3.00 [0.00, 7.00] 3.00 [0.00, 7.00] 0.00 1.00 [0.00, 5.00] 2.00 [0.00, 5.00] -0.16 1.62 (7.35) 2.31 (7.14) Number of Cardiologist visitsmean (sd) 9.25 (5.74) 9.28 (5.43) -0.01 1.02 (2.32) 1.03 (2.35) 0.00 3.58 (3.74) 3.60 (3.60) | |
| median [IQR] 3.00 [0.00, 7.00] 3.00 [0.00, 7.00] 0.00 1.00 [0.00, 5.00] 2.00 [0.00, 5.00] -0.16 1.62 (7.35) 2.31 (7.14) Number of Cardiologist visitsmean (sd) 9.25 (5.74) 9.28 (5.43) -0.01 1.02 (2.32) 1.03 (2.35) 0.00 3.58 (3.74) 3.60 (3.60) | |
| Number of Cardiologist visitsmean (sd) 9.25 (5.74) 9.28 (5.43) -0.01 1.02 (2.32) 1.03 (2.35) 0.00 3.58 (3.74) 3.60 (3.60) | -0.10 |
| mean (sd) 9.25 (5.74) 9.28 (5.43) -0.01 1.02 (2.32) 1.03 (2.35) 0.00 3.58 (3.74) 3.60 (3.60) | |
| median [IQR] 8.00 [6.00, 12.00] 8.00 [6.00, 12.00] 0.00 0.00 [0.00, 1.00] 0.00 [0.00, 1.00] 0.00 2.49 (3.74) 2.49 (3.60) | -0.01 |
| | 0.00 |
| Number electrocardiograms received | |
| mean (sd) 3.18 (2.35) 3.19 (2.39) 0.00 1.05 (1.36) 1.05 (1.41) 0.00 1.71 (1.73) 1.72 (1.77) | -0.01 |
| median [IQR] 3.00 [1.00, 4.00] 3.00 [1.00, 4.00] 0.00 1.00 [0.00, 2.00] 1.00 [0.00, 2.00] 0.00 1.62 (1.73) 1.62 (1.77) | 0.00 |
| Number of HbA1c tests ordered | |
| mean (sd) 0.30 (0.64) 0.31 (0.63) -0.02 0.23 (0.55) 0.23 (0.55) 0.00 0.25 (0.58) 0.25 (0.58) | 0.00 |
| median [IQR] 0.00 [0.00, 0.00] 0.00 [0.00, 0.00] 0.00 [0.00, 0.00] 0.00 [0.00, 0.00] 0.00 (0.58) | 0.00 |
| Number of glucose tests ordered | 0.00 |
| mean (sd) 0.13 (0.63) 0.15 (1.08) -0.02 0.11 (0.51) 0.12 (0.59) -0.02 0.12 (0.55) 0.13 (0.78) | -0.01 |
| median [IQR] 0.00 [0.00, 0.00] 0.00 [0.00, 0.00] 0.00 [0.00, 0.00] 0.00 [0.00, 0.00] 0.00 (0.55) 0.00 (0.78) | 0.00 |
| Number of lipid tests ordered | 0.00 |
| | 0.00 |
| | 0.00 |
| | 0.00 |
| Number of creatinine tests ordered 0.03 (0.35) 0.04 (0.34) 0.05 (0.33) 0.04 (0.34) 0.04 (0.34) | 0.00 |
| mean (sd) 0.03 (0.25) 0.03 (0.24) 0.00 0.05 (0.32) 0.04 (0.34) 0.03 0.04 (0.30) 0.04 (0.31) | 0.00 |
| median [IQR] 0.00 [0.00, 0.00] 0.00 [0.00, 0.00] 0.00 [0.00, 0.00] 0.00 [0.00, 0.00] 0.00 [0.00, 0.00] 0.00 (0.31) | 0.00 |
| Number of BUN tests ordered | 0.00 |
| mean (sd) 0.02 (0.16) 0.02 (0.38) 0.00 0.03 (0.26) 0.03 (0.25) 0.00 0.03 (0.23) 0.03 (0.30) | 0.00 |
| median [IQR] 0.00 [0.00, 0.00] 0.00 [0.00, 0.00] 0.00 [0.00, 0.00] 0.00 [0.00, 0.00] 0.00 [0.00, 0.00] 0.00 (0.23) 0.00 (0.30) | 0.00 |
| Number of tests for microalbuminuria | |
| mean (sd) 0.16 (0.57) 0.17 (0.62) -0.02 0.11 (0.48) 0.12 (0.49) -0.02 0.13 (0.51) 0.14 (0.53) | -0.02 |
| median [IQR] 0.00 [0.00, 0.00] 0.00 [0.00, 0.00] 0.00 [0.00, 0.00] 0.00 [0.00, 0.00] 0.00 (0.51) 0.00 (0.53) | 0.00 |
| Total N distinct ICD9/ICD10 diagnoses | |
| at the 3rd digit level | |
| mean (sd) 5.70 (8.02) 5.68 (8.21) 0.00 3.49 (6.39) 3.53 (6.48) -0.01 4.18 (6.94) 4.20 (7.06) | 0.00 |
| median [IQR] 0.00 [0.00, 10.00] 0.00 [0.00, 9.00] 0.00 0.00 [0.00, 4.00] 0.00 [0.00, 4.00] 0.00 (6.94) 0.00 (7.06) | 0.00 |
| For PS | |
| Hemorrhagic stroke+Other 52 (0.8%) 44 (0.6%) 0.02 47 (0.3%) 47 (0.3%) 0.00 99 (0.5%) 91 (0.4%) | 0.01 |
| cerebrovascular | |
| disease+Cerebrovascular procedure (for | |
| PS); n (%) | |

Table 1: Prasugrel 10 mg vs Clopidogrel 75 mg

| Occurrence of creatinine tests ordered (for PS); n (%) | 178 (2.6%) | 160 (2.3%) | 0.02 | 479 (3.2%) | 466 (3.1%) | 0.01 | 0,657 (3.0%) | 0,626 (2.9%) | 0.01 | |
|---|---|---|---|---|---|---|---|---|---|---|
| Occurrence of BUN tests ordered (for | 92 (1.3%) | 85 (1.2%) | 0.01 | 290 (1.9%) | 310 (2.1%) | -0.01 | 0,382 (1.7%) | 0,395 (1.8%) | -0.01 | |
| PS); n (%) | / | () | | | () | | / | | | |
| Occurrence of chronic renal | 298 (4.4%) | 320 (4.7%) | -0.01 | 304 (2.0%) | 298 (2.0%) | 0.00 | 0,602 (2.7%) | 0,618 (2.8%) | -0.01 | |
| insufficiency w/o CKD (for PS); n (%) | 02 (4. 20/) | 05 (4.20() | 0.00 | 404(0.70() | 400 (0.70/) | 0.00 | 407 (0.00() | 405 (0.00() | 0.04 | |
| Chronic kidney disease Stage 1-2 (for PS); n (%) | 83 (1.2%) | 85 (1.2%) | 0.00 | 104 (0.7%) | 100 (0.7%) | 0.00 | 187 (0.9%) | 185 (0.8%) | 0.01 | |
| Chronic kidney disease Stage 3-6 (for PS); n (%) | 306 (4.5%) | 322 (4.7%) | -0.01 | 298 (2.0%) | 309 (2.0%) | 0.00 | 0,604 (2.8%) | 0,631 (2.9%) | -0.01 | |
| Bladder stones+Kidney stones (for PS); n (%) | 140 (2.0%) | 148 (2.2%) | -0.01 | 274 (1.8%) | 260 (1.7%) | 0.01 | 0,414 (1.9%) | 0,408 (1.9%) | 0.00 | |
| Diabetes with peripheral circulatory disorders+Gangrene+Osteomyelitis(for PS) with ICD10; n (%) | 124 (1.8%) | 115 (1.7%) | 0.01 | 146 (1.0%) | 142 (0.9%) | 0.01 | 0,270 (1.2%) | 0,257 (1.2%) | 0.00 | |
| Alcohol abuse or dependence+Drug abuse or dependence (for PS); n (%) | 1 (0.0%) | 2 (0.0%) | #DIV/0! | 177 (1.2%) | 169 (1.1%) | 0.01 | 178 (0.8%) | 171 (0.8%) | 0.00 | |
| Diabetes with other ophthalmic manifestations+Retinal detachment, | 17 (0.2%) | 18 (0.3%) | -0.02 | 112 (0.7%) | 128 (0.8%) | -0.01 | 0,129 (0.6%) | 0,146 (0.7%) | -0.01 | |
| vitreous hemorrhage,<br>vitrectomy+Retinal laser coagulation<br>therapy (for PS); n (%) | | | | | | | | | | |
| Other atherosclerosis+Cardiac<br>conduction disorders+Other CVD (for<br>PS); n (%) | 2,350 (34.4%) | 2,362 (34.6%) | 0.00 | 3,918 (26.0%) | 3,941 (26.1%) | 0.00 | 6,268 (28.6%) | 6,303 (28.7%) | 0.00 | |
| Previous cardiac procedure (CABG or<br>PTCA or Stent) + History of CABG or<br>PTCA (for PS) ; n (%) | 6,773 (99.1%) | 6,772 (99.1%) | 0.00 | 14,900 (98.7%) | 14,889 (98.6%) | 0.01 | 21,673 (98.8%) | 21,661 (98.8%) | 0.00 | |
| Hyperthyroidism + Hypothyroidism +<br>Other disorders of thyroid gland (for<br>PS); n (%) | 739 (10.8%) | 750 (11.0%) | -0.01 | 1,153 (7.6%) | 1,132 (7.5%) | 0.00 | 1,892 (8.6%) | 1,882 (8.6%) | 0.00 | |
| Delirium + Psychosis (for PS); n (%) | 20 (0.3%) | 22 (0.3%) | 0.00 | 22 (0.1%) | 25 (0.2%) | -0.03 | 42 (0.2%) | 47 (0.2%) | 0.00 | |
| Any use of Meglitinides (for PS); n (%) | 11 (0.2%) | 16 (0.2%) | 0.00 | 36 (0.2%) | 37 (0.2%) | 0.00 | 47 (0.2%) | 53 (0.2%) | 0.00 | |
| Any use of AGIs (for PS); n (%) | 2 (0.0%) | 3 (0.0%) | #DIV/0! | 3,918 (26.0%) | 3,941 (26.1%) | 0.00 | 6,268 (28.6%) | 6,303 (28.7%) | 0.00 | |
| CKD stage 3-6 + dialysis (for PS); n (%) | 308 (4.5%) | 323 (4.7%) | -0.01 | 299 (2.0%) | 311 (2.1%) | -0.01 | 0,607 (2.8%) | 0,634 (2.9%) | -0.01 | |
| Use of thiazide; n (%) | 490 (7.2%) | 459 (6.7%) | 0.02 | 896 (5.9%) | 910 (6.0%) | 0.00 | 19,435 (88.6%) | 19,440 (88.6%) | 0.00 | |
| Use of beta blockers; n (%) | 5,945 (87.0%) | 5,953 (87.1%) | 0.00 | 13,490 (89.4%) | 13,487 (89.3%) | 0.00 | 3,472 (15.8%) | 3,490 (15.9%) | 0.00 | |
| Use of calcium channel blockers; n (%) | 1,164 (17.0%) | 1,160 (17.0%) | 0.00 | 2,308 (15.3%) | 2,330 (15.4%) | 0.00 | 4,161 (19.0%) | 4,142 (18.9%) | 0.00 | |
| All antidiabetic medications except Insulin; n (%) | 1,371 (20.1%) | 1,377 (20.1%) | 0.00 | 2,790 (18.5%) | 2,765 (18.3%) | 0.01 | 1,386 (6.3%) | 1,369 (6.2%) | 0.00 | |
| DM Medications - Insulin ; n (%) | 615 (9.0%) | 614 (9.0%) | 0.00 | 1,082 (7.2%) | 1,116 (7.4%) | -0.01 | 1,697 (7.7%) | 1,730 (7.9%) | -0.01 | |
| Use of Low Intensity Statins; n (%) | 2,279 (33.3%) | 2,243 (32.8%) | 0.01 | 5,230 (34.6%) | 5,227 (34.6%) | 0.00 | 7509 (34.2%) | 7,470 (34.1%) | 0.00 | 1 |
| Use of High Intensity Statins; n (%) | 4,447 (65.1%) | 4,598 (67.3%) | -0.05 | 9,372 (62.1%) | 9,575 (63.4%) | -0.03 | 13819 (63.0%) | 14,173 (64.6%) | -0.03 | 1 |
| Malignant hypertension; n (%) | 296 (4.3%) | 300 (4.4%) | 0.00 | 7,481 (49.6%) | 7,421 (49.2%) | 0.01 | 7777 (35.5%) | 7,721 (35.2%) | 0.01 | ĺ |
| Cardiovascular stress test; n (%) | 7 (0.1%) | 7 (0.1%) | 0.00 | 16 (0.1%) | 21 (0.1%) | 0.00 | 0,023 (0.1%) | 28 (0.1%) | 0.00 | ĺ |
| Echocardiogram; n (%) | 4,528 (66.2%) | 4,503 (65.9%) | 0.00 | 9,338 (61.9%) | 9,391 (62.2%) | -0.01 | 13,866 (63.2%) | 13894 (63.4%) | 0.00 | 1 |
| Number of BNP tests | 7,320 (00.270) | T,505 (05.570) | 0.01 | J,JJU (UI.J/0) | J,JJ± (UZ.Z/U) | 0.01 | 13,000 (03.2/0) | 13037 (03.470) | 0.00 | 1 |
| | | | | | | | | | | 1 |
| mean (sd) | 0.06 (0.32) | 0.06 (0.29) | 0.00 | 0.12 (0.37) | 0.12 (0.37) | 0.00 | 0.10 (0.36) | 0.10 (0.35) | 0.00 | |

Table 1: Prasugrel 10 mg vs Clopidogrel 75 mg

| median [IQR] | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 | 0.00 (0.36) | 0.00 (0.35) | 0.00 |
|---|---|---|---|---|---|---|---|---|---|
| Number of Cardiac biomarkers tests | | | | | | | | | |
| (tropnin, CK-MBs, Myoglobin, CPK) | | | | | | | | | |
| mean (sd) | 0.41 (1.47) | 0.42 (1.70) | -0.01 | 0.79 (1.65) | 0.80 (1.74) | -0.01 | 0.67 (1.60) | 0.68 (1.73) | -0.01 |
| median [IQR] | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 | 0.00 [0.00, 1.00] | 0.00 [0.00, 1.00] | 0.00 | 0.00 (1.60) | 0.00 (1.73) | 0.00 |
| Number of Ambulatory Blood pressure | | | | | | | | | |
| monitoring tests | | | | | | | | | |
| mean (sd) | 0.00 (0.02) | 0.00 (0.02) | 0.00 | 0.00 (0.03) | 0.00 (0.02) | 0.00 | 0.00 (0.03) | 0.00 (0.02) | 0.00 |
| median [IQR] | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 | 0.00 (0.03) | 0.00 (0.02) | 0.00 |
| N of days on antihypertensive | | | | | | | | | |
| medications during baseline | | | | | | | | | |
| mean (sd) | 67.42 (76.28) | 67.51 (76.88) | 0.00 | 62.89 (75.36) | 62.70 (75.54) | 0.00 | 64.30 (75.65) | 64.20 (75.96) | 0.00 |
| median [IQR] | 7.00 [1.00, 158.00] | 7.00 [1.00, 161.00] | 0.00 | 1.00 [1.00, 152.00] | 2.00 [1.00, 153.00] | -0.01 | 2.87 (75.65) | 3.56 (75.96) | -0.01 |
| N of days in database anytime prior | | | | | | | | | |
| mean (sd) | 1,616.01 (1,214.94) | 1,629.92 (1,231.27) | -0.01 | 1,708.25 (1,223.37) | 1,713.51 (1,215.39) | 0.00 | 1679.50 (1220.75) | 1687.46 (1220.36) | -0.01 |
| median [IQR] | 1,302.00 [622.00, | 1,298.00 [631.00, | 0.00 | 1,365.00 [681.00, | 1,375.00 [702.00, | -0.01 | 1345.37 (1220.75) | 1351.00 (1220.36) | 0.00 |
| | 2,331.00] | 2,369.00] | | 2,602.50] | 2,609.00] | | | | |
| Mean Copay for per prescription cost | | | | | | | | | |
| (charges in U.S. \$) (180-1 day prior) | | | | | | | | | |
| mean (sd) | 24.78 (29.15) | 25.15 (27.70) | -0.01 | 19.46 (24.18) | 19.56 (23.85) | 0.00 | 21.12 (25.83) | 21.30 (25.11) | -0.01 |
| median [IQR] | 17.32 [6.94, 33.33] | 17.92 [8.00, 33.33] | -0.02 | 13.33 [4.62, 26.99] | 13.25 [5.00, 26.42] | 0.00 | 14.57 (25.83) | 14.71 (25.11) | -0.01 |
| Missing; n (%) | 1,195 (17.5%) | 1,189 (17.4%) | 0.00 | 2,793 (18.5%) | 2,751 (18.2%) | 0.01 | 3,988 (18.2%) | 3940 (18.0%) | 0.01 |
| Colonos; n (%) | 233 (3.4%) | 218 (3.2%) | 0.01 | 476 (3.2%) | 473 (3.1%) | 0.01 | 0,709 (3.2%) | 691 (3.2%) | 0.00 |
| Fecal occult blood (FOB) test; n (%) | 215 (3.1%) | 216 (3.2%) | -0.01 | 432 (2.9%) | 404 (2.7%) | 0.01 | 0,647 (3.0%) | 620 (2.8%) | 0.01 |
| Flu vaccine; n (%) | 784 (11.5%) | 787 (11.5%) | 0.00 | 1,142 (7.6%) | 1,140 (7.6%) | 0.00 | 1,926 (8.8%) | 1927 (8.8%) | 0.00 |
| Mammogram; n (%) | 323 (4.7%) | 309 (4.5%) | 0.01 | 546 (3.6%) | 540 (3.6%) | 0.00 | 0,869 (4.0%) | 849 (3.9%) | 0.01 |
| Pap smear; n (%) | 141 (2.1%) | 138 (2.0%) | 0.01 | 362 (2.4%) | 347 (2.3%) | 0.01 | 0,503 (2.3%) | 485 (2.2%) | 0.01 |
| Pneumonia vaccine; n (%) | 716 (10.5%) | 723 (10.6%) | 0.00 | 678 (4.5%) | 649 (4.3%) | 0.01 | 1,394 (6.4%) | 1372 (6.3%) | 0.00 |
| PSA test or Prostate exam for DRE; n (%) | 1,042 (15.2%) | 1,040 (15.2%) | 0.00 | 2,105 (13.9%) | 2,048 (13.6%) | 0.01 | 3,147 (14.3%) | 3088 (14.1%) | 0.01 |
| Bone mineral density; n (%) | 107 (1.6%) | 105 (1.5%) | 0.01 | 119 (0.8%) | 103 (0.7%) | 0.01 | 0,226 (1.0%) | 208 (0.9%) | 0.01 |
| Use of Sympatomimetic agents; n (%) | 73 (1.1%) | 70 (1.0%) | 0.01 | 170 (1.1%) | 183 (1.2%) | -0.01 | 0,243 (1.1%) | 253 (1.2%) | -0.01 |
| Use of CNS stimulants; n (%) | 32 (0.5%) | 29 (0.4%) | 0.01 | 83 (0.5%) | 76 (0.5%) | 0.00 | 0,115 (0.5%) | 105 (0.5%) | 0.00 |
| Use of estrogens, progestins, androgens; n (%) | 274 (4.0%) | 261 (3.8%) | 0.01 | 634 (4.2%) | 643 (4.3%) | 0.00 | 0,908 (4.1%) | 904 (4.1%) | 0.00 |
| Use of Angiogenesis inhibitors; n (%) | 2 (0.0%) | 0 (0.0%) | #DIV/0! | 15 (0.1%) | 2 (0.0%) | 0.04 | 0,017 (0.1%) | 2 (0.0%) | 0.04 |
| Use of Oral Immunosuppressants; n (%) | 4 (0.1%) | 6 (0.1%) | 0.00 | 38 (0.3%) | 29 (0.2%) | 0.02 | 0,042 (0.2%) | 35 (0.2%) | 0.00 |
| Use of fondaparinux or Bivalirudin; n | 0 (0.0%) | 3 (0.0%) | #DIV/0! | 7 (0.0%) | 2 (0.0%) | #DIV/0! | 0,007 (0.0%) | 5 (0.0%) | #DIV/0! |
| (%) | | | | | | | | | |
| Use of other direct thrombin inhibitors | 0 (0.0%) | 0 (0.0%) | #DIV/0! | 0 (0.0%) | 0 (0.0%) | #DIV/0! | 0,000 (0.0%) | 0 (0.0%) | #DIV/0! |
| (lepirudin, desirudin, argatroban); n (%) | | | | | | | | | |
| Use of Prasugrel ON CED; n (%) | 90 (1.3%) | 82 (1.2%) | 0.01 | 104 (0.7%) | 122 (0.8%) | -0.01 | 0,194 (0.9%) | 204 (0.9%) | 0.00 |
| Use of Prasugrel 180 to 1 day prior; n | 94 (1.4%) | 90 (1.3%) | 0.01 | 112 (0.7%) | 134 (0.9%) | -0.02 | 0,206 (0.9%) | 224 (1.0%) | -0.01 |
| (%) | | | | | | | | | |
| Duration of index hospitalization (i.e. anchor hospitalization LOS) | | | | | | | | | |

Table 1: Prasugrel 10 mg vs Clopidogrel 75 mg

| mean (sd) | 3.38 (1.65) | 3.38 (1.50) | 0.00 | 3.39 (1.39) | 3.38 (1.34) | 0.01 | 3.39 (1.48) | 3.38 (1.39) | 0.01 |
|---|---|---|---|---|---|---|---|---|---|
| median [IQR] | 3.00 [3.00, 4.00] | 3.00 [3.00, 4.00] | 0.00 | 3.00 [3.00, 4.00] | 3.00 [3.00, 4.00] | 0.00 | 3.00 (1.48) | 3.00 (1.39) | 0.00 |
| Number of D-dimer tests | | | | | | | | | |
| mean (sd) | 0.02 (0.17) | 0.02 (0.17) | 0.00 | 0.06 (0.26) | 0.06 (0.26) | 0.00 | 0.05 (0.24) | 0.05 (0.24) | 0.00 |
| median [IQR] | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 | 0.00 (0.24) | 0.00 (0.24) | 0.00 |
| Numbe of CRP, high-sensitivity CRP | | | | | | | | | |
| tests | | | | | | | | | |
| mean (sd) | 0.04 (0.23) | 0.04 (0.24) | 0.00 | 0.04 (0.25) | 0.04 (0.28) | 0.00 | 0.04 (0.24) | 0.04 (0.27) | 0.00 |
| median [IQR] | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 | 0.00 (0.24) | 0.00 (0.27) | 0.00 |
| Number of PT or aPTTt tests | | | | | | | | | |
| mean (sd) | 0.22 (1.04) | 0.22 (0.99) | 0.00 | 0.43 (0.98) | 0.43 (1.00) | 0.00 | 0.36 (1.00) | 0.36 (1.00) | 0.00 |
| median [IQR] | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 | 0.00 (1.00) | 0.00 (1.00) | 0.00 |
| Number of Bleeding time tests | | | | | | | | | |
| mean (sd) | 0.00 (0.01) | 0.00 (0.01) | 0.00 | 0.00 (0.00) | 0.00 (0.01) | 0.00 | 0.00 (0.01) | 0.00 (0.01) | 0.00 |
| median [IQR] | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 | 0.00 (0.01) | 0.00 (0.01) | 0.00 |
| HAS-BLED Score (ICD-9 and ICD-10), | | | | | | | | | |
| 180 days | | | | | | | | | |
| mean (sd) | 3.41 (0.67) | 3.42 (0.67) | -0.01 | 3.16 (0.49) | 3.16 (0.50) | 0.00 | 3.24 (0.55) | 3.24 (0.56) | 0.00 |
| median [IQR] | 3.00 [3.00, 4.00] | 3.00 [3.00, 4.00] | 0.00 | 3.00 [3.00, 3.00] | 3.00 [3.00, 3.00] | 0.00 | 3.00 (0.55) | 3.00 (0.56) | 0.00 |
| Drug eluting stent; n (%) | 3,921 (57.4%) | 3,947 (57.7%) | -0.01 | 7,223 (47.8%) | 7,159 (47.4%) | 0.01 | 11,144 (50.8%) | 11106 (50.6%) | 0.00 |
| Bare metal stent; n (%) | 4,286 (62.7%) | 4,285 (62.7%) | 0.00 | 7,177 (47.5%) | 7,200 (47.7%) | 0.00 | 11,463 (52.3%) | 11485 (52.4%) | 0.00 |
| Use of CYP inhibitors; n (%) | 1,028 (15.0%) | 1,027 (15.0%) | 0.00 | 2,162 (14.3%) | 2,184 (14.5%) | -0.01 | 3,190 (14.5%) | 3211 (14.6%) | 0.00 |
| Use of CYP inducers; n (%) | 27 (0.4%) | 32 (0.5%) | -0.01 | 94 (0.6%) | 83 (0.5%) | 0.01 | 0,121 (0.6%) | 115 (0.5%) | 0.01 |
| Commercial vs Medicare Advantage- | | | | | | | | | |
| Business Type Code - CORRECT ONE - | | | | | | | | | |
| TRUVEN | | | | | | | | | |
| Commercial; n (%) | 4,740 (69.3%) | 4,686 (68.6%) | 0.02 | 2,090 (13.8%) | 2,184 (14.5%) | -0.02 | 6,830 (31.1%) | 6870 (31.3%) | 0.00 |
| Medicare Advantage; n (%) | 2,095 (30.7%) | 2,149 (31.4%) | -0.02 | 13,007 (86.2%) | 12,913 (85.5%) | 0.02 | 15,102 (68.9%) | 15062 (68.7%) | 0.00 |
| Commercial vs Medicare Advantage- | | | | | | | | | |
| Business Type Code | | | | | | | | | |
| COM = COMMERCIAL; n (%) | 4,740 (69.3%) | 4,686 (68.6%) | 0.02 | - | - | #VALUE! | 4,740 (69.3%) | 4,686 (68.6%) | 0.02 |
| MCR = MEDICARE; n (%) | 2,095 (30.7%) | 2,149 (31.4%) | -0.02 | - | - | #VALUE! | 2,095 (30.7%) | 2,149 (31.4%) | -0.02 |
| MCD = MEDICAID; n (%) | 0 (0.0%) | 0 (0.0%) | #DIV/0! | - | - | #VALUE! | 0 (0.0%) | 0 (0.0%) | #DIV/0! |
| NONE = NO BUSINESS LINE CODE | 0 (0.0%) | 0 (0.0%) | #DIV/0! | - | - | #VALUE! | 0 (0.0%) | 0 (0.0%) | #DIV/0! |
| (added in 2015); n (%) | | | | | | | | | |
| UNK = UNKNOWN (added in 2015); n | 0 (0.0%) | 0 (0.0%) | #DIV/0! | - | - | #VALUE! | 0 (0.0%) | 0 (0.0%) | #DIV/0! |
| (%) | | | | | | | | | |
| Commercial vs Medicare Advantage- | | | | | | | | | |
| Data Type | | | | | | | | | |
| 1 - Fee For Service; n (%) | - | - | #VALUE! | 11,534 (76.4%) | 11,465 (75.9%) | 0.01 | 11,534 (76.4%) | 11,465 (75.9%) | 0.01 |
| 2 - Encounter; n (%) | - | - | #VALUE! | 1,473 (9.8%) | 1,448 (9.6%) | 0.01 | 1,473 (9.8%) | 1,448 (9.6%) | 0.01 |
| 3 - Medicare; n (%) | - | - | #VALUE! | 1,821 (12.1%) | 1,920 (12.7%) | -0.02 | 1,821 (12.1%) | 1,920 (12.7%) | -0.02 |
| 4 - Medicare Encounter; n (%) | - | - | #VALUE! | 269 (1.8%) | 264 (1.7%) | 0.01 | 269 (1.8%) | 264 (1.7%) | 0.01 |
| Metropolitan Statistical Area - Urban | | | | | | | | | |
| (any MSA) vs Rural (non-MSA) | | | | | | | | | |
| Urban; n (%) | - | - | #VALUE! | 11,804 (78.2%) | 11,827 (78.3%) | 0.00 | 11,804 (78.2%) | 11,827 (78.3%) | 0.00 |
| Rural; n (%) | - | - | #VALUE! | 260 (1.7%) | 269 (1.8%) | -0.01 | 260 (1.7%) | 269 (1.8%) | -0.01 |
| Unknown/Missing; n (%) | - | - | #VALUE! | 3,033 (20.1%) | 3,001 (19.9%) | 0.01 | 3,033 (20.1%) | 3,001 (19.9%) | 0.01 |

Table 1: Prasugrel 10 mg vs Clopidogrel 75 mg

| N of Generic name drugs | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|
| mean (sd) | 11.18 (9.42) | 11.14 (10.51) | 0.00 | 9.48 (7.70) | 9.50 (8.54) | -0.00246 | 10.01 (8.27) | 10.01 (9.20) | 0.00 |
| median [IQR] | 8.00 [5.00, 15.00] | 8.00 [4.00, 15.00] | 0.00 | 7.00 [4.00, 12.00] | 7.00 [4.00, 12.00] | 0 | 7.31 (8.27) | 7.31 (9.20) | 0.00 |
| N of Brand name drugs | | | | | | | | | |
| mean (sd) | 3.70 (5.32) | 3.73 (4.20) | -0.01 | 3.86 (4.85) | 3.93 (3.99) | -0.02 | 3.81 (5.00) | 3.87 (4.06) | 0.05 |
| median [IQR] | 2.00 [1.00, 5.00] | 2.00 [1.00, 5.00] | 0.00 | 2.00 [1.00, 5.00] | 2.00 [2.00, 5.00] | 0 | 2.00 (5.00) | 2.00 (4.06) | 0.05 |